CLINICAL TRIAL: NCT04961541
Title: A Phase 1/2, Randomized, Observer-Blinded Study to Evaluate the Safety and Immunogenicity of a Quadrivalent Hemagglutinin Nanoparticle Influenza and SARS-CoV-2 rS Nanoparticle Combination Vaccine With Matrix M1™ Adjuvant in Healthy Participants ≥ 50 to ≤ 70 Years of Age
Brief Title: Evaluation of the Safety and Immunogenicity of Influenza and COVID-19 Combination Vaccine
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novavax (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2019nCoV-ICC-E-101
Record Dates: First submitted 2021-07-09; First posted 2021-07-14 (Actual); Results first posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: SARS-CoV Infection; Covid19
Keywords: Coronavirus
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; COVID-19; Coronavirus Infections | interventions — Matrix-M

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (14):
- Group A and Group C - ICC Vaccine Formulation (Experimental): 2 doses of Formulation 1. 1 dose each on Days 0 and Day 56.
  Interventions: Biological: ICC Vaccine
- Group B -ICC Vaccine Formulation (Experimental): 2 doses of Formulation 2. 1 dose each on Days 0 and Day 56.
  Interventions: Biological: ICC Vaccine
- Group D - ICC Vaccine Formulation (Experimental): 2 doses of Formulation 3. 1 dose each on Days 0 and Day 56.
  Interventions: Biological: ICC Vaccine
- Group E - ICC Vaccine Formulation (Experimental): 2 doses of Formulation 4. 1 dose each on Days 0 and Day 56.
  Interventions: Biological: ICC Vaccine
- Group F- ICC Vaccine Formulation (Experimental): 2 doses of Formulation 5. 1 dose each on Days 0 and Day 56.
  Interventions: Biological: ICC Vaccine
- Group G- ICC Vaccine Formulation (Experimental): 2 doses of Formulation 6. 1 dose each on Days 0 and Day 56.
  Interventions: Biological: ICC Vaccine
- Group H and Group N- ICC Vaccine Formulation (Experimental): 2 doses of Formulation 7. 1 dose each on Day 0 and Day 56.
  Interventions: Biological: ICC Vaccine
- Group I- ICC Vaccine Formulation (Experimental): 2 doses of Formulation 8. 1 dose each on Days 0 and Day 56.
  Interventions: Biological: ICC Vaccine
- Group J -ICC Vaccine Formulation (Experimental): 2 doses of Formulation 9. 1 dose each on Days 0 and Day 56.
  Interventions: Biological: ICC Vaccine
- Group K - ICC Vaccine Formulation (Experimental): 2 doses of Formulation 10. 1 dose each on Days 0 and Day 56.
  Interventions: Biological: ICC Vaccine
- Group L - ICC Vaccine Formulation (Experimental): 2 doses of Formulation 11. 1 dose each on Days 0 and Day 56.
  Interventions: Biological: ICC Vaccine
- Group M -ICC Vaccine Formulation (Experimental): 2 doses of Formulation 12. 1 dose each on Days 0 and Day 56.
  Interventions: Biological: ICC Vaccine
- Group O - qNIV with Matrix-M1 adjuvant (Experimental): 2 doses of Formulation 13. 1 dose each on Days 0 and Day 56 and an additional dose of 5 µg SARS-CoV-2 rS+50 µg Matrix-M1 at Day 70.
  Interventions: Biological: qNIV Nanoparticle Vaccine2 in-clinic mixed with Matrix-M1 Adjuvant
- Group P- SARS-CoV-2 rS with Matrix-M1 adjuvant (Experimental): 2 doses of Formulation 14. 1 dose each on Days 0 and Day 56.
  Interventions: Biological: SARS-CoV-2 rS Nanoparticle Vaccine in-clinic mixed with Matrix-M1 Adjuvant

INTERVENTIONS:
Biological: ICC Vaccine — Intramuscular (deltoid) injections of in-clinic mix of various doses of quadrivalent hemagglutinin nanoparticle influenza vaccine(qNIV2), SARS-CoV-2 rS, and 50 μg Matrix-M1 Adjuvant (ICC Vaccine) on Day 0 and Day 56.
  Arms: Group A and Group C - ICC Vaccine Formulation; Group B -ICC Vaccine Formulation; Group D - ICC Vaccine Formulation; Group E - ICC Vaccine Formulation; Group F- ICC Vaccine Formulation; Group G- ICC Vaccine Formulation; Group H and Group N- ICC Vaccine Formulation; Group I- ICC Vaccine Formulation; Group J -ICC Vaccine Formulation; Group K - ICC Vaccine Formulation; Group L - ICC Vaccine Formulation; Group M -ICC Vaccine Formulation
Biological: qNIV Nanoparticle Vaccine2 in-clinic mixed with Matrix-M1 Adjuvant — Intramuscular (deltoid) injections of 60 μg qNIV Nanoparticle Vaccine2 in-clinic mixed with 75 μg Matrix-M1 Adjuvant on Days 0, Day 56, and an additional dose on Day 70.
  Arms: Group O - qNIV with Matrix-M1 adjuvant
Biological: SARS-CoV-2 rS Nanoparticle Vaccine in-clinic mixed with Matrix-M1 Adjuvant — Intramuscular (deltoid) injections of 5 μg SARS-CoV-2 rS Nanoparticle Vaccine in-clinic mixed with 50 μg Matrix-M1 Adjuvant on Days 0 and Day 56.
  Arms: Group P- SARS-CoV-2 rS with Matrix-M1 adjuvant

SUMMARY:
This is a randomized, observer-blinded, Phase 1/2 study evaluating the safety and immunogenicity of a quadrivalent HA nanoparticle influenza and SARS-CoV-2 rS nanoparticle combination vaccine with Matrix-M1 adjuvant; this combination is referred to as ICC vaccine.

DETAILED DESCRIPTION:
This is a randomized, observer-blinded, Phase 1/2 study evaluating the safety and immunogenicity of a quadrivalent hemagglutinin (HA) nanoparticle influenza vaccine (qNIV) and severe acute respiratory syndrome coronavirus 2 (SARSCoV2) recombinant spike (rS) nanoparticle combination vaccine with Matrix-M1™ adjuvant; this combination vaccine is referred to as Influenza COVID-19 Combination (ICC) vaccine.

The study will enroll approximately 640 healthy (based on history and physical examination) adult male and female participants 50 to 70 years of age, inclusive, targeting participants who are baseline seropositive (either previously infected with SARS-CoV-2 ≥ 8 weeks prior to enrollment, or have been previously immunized against SARS-CoV-2 with a completed regimen of an authorized vaccine at ≥ 8 weeks prior to enrollment). Randomization will be stratified on age ≥ 50 to ≤60 or

≥ 60 to ≤ 70 years to distribute the proportions of each age stratum evenly across vaccine groups.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, medically stable adult males or females ≥ 50 to ≤ 70 years of age at screening.
2. Willing and able to give informed consent prior to study enrollment.
3. Able to attend study visits, comply with study requirements, and provide reliable and complete reports of AEs.
4. Participants must have been baseline seropositive to SARS-CoV-2 defined as either:

   • Having completed a primary vaccination series against SARS-CoV-2 with an authorized COVID-19 vaccine with receipt of second/final dose of authorized vaccine ≥ 8 weeks prior to enrollment (first study vaccination).

   OR

   • Previously infected with SARS CoV-2 ≥ 8 weeks prior to enrollment (first study vaccination).

   Note: Baseline SARS-CoV-2 serostatus determination at screening will be based on vaccination documentation (eg, vaccination card or vaccination registry) or participants' report of a previous SARS-CoV-2 infection.
5. Women of childbearing potential (defined as any female participant who is NOT surgically sterile [ie, hysterectomy, bilateral tubal ligation, or bilateral oophorectomy] or postmenopausal [defined as amenorrhea at least 12 consecutive months]) must agree to be heterosexually inactive from at least 28 days prior to enrollment and through the end of the study OR agree to consistently use a medically acceptable method of contraception listed below from at least 28 days prior to enrollment and through the end of the study.

   1. Condoms (male or female) with spermicide (if acceptable in-country)
   2. Diaphragm with spermicide
   3. Cervical cap with spermicide
   4. Intrauterine device
   5. Oral or patch contraceptives
   6. Norplant®, Depo-Provera®, or other in-country regulatory approved contraceptive method that is designed to protect against pregnancy
   7. Abstinence, as a form of contraception, is acceptable if in line with the participant's lifestyle
6. Participants must be healthy and medically stable, as determined by the investigator (based on a review of health status, vital signs [to include body temperature], medical history, and targeted physical examination [to include body weight]). Participants must have a body mass index (BMI) of 17 to 34 kg/m2, inclusive, at screening. Vital signs must be within medically acceptable ranges prior to the first vaccination.
7. Participants must agree to not participate in any other SARS-CoV-2 or influenza prevention or treatment studies for the duration of the study. Note: For participants who become hospitalized with COVID-19, participation in investigational treatment studies is permitted.

Exclusion Criteria:

1. Any ongoing, symptomatic acute, or chronic illness requiring medical or surgical care.

   * Asymptomatic chronic conditions or findings (eg, mild hypertension, dyslipidemia) that are not associated with evidence of end-organ damage are not exclusionary provided that they are being appropriately managed and are clinically stable (ie, unlikely to result in symptomatic illness within the time-course of this study), in the opinion of the investigator.
   * Acute or chronic illnesses or conditions which may be reasonably predicted to become symptomatic if treatment were withdrawn or interrupted are exclusionary, even if stable.
   * Acute or chronic illnesses reasonably expected to be associated with increased risks in the event of influenza or SARS-CoV-2 infection (eg, cardio-pulmonary diseases, diabetes mellitus, renal or hepatic dysfunction, hemoglobinopathies) are exclusionary, even if stable.
2. Participation in research involving an investigational product (drug/biologic/device) within 90 days before the planned date of the first injection.
3. Use of COVID-19 prophylactic or treatment monoclonal antibodies or antibody cocktails within 90 days prior to the planned date of the first injection.
4. History of a serious reaction to prior influenza vaccination or known allergy to constituents of influenza vaccines - including egg proteins - or polysorbate 80; or any known allergies to products contained in the investigational product.
5. Any history of anaphylaxis to any prior vaccine.
6. History of Guillain-Barré Syndrome within 6 weeks following a previous influenza vaccine.
7. Receipt of any vaccine in the 4 weeks preceding the study vaccination and any influenza vaccine within 2 months preceding the study vaccination. Note: Routine vaccinations will not be allowed until after study Day 70.
8. Any known or suspected autoimmune or immunosuppressive illness, congenital or acquired, based on medical history and/or physical examination.
9. Chronic administration (defined as more than 14 continuous days) of immunosuppressants or other immune-modifying drugs within 6 months prior to the administration of the study vaccines. An immunosuppressant dose of glucocorticoid will be defined as a systemic dose ≥ 10 mg of prednisone per day or equivalent. The use of topical, inhaled, and nasal glucocorticoids will be permitted.
10. Administration of immunoglobulins and/or any blood products within the 3 months preceding the administration of the study vaccine or during the study.
11. Active cancer (malignancy) therapy within 3 years prior to first study vaccination (with the exception of adequately treated non-melanomatous skin carcinoma or lentigo maligna and uterine cervical carcinoma in situ without evidence of disease, at the discretion of the investigator).
12. Participants who are breastfeeding, pregnant, or who plan to become pregnant prior to the EoS.
13. Known disturbance of coagulation.
14. Suspected or known history of alcohol abuse or drug addiction within 2 years prior to the first trial vaccine dose that, in the opinion of the investigator, might interfere with protocol compliance.
15. Acute disease at the time of enrollment (defined as the presence of a moderate or severe illness with or without fever, or an oral temperature > 38.0°C, on the planned day of vaccine administration).
16. Any condition that in the opinion of the investigator would pose a health risk to the participant if enrolled or could interfere with evaluation of the vaccine or interpretation of study results (including neurologic or psychiatric conditions deemed likely to impair the quality of safety reporting).
17. Study team member or immediate family member of any study team member (inclusive of Sponsor, Contract Research Organization, and study site personnel involved in the conduct or planning of the study).

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 637 (Actual)
Dates: Start 2021-09-08 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2022-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development, Study Director — Novavax
Locations (10):
- Australia (10):
  - Paratus Clinical Research - Canberra, Bruce, Australian Capital Territory
  - Paratus Clinical Research - Western Sydney, Blacktown, New South Wales
  - Northern Beaches Clinical Research, Brookvale, New South Wales
  - Paratus Clinical Research - Central Coast, Kanwal, New South Wales
  - Hunter Diabetes Centre, Merewether, New South Wales
  - University of the Sunshine Coast,Southbank, Brisbane, Queensland
  - University of the Sunshine Coast, Health Hub Morayfield, Morayfield, Queensland
  - University of the Sunshine Coast, Sippy Downs, Queensland
  - Austrials Pty Ltd - Taringa, Taringa, Queensland
  - Emeritus Research, Camberwell, Victoria

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A and Group C - ICC Vaccine Formulation: 2 doses of Formulation 1. 1 dose each on Days 0 and Day 56.
  ICC Vaccine: Intramuscular (deltoid) injections of in-clinic mix of various doses of qNIV2, SARS-CoV-2 rS, and 50 μg Matrix-M1 Adjuvant (ICC Vaccine) on Day 0 and Day 56.
- Group B -ICC Vaccine Formulation: 2 doses of Formulation 2. 1 dose each on Days 0 and Day 56.
  ICC Vaccine: Intramuscular (deltoid) injections of in-clinic mix of various doses of qNIV2, SARS-CoV-2 rS, and 50 μg Matrix-M1 Adjuvant (ICC Vaccine) on Day 0 and Day 56.
- Group D - ICC Vaccine Formulation: 2 doses of Formulation 3. 1 dose each on Days 0 and Day 56.
  ICC Vaccine: Intramuscular (deltoid) injections of in-clinic mix of various doses of qNIV2, SARS-CoV-2 rS, and 50 μg Matrix-M1 Adjuvant (ICC Vaccine) on Day 0 and Day 56.
- Group E - ICC Vaccine Formulation: 2 doses of Formulation 4. 1 dose each on Days 0 and Day 56.
  ICC Vaccine: Intramuscular (deltoid) injections of in-clinic mix of various doses of qNIV2, SARS-CoV-2 rS, and 50 μg Matrix-M1 Adjuvant (ICC Vaccine) on Day 0 and Day 56.
- Group F- ICC Vaccine Formulation: 2 doses of Formulation 5. 1 dose each on Days 0 and Day 56.
  ICC Vaccine: Intramuscular (deltoid) injections of in-clinic mix of various doses of qNIV2, SARS-CoV-2 rS, and 50 μg Matrix-M1 Adjuvant (ICC Vaccine) on Day 0 and Day 56.
- Group G- ICC Vaccine Formulation: 2 doses of Formulation 6. 1 dose each on Days 0 and Day 56.
  ICC Vaccine: Intramuscular (deltoid) injections of in-clinic mix of various doses of qNIV2, SARS-CoV-2 rS, and 50 μg Matrix-M1 Adjuvant (ICC Vaccine) on Day 0 and Day 56.
- Group H and Group N- ICC Vaccine Formulation: 2 doses of Formulation 7. 1 dose each on Day 0 and Day 56.
  ICC Vaccine: Intramuscular (deltoid) injections of in-clinic mix of various doses of qNIV2, SARS-CoV-2 rS, and 50 μg Matrix-M1 Adjuvant (ICC Vaccine) on Day 0 and Day 56.
- Group I- ICC Vaccine Formulation: 2 doses of Formulation 8. 1 dose each on Days 0 and Day 56.
  ICC Vaccine: Intramuscular (deltoid) injections of in-clinic mix of various doses of qNIV2, SARS-CoV-2 rS, and 50 μg Matrix-M1 Adjuvant (ICC Vaccine) on Day 0 and Day 56.
- Group J -ICC Vaccine Formulation: 2 doses of Formulation 9. 1 dose each on Days 0 and Day 56.
  ICC Vaccine: Intramuscular (deltoid) injections of in-clinic mix of various doses of qNIV2, SARS-CoV-2 rS, and 50 μg Matrix-M1 Adjuvant (ICC Vaccine) on Day 0 and Day 56.
- Group K - ICC Vaccine Formulation: 2 doses of Formulation 10. 1 dose each on Days 0 and Day 56.
  ICC Vaccine: Intramuscular (deltoid) injections of in-clinic mix of various doses of qNIV2, SARS-CoV-2 rS, and 50 μg Matrix-M1 Adjuvant (ICC Vaccine) on Day 0 and Day 56.
- Group L - ICC Vaccine Formulation: 2 doses of Formulation 11. 1 dose each on Days 0 and Day 56.
  ICC Vaccine: Intramuscular (deltoid) injections of in-clinic mix of various doses of qNIV2, SARS-CoV-2 rS, and 50 μg Matrix-M1 Adjuvant (ICC Vaccine) on Day 0 and Day 56.
- Group M -ICC Vaccine Formulation: 2 doses of Formulation 12. 1 dose each on Days 0 and Day 56.
  ICC Vaccine: Intramuscular (deltoid) injections of in-clinic mix of various doses of qNIV2, SARS-CoV-2 rS, and 50 μg Matrix-M1 Adjuvant (ICC Vaccine) on Day 0 and Day 56.
Period: Overall Study
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant | Group P- SARS-CoV-2 rS With Matrix-M1 Adjuvant
Started | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39 | 40
Completed | 80 | 40 | 35 | 36 | 41 | 40 | 80 | 38 | 39 | 38 | 40 | 41 | 38 | 40
Not Completed | 0 | 0 | 4 | 1 | 0 | 1 | 1 | 1 | 0 | 2 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant | Group P- SARS-CoV-2 rS With Matrix-M1 Adjuvant | Total
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39 | 40 | 637
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (5.3) | 59 (5.5) | 58 (5.5) | 60 (5.4) | 59 (6.1) | 59 (6.0) | 59 (6.1) | 59 (6.5) | 59 (5.7) | 59 (5.1) | 58 (6.3) | 59 (5.7) | 58 (5.5) | 59 (6.0) | 59 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 28 | 25 | 25 | 26 | 25 | 50 | 19 | 27 | 27 | 22 | 29 | 28 | 24 | 398
  Male | 37 | 12 | 14 | 12 | 15 | 16 | 31 | 20 | 12 | 13 | 18 | 12 | 11 | 16 | 239
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 8
  Not Hispanic or Latino | 79 | 39 | 39 | 36 | 39 | 40 | 80 | 39 | 39 | 38 | 40 | 41 | 39 | 39 | 627
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 1 | 0 | 1 | 0 | 0 | 2 | 3 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 76 | 39 | 37 | 36 | 41 | 39 | 76 | 39 | 39 | 38 | 39 | 39 | 38 | 39 | 615
  More than one race | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 4
  Unknown or Not Reported | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 7
Regimen of Previous COVID Vaccine [Count of Participants; unit: Participants]
  Pfizer-BioNtech | 30 | 11 | 12 | 8 | 16 | 14 | 29 | 8 | 11 | 16 | 10 | 9 | 13 | 11 | 198
  Oxford-AstraZeneca | 50 | 28 | 27 | 29 | 25 | 26 | 52 | 30 | 28 | 24 | 30 | 31 | 26 | 29 | 435
  Mixed or Other | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Local and Systemic Adverse Events (AE's)
Description: Numbers of participants with solicited local and systemic AEs over the 7 days post-injection after first and second doses.
Time Frame: Day 0 to Day 63
Population: Safety Analysis Set Population
Measure: Number; unit: participants
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant | Group P- SARS-CoV-2 rS With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39 | 40
participants
  Local AEs | 71 | 32 | 32 | 28 | 38 | 36 | 64 | 32 | 28 | 34 | 34 | 39 | 34 | 35
  Systemic AEs | 50 | 17 | 27 | 24 | 29 | 27 | 59 | 29 | 20 | 28 | 26 | 30 | 27 | 30

2. Primary Outcome: Number of Participants Reporting All AE's
Description: Number of participants reporting all AEs, (solicited and unsolicited), over 70 days after the first dose.
Time Frame: Day 0 to Day 70
Measure: Count of Participants; unit: Participants
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant | Group P- SARS-CoV-2 rS With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39 | 40
Participants
  Solicited AEs | 77 | 33 | 35 | 34 | 39 | 39 | 70 | 37 | 31 | 38 | 34 | 39 | 38 | 39
  Unsolicited AEs | 25 | 15 | 14 | 17 | 16 | 20 | 30 | 9 | 17 | 19 | 10 | 16 | 18 | 14

3. Primary Outcome: Number of Participants With MAAEs, AESIs (Including PIMMCs), SAEs
Description: Number of participants with Medical Attended Adverse Events (MAAE's), Adverse events (AESI's), Including potential immune-mediated medical conditions (PIMMCs), Serious Adverse Events SAEs.
Time Frame: Day 0 to Day 180
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant | Group P- SARS-CoV-2 rS With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39 | 40
Participants
  SAEs | 2 | 1 | 2 | 0 | 2 | 1 | 3 | 2 | 0 | 0 | 5 | 0 | 1 | 1
  AESIs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  MAAEs | 14 | 8 | 7 | 12 | 10 | 11 | 20 | 9 | 14 | 7 | 7 | 7 | 14 | 12

4. Secondary Outcome: Hemagglutination-Inhibition (HAI) Antibody Titers Specific for the Hemagglutinin (HA) Receptor Binding Domains of Vaccine Homologous Influenza A/Brisbane (H1N1 Subtype) Strain Expressed as Geometric Mean Titers (GMTs)
Description: Hemagglutination-inhibition (HAI) antibody titers specific for the hemagglutinin (HA) receptor binding domains of vaccine homologous Influenza A/Brisbane (H1N1 Subtype) strain calculated as GMT, defined as the antilog of the mean of the log-transformed HAI titers on Days 56, 70, and other follow-up time points.
Time Frame: Day 0 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean Titers
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
Geometric Mean Titers
  Day 0 | 83.6 [66.4 to 105.3] | 66.7 [49.8 to 89.3] | 62.4 [44.8 to 86.9] | 91.2 [67.7 to 122.8] | 85.6 [62.6 to 117.1] | 77.3 [54.9 to 108.7] | 78.3 [61.6 to 99.4] | 89.8 [64.1 to 125.7] | 77.9 [55.4 to 109.5] | 96.8 [71.1 to 131.8] | 97.3 [68.1 to 138.9] | 81.4 [62.2 to 106.4] | 83.6 [60.1 to 116.4]
  Day 28 | 141.1 [116.9 to 170.4] | 91.9 [67.8 to 103.8] | 81.5 [63.9 to 103.8] | 107.0 [83.6 to 136.8] | 112.2 [84.6 to 148.8] | 106.6 [78.1 to 145.6] | 126.4 [103.0 to 155.2] | 105.4 [79.1 to 140.4] | 105.4 [61.5 to 111.8] | 141.3 [107.0 to 186.6] | 129.3 [93.7 to 178.3] | 103.1 [80.7 to 131.7] | 133.9 [104.2 to 172.2]
  Day 56 | 129.1 [107.5 to 154.9] | 86.7 [64.9 to 115.8] | 84.8 [63.9 to 112.4] | 100.8 [75.6 to 134.3] | 100.2 [75.4 to 133.2] | 95.1 [71.5 to 126.7] | 107.3 [88.4 to 130.4] | 94.7 [70.5 to 127.2] | 73.7 [54.3 to 100.1] | 126.6 [90.1 to 177.9] | 109.1 [77.4 to 153.7] | 99.3 [77.3 to 127.6] | 118.3 [90.5 to 154.6]
  Day 70 | 149.6 [123.6 to 181.0] | 124.8 [93.9 to 165.8] | 113.1 [84.4 to 151.7] | 142.5 [105.7 to 192.3] | 135.7 [101.3 to 181.9] | 113.1 [86.7 to 147.6] | 128.5 [105.2 to 157.1] | 123.9 [96.6 to 159.0] | 95.1 [72.8 to 124.3] | 156.9 [118.8 to 207.4] | 148.4 [105.6 to 208.6] | 129.5 [106.9 to 157.0] | 119.5 [93.0 to 153.5]
  Day 84 | 107.7 [89.2 to 130.1] | 85.1 [63.3 to 114.5] | 96.1 [73.6 to 125.5] | 98.5 [75.4 to 128.6] | 101.7 [72.4 to 142.8] | 68.5 [50.6 to 92.7] | 99.1 [80.6 to 122.0] | 75.1 [59.1 to 95.2] | 74.4 [58.7 to 94.3] | 103.2 [75.7 to 140.7] | 110.0 [76.1 to 158.9] | 89.3 [70.8 to 112.7] | 90.1 [68.0 to 119.3]
  Day 182 | 85.0 [69.8 to 103.4] | 57.1 [41.7 to 78.1] | 68.7 [51.1 to 92.2] | 72.5 [54.6 to 96.1] | 70.6 [51.3 to 97.3] | 60.9 [43.8 to 84.5] | 67.4 [53.9 to 84.3] | 58.7 [43.4 to 79.5] | 56.6 [43.9 to 72.9] | 83.1 [57.0 to 121.2] | 76.4 [53.9 to 108.3] | 65.2 [49.7 to 85.6] | 66.1 [48.5 to 90.0]

5. Secondary Outcome: Hemagglutination-Inhibition (HAI) Antibody Titers Specific for the HA Receptor Binding Domains of Vaccine Homologous Influenza A/Kansas (H3N2 Subtype) Strain Expressed as GMTs
Description: Hemagglutination-inhibition (HAI) antibody titers specific for the HA receptor binding domains of vaccine homologous Influenza A/Kansas (H3N2 Subtype) strain calculated as GMT, defined as the antilog of the mean of the log-transformed HAI titers on Days 56, 70, and other follow-up time points.
Time Frame: Day 0 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean Titers
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
Geometric Mean Titers
  Day 0 | 27.1 [22.7 to 32.3] | 27.1 [20.4 to 35.9] | 21.1 [16.0 to 27.7] | 31.1 [22.9 to 42.2] | 32.4 [24.3 to 43.2] | 29.8 [22.8 to 38.9] | 26.0 [21.3 to 31.8] | 32.9 [24.5 to 44.2] | 37.3 [27.5 to 50.4] | 26.4 [20.9 to 33.3] | 28.3 [21.3 to 37.6] | 30.5 [23.5 to 39.6] | 27.1 [20.2 to 36.2]
  Day 28 | 110.7 [88.5 to 138.5] | 96.8 [60.1 to 155.9] | 58.1 [39.9 to 84.7] | 77.1 [53.8 to 110.3] | 110.3 [77.2 to 157.7] | 80.7 [60.1 to 108.4] | 104.9 [82.7 to 133.1] | 75.8 [55.8 to 103.1] | 81.4 [58.8 to 112.7] | 116.2 [78.5 to 172.0] | 112.1 [82.4 to 152.7] | 109.4 [80.6 to 148.4] | 145.1 [103.0 to 204.4]
  Day 56 | 98.8 [78.0 to 125.0] | 79.3 [50.7 to 124.0] | 60.5 [41.3 to 88.6] | 71.3 [49.7 to 102.3] | 82.8 [58.6 to 117.1] | 65.5 [49.6 to 86.7] | 93.7 [74.6 to 117.6] | 67.0 [48.8 to 91.9] | 80.7 [59.7 to 109.1] | 87.0 [57.5 to 131.8] | 91.7 [64.8 to 129.9] | 96.8 [69.7 to 134.5] | 111.1 [79.7 to 155.1]
  Day 70 | 122.1 [99.6 to 149.8] | 115.2 [75.9 to 174.6] | 77.7 [52.6 to 114.6] | 111.0 [81.9 to 150.5] | 127.7 [92.9 to 175.6] | 98.5 [74.9 to 129.5] | 125.6 [101.8 to 155.1] | 104.2 [80.6 to 134.8] | 102.3 [75.8 to 138.2] | 115.3 [78.0 to 170.6] | 111.0 [81.4 to 151.5] | 113.1 [83.2 to 153.9] | 116.3 [81.8 to 165.3]
  Day 84 | 110.7 [90.3 to 135.5] | 104.4 [72.2 to 151.0] | 82.5 [58.1 to 117.1] | 85.7 [63.5 to 115.7] | 118.3 [88.3 to 158.4] | 88.4 [65.6 to 119.2] | 114.2 [94.7 to 137.6] | 88.4 [65.6 to 119.2] | 93.4 [68.9 to 126.6] | 90.4 [64.6 to 126.6] | 101.1 [74.2 to 137.8] | 104.8 [77.6 to 141.7] | 99.6 [73.2 to 135.5]
  Day 182 | 83.8 [68.6 to 102.4] | 74.5 [51.5 to 107.9] | 57.7 [40.7 to 81.9] | 57.1 [44.0 to 74.1] | 82.2 [62.6 to 107.8] | 65.5 [48.5 to 88.3] | 75.0 [61.7 to 91.2] | 68.2 [51.8 to 89.8] | 80.0 [61.5 to 104.0] | 68.6 [50.9 to 92.3] | 70.4 [52.0 to 95.3] | 80.7 [59.5 to 109.4] | 68.5 [50.6 to 92.7]

6. Secondary Outcome: Hemagglutination-Inhibition (HAI) Antibody Titers Specific for the HA Receptor Binding Domains of Vaccine Homologous Influenza A/Wisconsin (H1N1 Subtype) Strain Expressed as GMTs
Description: Hemagglutination-inhibition (HAI) antibody titers specific for the HA receptor binding domains of vaccine homologous Influenza A/Wisconsin (H1N1 Subtype) strain calculated as GMT, defined as the antilog of the mean of the log-transformed HAI titers on Days 56, 70, and other follow-up time points.
Time Frame: Day 0 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean Titers
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
Geometric Mean Titers
  Day 0 | 96.6 [79.9 to 116.8] | 85.0 [67.8 to 106.5] | 87.4 [70.2 to 108.9] | 100.2 [77.6 to 129.4] | 90.8 [67.9 to 121.5] | 96.0 [73.8 to 124.7] | 102.3 [82.6 to 126.6] | 89.0 [67.9 to 116.6] | 108.2 [83.5 to 140.2] | 104.6 [81.0 to 135.3] | 111.1 [83.1 to 148.6] | 87.8 [68.2 to 113.1] | 115.2 [87.3 to 152.0]
  Day 28 | 139.9 [118.1 to 165.7] | 108.3 [87.3 to 134.5] | 98.7 [80.6 to 120.8] | 111.0 [87.2 to 141.4] | 124.2 [100.0 to 154.1] | 117.0 [91.2 to 150.1] | 138.8 [116.3 to 165.6] | 100.8 [79.4 to 127.9] | 115.2 [91.9 to 144.4] | 132.8 [103.2 to 170.9] | 130.4 [98.7 to 172.3] | 114.1 [89.8 to 144.9] | 146.4 [117.3 to 182.7]
  Day 56 | 127.4 [106.8 to 151.8] | 95.6 [75.3 to 121.3] | 93.3 [73.9 to 117.9] | 105.8 [81.7 to 136.9] | 107.4 [82.9 to 139.2] | 100.2 [77.1 to 130.3] | 119.3 [101.4 to 140.2] | 98.1 [77.6 to 124.1] | 102.3 [79.7 to 131.4] | 126.6 [98.2 to 163.2] | 119.5 [91.2 to 156.7] | 98.5 [78.8 to 123.1] | 135.1 [104.2 to 175.3]
  Day 70 | 148.2 [123.4 to 178.0] | 109.2 [87.4 to 136.4] | 107.7 [85.3 to 135.9] | 125.8 [98.4 to 160.8] | 140.5 [107.5 to 183.6] | 107.4 [84.3 to 136.9] | 138.9 [116.5 to 165.6] | 114.2 [90.8 to 143.5] | 110.1 [88.9 to 136.4] | 146.7 [114.7 to 187.7] | 140.3 [108.2 to 182.1] | 121.1 [99.8 to 146.8] | 137.0 [105.2 to 178.5]
  Day 84 | 87.4 [73.2 to 104.5] | 68.2 [53.8 to 86.3] | 62.6 [47.8 to 82.1] | 69.6 [53.0 to 91.5] | 81.4 [62.0 to 107.0] | 72.4 [54.7 to 95.8] | 86.4 [71.0 to 105.3] | 66.7 [52.1 to 85.3] | 58.7 [46.1 to 74.7] | 79.2 [57.3 to 109.3] | 79.3 [55.7 to 112.7] | 74.1 [58.4 to 94.0] | 75.7 [57.1 to 100.4]
  Day 182 | 70.9 [59.1 to 85.2] | 50.4 [40.7 to 62.5] | 50.6 [38.4 to 66.5] | 57.1 [48.2 to 76.3] | 65.2 [49.8 to 85.4] | 60.3 [45.9 to 79.2] | 65.0 [53.6 to 78.7] | 54.0 [41.6 to 70.1] | 49.6 [39.2 to 62.8] | 70.6 [52.8 to 94.4] | 60.9 [44.5 to 83.3] | 61.3 [48.0 to 78.3] | 64.9 [48.6 to 86.6]

7. Secondary Outcome: Hemagglutination-Inhibition (HAI) Antibody Titers Specific for the HA Receptor Binding Domains of Vaccine Homologous Influenza A/Cambodia (H3N2 Subtype) Strain Expressed as GMTs
Description: Hemagglutination-inhibition (HAI) antibody titers specific for the HA receptor binding domains of vaccine homologous Influenza A/Cambodia (H3N2 Subtype) strain calculated as GMT, defined as the antilog of the mean of the log-transformed HAI titers on Days 56, 70, and other follow-up time points.
Time Frame: Day 0 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean Titers
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
Geometric Mean Titers
  Day 0 | 43.9 [36.6 to 52.5] | 41.8 [31.3 to 55.7] | 40.4 [30.1 to 54.2] | 42.3 [32.8 to 54.6] | 42.1 [32.5 to 54.4] | 45.6 [35.2 to 58.9] | 35.5 [29.7 to 42.5] | 40.7 [30.0 to 55.2] | 46.1 [34.0 to 62.5] | 36.4 [27.8 to 47.6] | 45.3 [34.1 to 60.1] | 41.4 [32.4 to 52.8] | 46.9 [35.3 to 62.4]
  Day 28 | 98.1 [77.3 to 124.4] | 90.3 [55.7 to 146.3] | 67.9 [46.8 to 98.4] | 70.2 [51.2 to 96.2] | 93.9 [64.9 to 135.9] | 84.2 [63.8 to 110.9] | 78.2 [61.7 to 99.2] | 66.4 [47.1 to 93.5] | 79.3 [55.8 to 112.7] | 89.0 [59.1 to 134.1] | 110.2 [76.9 to 157.8] | 76.0 [56.0 to 103.2] | 104.4 [77.4 to 141.0]
  Day 56 | 85.8 [66.9 to 110.1] | 80.0 [5.0 to 2560.0] | 68.3 [5.0 to 640.0] | 48.3 [10.0 to 640.0] | 73.4 [53.1 to 101.3] | 80.0 [10.0 to 1280.0] | 68.0 [53.8 to 85.9] | 40.0 [5.0 to 640.0] | 40.0 [5.0 to 640.0] | 79.3 [51.1 to 123.0] | 88.4 [59.5 to 131.5] | 64.4 [47.1 to 88.1] | 89.0 [65.0 to 121.9]
  Day 70 | 94.5 [75.3 to 118.6] | 92.2 [58.6 to 145.3] | 78.4 [53.3 to 115.4] | 74.1 [53.9 to 101.9] | 92.7 [67.6 to 127.2] | 85.7 [63.8 to 115.2] | 78.2 [62.0 to 98.6] | 83.0 [59.6 to 115.6] | 77.1 [52.9 to 112.6] | 85.6 [56.7 to 129.1] | 97.4 [67.7 to 140.1] | 79.3 [59.4 to 105.9] | 94.3 [70.0 to 127.0]
  Day 84 | 56.8 [45.0 to 71.7] | 65.2 [42.3 to 100.6] | 48.1 [33.0 to 69.9] | 45.5 [32.1 to 64.5] | 57.1 [40.7 to 80.1] | 55.5 [40.3 to 76.6] | 50.7 [40.4 to 63.6] | 51.6 [36.8 to 72.4] | 48.4 [33.3 to 70.6] | 53.8 [35.0 to 82.7] | 70.8 [48.7 to 102.9] | 46.6 [34.4 to 63.0] | 51.2 [36.6 to 71.6]
  Day 182 | 50.4 [40.5 to 62.7] | 55.6 [36.2 to 85.4] | 38.0 [25.7 to 56.2] | 33.5 [23.7 to 47.2] | 45.7 [33.9 to 61.6] | 42.6 [31.0 to 58.6] | 38.0 [30.6 to 47.3] | 44.8 [31.6 to 63.4] | 46.0 [32.9 to 64.5] | 44.9 [31.3 to 64.4] | 47.6 [33.3 to 68.0] | 38.6 [28.6 to 52.1] | 41.9 [30.1 to 58.2]

8. Secondary Outcome: Hemagglutination-Inhibition (HAI) Antibody Titers Specific for the HA Receptor Binding Domains of Vaccine Homologous Influenza A/Hong Kong (H3N2 Subtype) Strain Expressed as GMTs
Description: Hemagglutination-inhibition (HAI) antibody titers specific for the HA receptor binding domains of vaccine homologous Influenza A/Hong Kong (H3N2 Subtype) strain calculated as GMT, defined as the antilog of the mean of the log-transformed HAI titers on Days 56, 70, and other follow-up time points.
Time Frame: Day 0 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean Titers
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
Geometric Mean Titers
  Day 0 | 71.4 [61.1 to 83.4] | 69.6 [55.0 to 88.2] | 68.2 [53.4 to 87.0] | 70.8 [54.6 to 91.9] | 78.0 [62.0 to 98.2] | 79.3 [60.5 to 104.0] | 58.6 [49.6 to 69.2] | 73.2 [56.5 to 94.8] | 77.2 [58.0 to 102.8] | 56.6 [45.2 to 70.8] | 81.4 [63.2 to 105.0] | 67.6 [52.6 to 86.7] | 74.5 [57.1 to 97.3]
  Day 28 | 134.0 [110.9 to 161.8] | 126.6 [83.9 to 191.2] | 98.7 [73.3 to 132.8] | 100.2 [73.9 to 135.9] | 134.0 [95.0 to 189.0] | 113.1 [88.6 to 144.5] | 115.7 [95.0 to 140.9] | 107.3 [82.0 to 140.3] | 125.9 [91.5 to 173.2] | 117.2 [86.4 to 159.0] | 150.4 [107.1 to 211.0] | 117.0 [88.5 to 154.8] | 142.5 [107.2 to 189.6]
  Day 56 | 121.9 [99.4 to 149.6] | 111.1 [74.1 to 166.6] | 91.5 [68.1 to 123.0] | 95.1 [69.7 to 129.9] | 102.9 [76.3 to 138.7] | 110.2 [84.0 to 144.7] | 104.1 [85.2 to 127.2] | 93.9 [70.2 to 125.5] | 113.1 [82.8 to 154.6] | 95.6 [68.7 to 133.1] | 130.9 [94.3 to 181.8] | 103.7 [79.6 to 135.3] | 121.5 [92.2 to 160.0]
  Day 70 | 137.9 [112.2 to 169.5] | 142.5 [95.4 to 212.9] | 115.4 [83.4 to 159.8] | 117.6 [89.4 to 154.7] | 131.1 [96.9 to 177.3] | 127.7 [98.0 to 166.5] | 112.1 [91.6 to 137.1] | 112.1 [85.7 to 146.6] | 123.9 [88.1 to 174.3] | 111.0 [82.0 to 150.3] | 155.0 [111.2 to 216.2] | 115.1 [86.8 to 152.6] | 132.1 [101.4 to 172.1]
  Day 84 | 88.6 [70.5 to 111.3] | 99.0 [66.4 to 147.6] | 76.0 [51.4 to 112.4] | 80.8 [57.3 to 113.9] | 97.3 [69.2 to 136.8] | 90.9 [64.8 to 127.5] | 86.8 [69.5 to 108.5] | 83.7 [60.3 to 116.3] | 83.7 [58.1 to 120.8] | 79.2 [52.7 to 118.9] | 113.1 [77.0 to 166.3] | 93.1 [68.4 to 126.8] | 87.6 [64.6 to 118.9]
  Day 182 | 72.6 [58.6 to 89.9] | 81.4 [54.3 to 122.1] | 59.5 [42.1 to 84.2] | 62.5 [44.6 to 87.5] | 77.9 [57.1 to 106.3] | 69.8 [50.3 to 96.8] | 61.8 [50.3 to 75.8] | 69.5 [50.7 to 95.3] | 74.9 [53.8 to 104.3] | 66.6 [48.4 to 91.7] | 85.3 [60.1 to 120.9] | 72.5 [52.2 to 100.8] | 73.0 [53.7 to 99.3]

9. Secondary Outcome: Hemagglutination-Inhibition (HAI) Antibody Titers Specific for the HA Receptor Binding Domains of Vaccine Homologous Influenza B/Maryland (Victoria Subtype) Strain Expressed as GMTs
Description: Hemagglutination-inhibition (HAI) antibody titers specific for the HA receptor binding domains of vaccine homologous Influenza B/Maryland (Victoria Subtype) strain calculated as GMT, defined as the antilog of the mean of the log-transformed HAI titers on Days 56, 70, and other follow-up time points.
Time Frame: Day 0 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean Titers
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
Geometric Mean Titers
  Day 0 | 46.6 [38.7 to 56.2] | 40.3 [31.1 to 52.3] | 36.6 [36.6 to 48.8] | 39.3 [30.9 to 49.9] | 34.6 [27.0 to 44.4] | 36.4 [27.6 to 47.9] | 38.1 [31.2 to 46.6] | 41.4 [31.5 to 54.6] | 38.9 [28.2 to 53.7] | 45.9 [34.9 to 60.5] | 41.1 [31.8 to 53.1] | 42.1 [32.9 to 53.8] | 36.0 [26.8 to 48.2]
  Day 28 | 73.7 [62.3 to 87.2] | 63.3 [48.0 to 83.5] | 40.7 [31.2 to 53.2] | 52.0 [40.1 to 67.4] | 53.3 [40.2 to 70.8] | 47.0 [36.3 to 60.7] | 61.0 [51.0 to 73.0] | 49.1 [37.7 to 63.9] | 45.3 [33.4 to 61.4] | 59.7 [46.4 to 76.8] | 56.6 [42.6 to 75.1] | 58.0 [44.9 to 75.0] | 65.8 [48.4 to 89.5]
  Day 56 | 69.5 [58.1 to 83.2] | 54.6 [41.3 to 72.1] | 43.6 [32.7 to 58.2] | 55.5 [43.1 to 71.5] | 42.5 [31.7 to 56.9] | 44.8 [34.7 to 57.7] | 57.3 [47.7 to 68.8] | 47.8 [37.4 to 61.0] | 44.6 [33.4 to 59.6] | 57.1 [44.0 to 74.1] | 48.4 [36.2 to 64.8] | 52.3 [41.0 to 66.7] | 58.1 [43.8 to 77.0]
  Day 70 | 77.5 [64.8 to 92.8] | 65.2 [48.5 to 87.8] | 47.8 [34.6 to 66.1] | 61.1 [47.4 to 78.8] | 58.1 [44.2 to 76.3] | 50.5 [39.5 to 64.7] | 63.4 [53.3 to 75.4] | 55.5 [41.6 to 74.1] | 50.7 [38.9 to 66.1] | 66.0 [50.5 to 86.1] | 60.4 [45.2 to 80.8] | 64.2 [50.5 to 81.6] | 58.1 [43.6 to 77.5]
  Day 84 | 76.2 [63.2 to 91.9] | 69.4 [54.5 to 88.3] | 56.6 [41.9 to 76.4] | 57.7 [44.1 to 75.4] | 61.8 [47.8 to 80.0] | 56.6 [43.4 to 73.7] | 74.0 [62.5 to 87.7] | 51.6 [39.1 to 68.1] | 52.1 [39.9 to 68.0] | 65.2 [48.8 to 87.2] | 67.6 [51.9 to 88.0] | 65.3 [51.3 to 83.1] | 63.1 [49.4 to 80.6]
  Day 182 | 71.3 [59.5 to 85.3] | 60.2 [47.9 to 75.7] | 49.0 [37.0 to 65.0] | 50.7 [37.7 to 68.2] | 52.2 [40.8 to 66.9] | 48.0 [37.0 to 62.3] | 62.6 [52.1 to 75.2] | 49.6 [38.0 to 64.7] | 52.0 [41.0 to 66.0] | 55.5 [42.0 to 73.3] | 54.0 [40.5 to 72.2] | 55.1 [43.7 to 69.4] | 56.1 [43.9 to 71.5]

10. Secondary Outcome: Hemagglutination-Inhibition (HAI) Antibody Titers Specific for the HA Receptor Binding Domains of Vaccine Homologous Influenza B/Phuket (Yamagata Subtype) Strain Expressed as GMTs
Description: Hemagglutination-inhibition (HAI) antibody titers specific for the HA receptor binding domains of vaccine homologous Influenza B/Phuket (Yamagata Subtype) strain calculated as GMT, defined as the antilog of the mean of the log-transformed HAI titers on Days 56, 70, and other follow-up time points.
Time Frame: Day 0 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean Titers
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
Geometric Mean Titers
  Day 0 | 40.4 [33.7 to 48.3] | 36.1 [27.1 to 47.9] | 24.3 [18.3 to 32.4] | 33.2 [24.4 to 45.2] | 35.8 [27.5 to 46.7] | 35.4 [26.4 to 47.6] | 31.3 [25.7 to 38.1] | 38.3 [29.6 to 49.4] | 36.9 [28.9 to 47.2] | 36.1 [29.0 to 44.8] | 33.5 [26.9 to 41.7] | 35.5 [27.8 to 45.5] | 40.0 [5.0 to 640.0]
  Day 28 | 78.3 [65.2 to 93.9] | 57.6 [43.5 to 76.2] | 35.2 [26.7 to 46.4] | 47.8 [36.6 to 62.4] | 67.6 [53.0 to 86.2] | 50.7 [39.1 to 65.7] | 58.1 [48.5 to 69.6] | 60.2 [47.8 to 75.8] | 48.6 [38.1 to 62.0] | 59.7 [48.2 to 73.9] | 57.6 [45.9 to 72.2] | 68.7 [53.3 to 88.6] | 100.8 [81.8 to 124.1]
  Day 56 | 72.3 [60.5 to 86.4] | 53.2 [40.0 to 70.7] | 36.0 [26.7 to 48.5] | 44.5 [33.6 to 58.8] | 58.6 [45.0 to 76.3] | 47.2 [36.2 to 61.4] | 52.7 [43.8 to 63.4] | 57.1 [45.8 to 71.1] | 44.6 [35.8 to 55.6] | 55.5 [43.9 to 70.3] | 49.8 [39.1 to 63.3] | 62.2 [48.4 to 80.1] | 86.7 [69.2 to 108.6]
  Day 70 | 87.9 [71.9 to 107.6] | 72.5 [55.4 to 94.9] | 45.0 [32.8 to 61.9] | 61.7 [48.1 to 79.1] | 84.3 [64.8 to 109.6] | 59.1 [46.2 to 75.5] | 65.8 [54.6 to 79.2] | 67.9 [54.4 to 84.7] | 56.1 [44.6 to 70.5] | 69.9 [54.1 to 90.4] | 63.3 [49.9 to 80.3] | 74.1 [58.6 to 93.8] | 85.3 [66.8 to 108.8]
  Day 84 | 86.7 [73.0 to 102.9] | 71.9 [57.2 to 90.4] | 52.1 [39.9 to 68.1] | 60.6 [46.8 to 78.6] | 87.4 [69.8 to 109.6] | 63.7 [51.3 to 79.0] | 72.7 [60.9 to 86.7] | 65.5 [53.3 to 80.3] | 60.3 [47.9 to 75.9] | 73.0 [56.0 to 95.1] | 72.8 [57.1 to 92.9] | 76.7 [61.0 to 96.4] | 89.3 [72.3 to 110.2]
  Day 182 | 77.1 [64.4 to 92.3] | 61.3 [49.3 to 76.2] | 43.8 [33.4 to 57.6] | 53.3 [41.3 to 68.7] | 70.0 [54.9 to 89.2] | 52.6 [41.1 to 67.3] | 55.5 [46.8 to 65.9] | 57.1 [46.8 to 69.7] | 54.5 [44.1 to 67.3] | 61.7 [50.7 to 75.1] | 54.0 [42.9 to 68.1] | 60.7 [49.0 to 75.3] | 68.5 [55.3 to 84.9]

11. Secondary Outcome: Hemagglutination-Inhibition (HAI) Antibody Titers Specific for the HA Receptor Binding Domains of Vaccine Homologous Influenza B/Washington (Victoria Subtype) Strain Expressed as GMTs
Description: Hemagglutination-inhibition (HAI) antibody titers specific for the HA receptor binding domains of vaccine homologous Influenza B/Washington (Victoria Subtype) strain calculated as GMT, defined as the antilog of the mean of the log-transformed HAI titers on Days 56, 70, and other follow-up time points.
Time Frame: Day 0 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean Titers
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
Geometric Mean Titers
  Day 0 | 75.9 [65.7 to 87.7] | 67.9 [54.4 to 84.6] | 75.8 [60.7 to 94.7] | 67.6 [54.5 to 83.8] | 62.1 [49.2 to 78.3] | 65.5 [52.3 to 82.1] | 69.5 [59.9 to 80.7] | 65.2 [50.9 to 83.5] | 67.6 [51.3 to 89.1] | 72.7 [56.3 to 93.9] | 75.2 [60.9 to 92.8] | 74.8 [60.1 to 93.1] | 64.6 [51.9 to 80.5]
  Day 28 | 101.5 [88.4 to 116.6] | 84.3 [67.8 to 104.7] | 82.2 [65.0 to 103.9] | 81.5 [64.5 to 103.0] | 83.5 [67.0 to 103.9] | 78.0 [63.0 to 96.6] | 89.4 [75.3 to 106.2] | 73.9 [58.8 to 92.8] | 75.8 [58.9 to 97.7] | 87.4 [68.7 to 111.3] | 88.2 [67.4 to 115.4] | 90.8 [71.3 to 115.7] | 99.9 [80.2 to 124.4]
  Day 56 | 91.7 [79.2 to 106.1] | 83.6 [66.3 to 105.5] | 73.4 [57.6 to 93.4] | 80.8 [64.1 to 101.9] | 70.3 [56.6 to 87.1] | 70.3 [56.0 to 88.1] | 85.4 [72.6 to 100.5] | 70.0 [55.5 to 88.4] | 77.1 [59.8 to 99.6] | 77.8 [61.0 to 99.1] | 82.2 [62.9 to 107.5] | 85.7 [69.0 to 106.6] | 91.4 [72.8 to 114.7]
  Day 70 | 107.2 [92.8 to 123.8] | 89.8 [69.0 to 116.8] | 88.3 [68.6 to 113.7] | 91.5 [71.3 to 117.5] | 85.0 [66.5 to 108.7] | 77.3 [62.1 to 96.1] | 93.4 [79.0 to 110.4] | 75.1 [60.1 to 93.6] | 80.7 [60.9 to 107.0] | 95.1 [76.0 to 119.2] | 92.9 [70.5 to 122.4] | 90.8 [74.3 to 111.1] | 94.3 [73.7 to 120.6]
  Day 84 | 63.5 [53.5 to 75.4] | 62.4 [48.0 to 81.1] | 57.1 [42.5 to 76.8] | 54.9 [41.9 to 72.0] | 58.6 [46.0 to 74.7] | 48.4 [38.8 to 60.5] | 66.1 [54.9 to 79.5] | 48.4 [36.0 to 65.3] | 50.2 [37.6 to 67.1] | 58.3 [43.8 to 77.6] | 67.0 [51.3 to 87.4] | 63.1 [50.0 to 79.7] | 65.5 [49.4 to 86.7]
  Day 182 | 61.2 [51.8 to 72.3] | 52.7 [40.7 to 68.2] | 50.6 [37.4 to 68.4] | 49.7 [37.4 to 66.1] | 48.2 [37.5 to 62.0] | 43.4 [34.2 to 55.1] | 55.8 [46.2 to 67.3] | 45.6 [34.5 to 60.2] | 50.1 [39.2 to 63.9] | 56.0 [43.5 to 72.2] | 51.6 [38.4 to 69.4] | 57.1 [45.0 to 72.3] | 58.7 [44.6 to 77.1]

12. Secondary Outcome: Hemagglutination-Inhibition (HAI) Antibody Titers Specific for the HA Receptor Binding Domains of Vaccine Homologous Influenza A/Brisbane (H1N1 Subtype) Expressed as Geometric Mean Fold Rise (GMFRPost/Pre)
Description: Hemagglutination-inhibition (HAI) antibody titers specific for the HA receptor binding domains of vaccine homologous Influenza A/Brisbane (H1N1 Subtype) calculated as (GMFRPost/Pre), defined as the within-group ratio of post-vaccination to pre-vaccination (Day 0) HAI GMTs within the same vaccine group on Days 56, 70, and other follow-up time points.
Time Frame: Day 28 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean fold rise
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
geometric mean fold rise
  Day 28 | 1.7 [1.4 to 2.0] | 1.4 [1.0 to 1.4] | 1.3 [1.1 to 1.6] | 1.2 [1.0 to 1.4] | 1.3 [1.0 to 1.6] | 1.3 [1.1 to 1.5] | 1.6 [1.4 to 1.8] | 1.2 [1.0 to 1.4] | 1.1 [0.9 to 1.2] | 1.5 [1.2 to 1.8] | 1.3 [1.1 to 1.6] | 1.3 [1.1 to 1.5] | 1.6 [1.3 to 2.0]
  Day 56 | 1.5 [1.3 to 1.8] | 1.3 [1.0 to 1.8] | 1.3 [1.0 to 1.6] | 1.1 [1.0 to 1.2] | 1.1 [1.0 to 1.3] | 1.2 [1.1 to 1.4] | 1.4 [1.2 to 1.6] | 1.1 [0.9 to 1.3] | 1.0 [0.9 to 1.2] | 1.3 [1.0 to 1.6] | 1.1 [0.9 to 1.4] | 1.2 [1.1 to 1.5] | 1.4 [1.1 to 1.8]
  Day 70 | 1.7 [1.4 to 2.1] | 1.9 [1.4 to 2.6] | 1.7 [1.4 to 2.1] | 1.6 [1.3 to 1.9] | 1.5 [1.2 to 1.9] | 1.5 [1.2 to 1.8] | 1.6 [1.4 to 1.9] | 1.4 [1.1 to 1.7] | 1.3 [1.1 to 1.6] | 1.5 [1.2 to 1.9] | 1.5 [1.2 to 1.9] | 1.6 [1.3 to 1.9] | 1.5 [1.2 to 1.8]
  Day 84 | 1.3 [1.0 to 1.6] | 1.3 [0.9 to 1.8] | 1.4 [1.1 to 1.7] | 1.1 [0.9 to 1.3] | 1.1 [0.9 to 1.5] | 0.9 [0.7 to 1.2] | 1.3 [1.1 to 1.5] | 0.8 [0.6 to 1.0] | 1.0 [0.8 to 1.3] | 1.0 [0.8 to 1.2] | 1.1 [0.8 to 1.4] | 1.1 [0.9 to 1.4] | 1.1 [0.8 to 1.5]
  Day 182 | 1.0 [0.8 to 1.3] | 0.9 [0.6 to 1.2] | 1.0 [0.8 to 1.2] | 0.8 [0.7 to 0.9] | 0.8 [0.6 to 1.0] | 0.8 [0.6 to 1.0] | 0.9 [0.7 to 1.0] | 0.6 [0.5 to 0.8] | 0.8 [0.6 to 0.9] | 0.8 [0.6 to 1.0] | 0.8 [0.6 to 1.0] | 0.8 [0.7 to 1.0] | 0.8 [0.6 to 1.0]

13. Secondary Outcome: Hemagglutination-Inhibition (HAI) Antibody Titers Specific for the HA Receptor Binding Domains of Vaccine Homologous Influenza A/Kansas (H3N2 Subtype) Expressed as (GMFRPost/Pre)
Description: Hemagglutination-inhibition (HAI) antibody titers specific for the HA receptor binding domains of vaccine homologous Influenza A/Kansas (H3N2 Subtype) calculated as (GMFRPost/Pre), defined as the within-group ratio of post-vaccination to pre-vaccination (Day 0) HAI GMTs within the same vaccine group on Days 56, 70, and other follow-up time points.
Time Frame: Day 28 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean fold rise
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
geometric mean fold rise
  Day 28 | 4.1 [3.3 to 4.9] | 3.6 [2.3 to 5.5] | 2.7 [2.1 to 3.5] | 2.5 [1.9 to 3.2] | 3.4 [2.4 to 4.7] | 2.7 [2.0 to 3.5] | 4.1 [3.3 to 5.0] | 2.3 [1.8 to 3.0] | 2.2 [1.7 to 2.8] | 4.4 [3.1 to 6.1] | 4.0 [3.2 to 5.0] | 3.6 [2.7 to 4.8] | 5.4 [3.8 to 7.5]
  Day 56 | 3.6 [3.0 to 4.4] | 3.0 [2.0 to 4.4] | 2.9 [2.2 to 3.7] | 2.2 [1.8 to 2.8] | 2.6 [1.9 to 3.6] | 2.2 [1.7 to 2.8] | 3.6 [3.0 to 4.4] | 2.0 [1.6 to 2.6] | 2.1 [1.6 to 2.8] | 3.3 [2.4 to 4.5] | 3.2 [2.5 to 4.1] | 3.2 [2.5 to 4.2] | 4.1 [3.1 to 5.5]
  Day 70 | 4.5 [3.7 to 5.4] | 4.3 [2.9 to 6.4] | 3.8 [2.7 to 5.2] | 3.5 [2.8 to 4.3] | 4.0 [2.9 to 5.4] | 3.3 [2.5 to 4.3] | 4.8 [3.9 to 5.9] | 3.1 [2.4 to 4.0] | 2.7 [2.1 to 3.5] | 4.4 [3.1 to 6.2] | 3.8 [3.0 to 4.7] | 3.7 [2.8 to 4.8] | 4.2 [3.0 to 5.8]
  Day 84 | 4.1 [3.4 to 4.9] | 3.9 [2.7 to 5.6] | 3.9 [3.1 to 5.0] | 2.6 [2.1 to 3.3] | 3.6 [2.6 to 4.9] | 2.8 [2.1 to 3.7] | 4.4 [3.6 to 5.4] | 2.6 [2.1 to 3.2] | 2.5 [1.9 to 3.2] | 3.5 [2.8 to 4.3] | 3.4 [2.7 to 4.3] | 3.4 [2.7 to 4.4] | 3.6 [2.7 to 4.8]
  Day 182 | 3.1 [2.6 to 3.7] | 2.8 [2.0 to 3.9] | 2.8 [2.2 to 3.5] | 1.8 [1.4 to 2.2] | 2.5 [1.9 to 3.2] | 2.2 [1.6 to 3.0] | 3.0 [2.5 to 3.6] | 2.1 [1.7 to 2.6] | 2.1 [1.7 to 2.5] | 2.6 [2.1 to 3.2] | 2.5 [2.0 to 3.1] | 2.8 [2.2 to 3.5] | 2.5 [1.9 to 3.3]

14. Secondary Outcome: Hemagglutination-Inhibition (HAI) Antibody Titers Specific for the HA Receptor Binding Domains of Vaccine Homologous Influenza A/Wisconsin (H1N1 Subtype) Expressed as (GMFRPost/Pre)
Description: Hemagglutination-inhibition (HAI) antibody titers specific for the HA receptor binding domains of vaccine homologous Influenza A/Wisconsin (H1N1 Subtype) calculated as (GMFRPost/Pre), defined as the within-group ratio of post-vaccination to pre-vaccination (Day 0) HAI GMTs within the same vaccine group on Days 56, 70, and other follow-up time points.
Time Frame: Day 28 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean fold rise
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
geometric mean fold rise
  Day 28 | 1.4 [1.3 to 1.6] | 1.3 [1.1 to 1.5] | 1.2 [1.0 to 1.3] | 1.1 [1.0 to 1.2] | 1.4 [1.2 to 1.6] | 1.2 [1.1 to 1.3] | 1.4 [1.2 to 1.5] | 1.1 [1.0 to 1.3] | 1.1 [0.9 to 1.2] | 1.3 [1.1 to 1.5] | 1.2 [1.1 to 1.3] | 1.3 [1.1 to 1.5] | 1.3 [1.1 to 1.5]
  Day 56 | 1.3 [1.2 to 1.5] | 1.1 [0.9 to 1.4] | 1.1 [0.9 to 1.2] | 1.0 [1.0 to 1.2] | 1.1 [1.0 to 1.3] | 1.0 [0.9 to 1.2] | 1.2 [1.0 to 1.3] | 1.1 [0.9 to 1.3] | 1.0 [0.9 to 1.1] | 1.2 [1.0 to 1.4] | 1.1 [1.0 to 1.2] | 1.1 [1.0 to 1.3] | 1.2 [1.0 to 1.4]
  Day 70 | 1.5 [1.3 to 1.8] | 1.3 [1.0 to 1.6] | 1.2 [1.1 to 1.4] | 1.2 [1.1 to 1.4] | 1.5 [1.2 to 1.8] | 1.1 [1.0 to 1.3] | 1.4 [1.2 to 1.5] | 1.3 [1.1 to 1.5] | 1.1 [1.0 to 1.2] | 1.3 [1.1 to 1.6] | 1.2 [1.1 to 1.4] | 1.4 [1.2 to 1.6] | 1.2 [1.0 to 1.4]
  Day 84 | 0.9 [0.8 to 1.0] | 0.8 [0.6 to 1.0] | 0.7 [0.6 to 0.8] | 0.7 [0.6 to 0.8] | 0.9 [0.7 to 1.0] | 0.8 [0.6 to 1.0] | 0.8 [0.7 to 1.0] | 0.7 [0.6 to 0.9] | 0.6 [0.5 to 0.7] | 0.7 [0.5 to 0.9] | 0.7 [0.6 to 0.8] | 0.8 [0.7 to 1.0] | 0.7 [0.6 to 0.8]
  Day 182 | 0.8 [0.6 to 0.9] | 0.6 [0.5 to 0.7] | 0.6 [0.5 to 0.7] | 0.6 [0.5 to 0.7] | 0.7 [0.6 to 0.8] | 0.6 [0.5 to 0.8] | 0.7 [0.6 to 0.7] | 0.6 [0.5 to 0.7] | 0.5 [0.4 to 0.6] | 0.6 [0.5 to 0.8] | 0.6 [0.5 to 0.6] | 0.7 [0.6 to 0.8] | 0.6 [0.5 to 0.7]

15. Secondary Outcome: Hemagglutination-Inhibition (HAI) Antibody Titers Specific for the HA Receptor Binding Domains of Vaccine Homologous Influenza A/Cambodia (H3N2 Subtype) Expressed as (GMFRPost/Pre)
Description: Hemagglutination-inhibition (HAI) antibody titers specific for the HA receptor binding domains of vaccine homologous Influenza A/Cambodia (H3N2 Subtype) calculated as (GMFRPost/Pre), defined as the within-group ratio of post-vaccination to pre-vaccination (Day 0) HAI GMTs within the same vaccine group on Days 56, 70, and other follow-up time points.
Time Frame: Day 28 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean fold rise
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
geometric mean fold rise
  Day 28 | 2.2 [1.9 to 2.6] | 2.2 [1.4 to 3.2] | 1.7 [1.3 to 2.1] | 1.7 [1.3 to 2.0] | 2.2 [1.6 to 3.0] | 1.8 [1.4 to 2.4] | 2.2 [1.9 to 2.6] | 1.6 [1.3 to 2.0] | 1.7 [1.4 to 2.1] | 2.4 [1.8 to 3.3] | 2.4 [1.9 to 3.0] | 1.8 [1.5 to 2.3] | 2.2 [1.7 to 3.0]
  Day 56 | 1.9 [1.6 to 2.3] | 1.9 [1.3 to 2.7] | 1.6 [1.3 to 2.0] | 1.5 [1.2 to 1.9] | 1.8 [1.4 to 2.3] | 1.6 [1.3 to 1.9] | 1.9 [1.6 to 2.2] | 1.5 [1.2 to 1.8] | 1.5 [1.2 to 1.9] | 2.2 [1.6 to 3.1] | 2.0 [1.6 to 2.5] | 1.6 [1.3 to 2.1] | 1.9 [1.5 to 2.5]
  Day 70 | 2.1 [1.8 to 2.5] | 2.2 [1.5 to 3.2] | 1.9 [1.5 to 2.4] | 1.7 [1.4 to 2.1] | 2.2 [1.7 to 3.0] | 1.9 [1.5 to 2.4] | 2.2 [1.8 to 2.5] | 1.9 [1.6 to 2.4] | 1.7 [1.3 to 2.1] | 2.5 [1.8 to 3.5] | 2.1 [1.7 to 2.7] | 1.9 [1.5 to 2.4] | 2.1 [1.6 to 2.6]
  Day 84 | 1.3 [1.1 to 1.5] | 1.6 [1.1 to 2.3] | 1.2 [0.9 to 1.5] | 1.1 [0.8 to 1.4] | 1.4 [1.0 to 1.8] | 1.2 [0.9 to 1.6] | 1.4 [1.2 to 1.7] | 1.2 [1.0 to 1.5] | 1.0 [0.8 to 1.4] | 1.6 [1.2 to 2.2] | 1.6 [1.2 to 1.9] | 1.1 [0.9 to 1.4] | 1.1 [0.9 to 1.4]
  Day 182 | 1.2 [1.0 to 1.4] | 1.3 [0.9 to 1.9] | 0.9 [0.7 to 1.2] | 0.8 [0.6 to 1.0] | 1.1 [0.8 to 1.4] | 0.9 [0.7 to 1.2] | 1.1 [0.9 to 1.3] | 1.0 [0.8 to 1.2] | 1.0 [0.8 to 1.2] | 1.3 [1.0 to 1.7] | 1.1 [0.8 to 1.4] | 0.9 [0.8 to 1.2] | 0.9 [0.7 to 1.2]

16. Secondary Outcome: Hemagglutination-Inhibition (HAI) Antibody Titers Specific for the HA Receptor Binding Domains of Vaccine Homologous Influenza A/Hong Kong (H3N2 Subtype) Expressed as (GMFRPost/Pre)
Description: Hemagglutination-inhibition (HAI) antibody titers specific for the HA receptor binding domains of vaccine homologous Influenza A/Hong Kong (H3N2 Subtype) calculated as (GMFRPost/Pre), defined as the within-group ratio of post-vaccination to pre-vaccination (Day 0) HAI GMTs within the same vaccine group on Days 56, 70, and other follow-up time points.
Time Frame: Day 28 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean fold rise
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
geometric mean fold rise
  Day 28 | 1.9 [1.6 to 2.2] | 1.8 [1.3 to 2.5] | 1.4 [1.2 to 1.7] | 1.4 [1.2 to 1.7] | 1.7 [1.3 to 2.2] | 1.4 [1.2 to 1.7] | 1.9 [1.7 to 2.3] | 1.5 [1.2 to 1.7] | 1.6 [1.4 to 2.0] | 2.1 [1.7 to 2.5] | 1.8 [1.5 to 2.3] | 1.7 [1.4 to 2.1] | 1.9 [1.4 to 2.5]
  Day 56 | 1.7 [1.5 to 2.0] | 1.6 [1.2 to 2.2] | 1.4 [1.2 to 1.6] | 1.3 [1.1 to 1.6] | 1.3 [1.1 to 1.6] | 1.4 [1.2 to 1.6] | 1.8 [1.5 to 2.1] | 1.3 [1.1 to 1.5] | 1.5 [1.2 to 1.7] | 1.7 [1.4 to 2.1] | 1.6 [1.3 to 2.0] | 1.6 [1.3 to 1.9] | 1.6 [1.3 to 2.1]
  Day 70 | 1.9 [1.6 to 2.2] | 2.1 [1.5 to 2.8] | 1.8 [1.4 to 2.2] | 1.6 [1.3 to 2.0] | 1.7 [1.4 to 2.1] | 1.6 [1.3 to 1.9] | 1.9 [1.6 to 2.2] | 1.5 [1.2 to 1.8] | 1.6 [1.3 to 1.9] | 2.0 [1.7 to 2.5] | 1.9 [1.5 to 2.4] | 1.7 [1.4 to 2.1] | 1.8 [1.4 to 2.2]
  Day 84 | 1.2 [1.1 to 1.5] | 1.4 [1.1 to 1.9] | 1.1 [0.9 to 1.5] | 1.1 [0.9 to 1.4] | 1.2 [1.0 to 1.6] | 1.1 [0.9 to 1.4] | 1.5 [1.2 to 1.8] | 1.1 [0.9 to 1.3] | 1.1 [0.8 to 1.4] | 1.5 [1.1 to 2.0] | 1.4 [1.1 to 1.7] | 1.4 [1.1 to 1.8] | 1.2 [0.9 to 1.5]
  Day 182 | 1.0 [0.9 to 1.2] | 1.2 [0.8 to 1.6] | 0.9 [0.7 to 1.1] | 0.9 [0.7 to 1.1] | 1.0 [0.8 to 1.2] | 0.9 [0.7 to 1.2] | 1.1 [0.9 to 1.3] | 0.9 [0.8 to 1.1] | 1.0 [0.8 to 1.2] | 1.2 [1.0 to 1.5] | 1.1 [0.9 to 1.3] | 1.1 [0.8 to 1.4] | 1.0 [0.8 to 1.3]

17. Secondary Outcome: Hemagglutination-Inhibition (HAI) Antibody Titers Specific for the HA Receptor Binding Domains of Vaccine Homologous Influenza B/Maryland (Victoria Subtype) Expressed as (GMFRPost/Pre)
Description: Hemagglutination-inhibition (HAI) antibody titers specific for the HA receptor binding domains of vaccine homologous Influenza B/Maryland (Victoria Subtype) calculated as (GMFRPost/Pre), defined as the within-group ratio of post-vaccination to pre-vaccination (Day 0) HAI GMTs within the same vaccine group on Days 56, 70, and other follow-up time points.
Time Frame: Day 28 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean fold rise
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
geometric mean fold rise
  Day 28 | 1.6 [1.4 to 1.9] | 1.6 [1.3 to 2.0] | 1.1 [0.9 to 1.4] | 1.3 [1.1 to 1.6] | 1.5 [1.2 to 1.9] | 1.3 [1.1 to 1.5] | 1.6 [1.4 to 1.9] | 1.2 [1.0 to 1.3] | 1.2 [1.0 to 1.3] | 1.3 [1.1 to 1.6] | 1.4 [1.1 to 1.7] | 1.4 [1.2 to 1.6] | 1.8 [1.4 to 2.4]
  Day 56 | 1.5 [1.3 to 1.8] | 1.3 [1.1 to 1.6] | 1.2 [1.0 to 1.4] | 1.4 [1.2 to 1.6] | 1.2 [1.0 to 1.5] | 1.2 [1.1 to 1.4] | 1.5 [1.3 to 1.7] | 1.2 [1.0 to 1.3] | 1.1 [1.0 to 1.3] | 1.3 [1.1 to 1.6] | 1.2 [1.0 to 1.4] | 1.3 [1.2 to 1.4] | 1.6 [1.3 to 2.0]
  Day 70 | 1.7 [1.4 to 2.0] | 1.6 [1.3 to 1.9] | 1.3 [1.1 to 1.5] | 1.5 [1.3 to 1.8] | 1.7 [1.4 to 2.0] | 1.4 [1.2 to 1.6] | 1.6 [1.4 to 1.8] | 1.4 [1.2 to 1.6] | 1.3 [1.1 to 1.5] | 1.5 [1.3 to 1.8] | 1.4 [1.2 to 1.7] | 1.5 [1.3 to 1.8] | 1.6 [1.3 to 1.9]
  Day 84 | 1.7 [1.4 to 2.1] | 1.7 [1.4 to 2.0] | 1.5 [1.2 to 1.9] | 1.4 [1.2 to 1.7] | 1.8 [1.4 to 2.2] | 1.6 [1.3 to 1.9] | 1.9 [1.7 to 2.2] | 1.3 [1.1 to 1.5] | 1.3 [1.0 to 1.6] | 1.5 [1.3 to 1.8] | 1.6 [1.3 to 1.9] | 1.6 [1.3 to 1.8] | 1.7 [1.4 to 2.1]
  Day 182 | 1.6 [1.3 to 1.9] | 1.5 [1.2 to 1.7] | 1.3 [1.1 to 1.6] | 1.3 [1.0 to 1.5] | 1.5 [1.2 to 1.8] | 1.3 [1.1 to 1.5] | 1.6 [1.4 to 1.8] | 1.3 [1.1 to 1.5] | 1.3 [1.1 to 1.6] | 1.3 [1.1 to 1.5] | 1.3 [1.1 to 1.5] | 1.3 [1.1 to 1.6] | 1.5 [1.2 to 1.8]

18. Secondary Outcome: Hemagglutination-Inhibition (HAI) Antibody Titers Specific for the HA Receptor Binding Domains of Vaccine Homologous Influenza B/Phuket (Yamagata Subtype) Expressed as (GMFRPost/Pre)
Description: Hemagglutination-inhibition (HAI) antibody titers specific for the HA receptor binding domains of vaccine homologous Influenza B/Phuket (Yamagata Subtype) calculated as (GMFRPost/Pre), defined as the within-group ratio of post-vaccination to pre-vaccination (Day 0) HAI GMTs within the same vaccine group on Days 56, 70, and other follow-up time points.
Time Frame: Day 28 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean fold rise
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
geometric mean fold rise
  Day 28 | 2.0 [1.6 to 2.3] | 1.6 [1.3 to 2.0] | 1.4 [1.1 to 1.7] | 1.4 [1.2 to 1.8] | 1.9 [1.4 to 2.5] | 1.4 [1.1 to 1.7] | 1.9 [1.6 to 2.2] | 1.6 [1.3 to 1.9] | 1.3 [1.1 to 1.5] | 1.6 [1.3 to 2.0] | 1.7 [1.4 to 2.0] | 1.9 [1.6 to 2.4] | 2.7 [2.0 to 3.6]
  Day 56 | 1.8 [1.5 to 2.1] | 1.5 [1.2 to 1.8] | 1.5 [1.2 to 1.8] | 1.3 [1.1 to 1.6] | 1.6 [1.2 to 2.1] | 1.3 [1.1 to 1.6] | 1.7 [1.5 to 1.9] | 1.5 [1.3 to 1.8] | 1.2 [1.0 to 1.4] | 1.5 [1.3 to 1.9] | 1.5 [1.3 to 1.8] | 1.8 [1.5 to 2.2] | 2.3 [1.8 to 3.0]
  Day 70 | 2.3 [1.9 to 2.7] | 2.0 [1.6 to 2.4] | 1.9 [1.5 to 2.3] | 1.8 [1.5 to 2.3] | 2.3 [1.8 to 3.1] | 1.7 [1.4 to 2.0] | 2.1 [1.8 to 2.4] | 1.8 [1.5 to 2.2] | 1.5 [1.3 to 1.7] | 2.0 [1.6 to 2.5] | 1.9 [1.6 to 2.3] | 2.1 [1.7 to 2.5] | 2.3 [1.7 to 3.0]
  Day 84 | 2.2 [1.8 to 2.6] | 2.0 [1.6 to 2.4] | 2.1 [1.8 to 2.6] | 1.8 [1.4 to 2.3] | 2.5 [1.9 to 3.2] | 1.8 [1.4 to 2.2] | 2.3 [2.0 to 2.7] | 1.7 [1.4 to 2.1] | 1.6 [1.3 to 1.9] | 2.2 [1.8 to 2.6] | 2.2 [1.8 to 2.7] | 2.2 [1.8 to 2.6] | 2.4 [1.8 to 3.1]
  Day 182 | 2.0 [1.6 to 2.4] | 1.7 [1.4 to 2.0] | 1.8 [1.5 to 2.2] | 1.6 [1.2 to 2.0] | 2.0 [1.5 to 2.5] | 1.5 [1.2 to 1.9] | 1.8 [1.6 to 2.1] | 1.5 [1.2 to 1.9] | 1.5 [1.3 to 1.7] | 1.7 [1.5 to 2.0] | 1.6 [1.4 to 1.9] | 1.8 [1.5 to 2.3] | 1.8 [1.4 to 2.3]

19. Secondary Outcome: Hemagglutination-Inhibition (HAI) Antibody Titers Specific for the HA Receptor Binding Domains of Vaccine Homologous Influenza B/Washington (Victoria Subtype) Expressed as (GMFRPost/Pre)
Description: Hemagglutination-inhibition (HAI) antibody titers specific for the HA receptor binding domains of vaccine homologous Influenza B/Washington (Victoria Subtype) calculated as (GMFRPost/Pre), defined as the within-group ratio of post-vaccination to pre-vaccination (Day 0) HAI GMTs within the same vaccine group on Days 56, 70, and other follow-up time points.
Time Frame: Day 28 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean fold rise
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
geometric mean fold rise
  Day 28 | 1.3 [1.2 to 1.5] | 1.2 [1.1 to 1.4] | 1.1 [1.0 to 1.2] | 1.2 [1.0 to 1.4] | 1.3 [1.1 to 1.6] | 1.2 [1.0 to 1.4] | 1.3 [1.1 to 1.4] | 1.1 [1.0 to 1.3] | 1.1 [1.0 to 1.3] | 1.2 [1.1 to 1.4] | 1.2 [1.0 to 1.4] | 1.2 [1.1 to 1.4] | 1.5 [1.2 to 2.0]
  Day 56 | 1.2 [1.1 to 1.4] | 1.2 [1.1 to 1.4] | 1.0 [0.9 to 1.1] | 1.2 [1.0 to 1.4] | 1.1 [1.0 to 1.3] | 1.1 [0.9 to 1.2] | 1.2 [1.1 to 1.3] | 1.1 [1.0 to 1.2] | 1.1 [1.0 to 1.2] | 1.1 [1.0 to 1.3] | 1.1 [0.9 to 1.3] | 1.2 [1.1 to 1.3] | 1.4 [1.1 to 1.8]
  Day 70 | 1.4 [1.3 to 1.6] | 1.3 [1.2 to 1.5] | 1.2 [1.0 to 1.4] | 1.3 [1.1 to 1.6] | 1.4 [1.1 to 1.6] | 1.2 [1.0 to 1.4] | 1.3 [1.2 to 1.5] | 1.2 [1.1 to 1.3] | 1.2 [1.0 to 1.3] | 1.4 [1.2 to 1.6] | 1.2 [1.0 to 1.5] | 1.2 [1.1 to 1.4] | 1.5 [1.2 to 1.9]
  Day 84 | 0.9 [0.8 to 1.0] | 0.9 [0.8 to 1.0] | 0.8 [0.7 to 0.9] | 0.8 [0.7 to 1.0] | 0.9 [0.8 to 1.1] | 0.7 [0.6 to 0.9] | 0.9 [0.8 to 1.1] | 0.8 [0.6 to 0.9] | 0.7 [0.6 to 0.9] | 0.9 [0.7 to 1.0] | 0.9 [0.7 to 1.1] | 0.8 [0.7 to 1.0] | 1.0 [0.8 to 1.3]
  Day 182 | 0.8 [0.7 to 0.9] | 0.8 [0.7 to 0.9] | 0.7 [0.6 to 0.8] | 0.7 [0.6 to 0.9] | 0.7 [0.6 to 0.9] | 0.7 [0.5 to 0.8] | 0.8 [0.7 to 0.9] | 0.7 [0.6 to 0.9] | 0.7 [0.6 to 0.9] | 0.8 [0.7 to 1.0] | 0.7 [0.6 to 0.8] | 0.8 [0.7 to 0.9] | 0.9 [0.7 to 1.2]

20. Secondary Outcome: Hemagglutination-Inhibition (HAI) Antibody Titers Specific for the HA Receptor Binding Domains of Vaccine Homologous Influenza A/Brisbane (H1N1 Subtype) Strain Expressed as Seroconversion Rate (SCR)
Description: Hemagglutination-Inhibition (HAI) Antibody titers specific for the HA receptor binding domains of vaccine homologous Influenza A/Brisbane (H1N1 Subtype) strain(s) calculated as SCR defined as the proportion of participants in a given treatment group with either a baseline reciprocal (Day 0) titer of < 10 and a post-vaccination reciprocal titer ≥ 40, or a baseline reciprocal (Day 0) titer of ≥ 10 and a post-vaccination titer ≥ 4-fold higher than the baseline titer as measured on Days 56, 70, and other follow-up time points.
Time Frame: Day 28 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
percentage of participants
  Day 28 | 15.2 [8.1 to 25.0] | 10.0 [2.8 to 23.7] | 5.3 [0.6 to 17.7] | 2.7 [0.1 to 14.2] | 12.2 [4.1 to 26.2] | 5.0 [0.6 to 16.9] | 14.1 [7.3 to 23.8] | 5.1 [0.6 to 17.3] | 0 [0.0 to 9.0] | 12.8 [4.3 to 27.4] | 7.7 [1.6 to 20.9] | 4.9 [0.6 to 16.5] | 15.4 [5.9 to 30.5]
  Day 56 | 12.8 [6.3 to 22.3] | 7.7 [1.6 to 20.9] | 8.3 [1.8 to 22.5] | 0 [0.0 to 9.7] | 5.0 [0.6 to 16.9] | 5.0 [0.6 to 16.9] | 10.1 [4.5 to 19.0] | 5.1 [0.6 to 17.3] | 0 [0.0 to 9.3] | 8.1 [1.7 to 21.9] | 5.3 [0.6 to 17.7] | 5.0 [0.6 to 16.9] | 10.3 [2.9 to 24.2]
  Day 70 | 17.1 [9.4 to 27.5] | 15.4 [5.9 to 30.5] | 17.1 [6.6 to 33.6] | 11.1 [3.1 to 26.1] | 10.0 [2.8 to 23.7] | 7.5 [1.6 to 20.4] | 15.8 [8.4 to 26.0] | 10.5 [2.9 to 24.8] | 5.3 [0.6 to 17.7] | 13.9 [4.7 to 29.5] | 13.5 [4.5 to 28.8] | 17.1 [7.2 to 32.1] | 10.5 [2.9 to 24.8]
  Day 84 | 14.5 [7.5 to 24.4] | 20.5 [9.3 to 36.5] | 11.8 [3.3 to 27.5] | 0 [0.0 to 10.0] | 7.7 [1.6 to 20.9] | 2.6 [0.1 to 13.8] | 14.5 [7.5 to 24.4] | 2.6 [0.1 to 13.8] | 5.3 [0.6 to 17.7] | 5.9 [0.7 to 19.7] | 10.8 [3.0 to 25.4] | 7.3 [1.5 to 19.9] | 7.9 [1.7 to 21.4]
  Day 182 | 10.8 [0.1 to 13.8] | 10.3 [2.9 to 24.2] | 2.9 [0.1 to 15.3] | 0 [0.0 to 10.0] | 2.6 [0.1 to 13.5] | 0 [0.0 to 9.3] | 6.7 [2.2 to 14.9] | 2.7 [0.1 to 14.2] | 0 [0.0 to 9.5] | 0 [0.0 to 9.7] | 5.3 [0.6 to 17.7] | 2.6 [0.1 to 13.5] | 2.6 [0.1 to 13.8]

21. Secondary Outcome: Hemagglutination-Inhibition (HAI) Antibody Titers Specific for the HA Receptor Binding Domains of Vaccine Homologous Influenza A/Kansas (H3N2 Subtype) Strain Expressed as SCR
Description: Hemagglutination-Inhibition (HAI) Antibody titers specific for the HA receptor binding domains of vaccine homologous Influenza A/Kansas (H3N2 Subtype) strain(s) calculated as SCR defined as the proportion of participants in a given treatment group with either a baseline reciprocal (Day 0) titer of < 10 and a post-vaccination reciprocal titer ≥ 40, or a baseline reciprocal (Day 0) titer of ≥ 10 and a post-vaccination titer ≥ 4-fold higher than the baseline titer as measured on Days 56, 70, and other follow-up time points.
Time Frame: Day 28 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
percentage of participants
  Day 28 | 63.3 [51.7 to 73.9] | 45.0 [29.3 to 61.5] | 42.1 [26.3 to 59.2] | 37.8 [22.5 to 55.2] | 51.2 [35.1 to 67.1] | 37.5 [22.7 to 54.2] | 56.4 [44.7 to 67.6] | 33.3 [19.1 to 50.2] | 28.2 [15.0 to 44.9] | 51.3 [34.8 to 67.6] | 61.5 [44.6 to 76.6] | 51.2 [35.1 to 67.1] | 69.2 [52.4 to 83.0]
  Day 56 | 60.3 [48.5 to 71.2] | 38.5 [23.4 to 55.4] | 41.7 [25.5 to 59.2] | 27.8 [14.2 to 45.2] | 37.5 [22.7 to 54.2] | 30.0 [16.6 to 46.5] | 51.9 [40.4 to 63.3] | 25.6 [13.0 to 42.1] | 26.3 [13.4 to 43.1] | 45.9 [29.5 to 63.1] | 44.7 [28.6 to 61.7] | 45.0 [29.3 to 61.5] | 61.5 [44.6 to 76.6]
  Day 70 | 71.1 [59.5 to 80.9] | 53.8 [37.2 to 69.9] | 54.3 [36.6 to 71.2] | 61.1 [43.5 to 76.9] | 67.5 [50.9 to 81.4] | 47.5 [31.5 to 63.9] | 65.8 [54.0 to 76.3] | 52.6 [35.8 to 69.0] | 39.5 [24.0 to 56.6] | 55.6 [38.1 to 72.1] | 64.9 [47.5 to 79.8] | 56.1 [39.7 to 71.5] | 57.9 [40.8 to 73.7]
  Day 84 | 67.5 [55.9 to 77.8] | 46.2 [30.1 to 62.8] | 52.9 [35.1 to 70.2] | 42.9 [26.3 to 60.6] | 53.8 [37.2 to 69.9] | 42.1 [26.3 to 59.2] | 65.8 [54.0 to 76.3] | 39.5 [24.0 to 56.6] | 36.8 [21.8 to 54.0] | 58.8 [40.7 to 75.4] | 54.1 [36.9 to 70.5] | 51.2 [35.1 to 67.1] | 52.6 [35.8 to 69.0]
  Day 182 | 39.2 [28.0 to 51.2] | 33.3 [19.1 to 50.2] | 41.2 [24.6 to 59.3] | 20.0 [8.4 to 36.9] | 38.5 [23.4 to 55.4] | 28.9 [15.4 to 45.9] | 46.7 [35.1 to 58.7] | 21.6 [9.8 to 38.2] | 21.6 [9.8 to 38.2] | 38.9 [23.1 to 56.5] | 28.9 [15.4 to 45.9] | 43.6 [27.8 to 60.4] | 34.2 [19.6 to 51.4]

22. Secondary Outcome: Hemagglutination-Inhibition (HAI) Antibody Titers Specific for the HA Receptor Binding Domains of Vaccine Homologous Influenza A/Wisconsin (H1N1 Subtype) Strain Expressed as SCR
Description: Hemagglutination-Inhibition (HAI) Antibody titers specific for the HA receptor binding domains of vaccine homologous Influenza A/Wisconsin (H1N1 Subtype) strain(s) calculated as SCR defined as the proportion of participants in a given treatment group with either a baseline reciprocal (Day 0) titer of < 10 and a post-vaccination reciprocal titer ≥ 40, or a baseline reciprocal (Day 0) titer of ≥ 10 and a post-vaccination titer ≥ 4-fold higher than the baseline titer as measured on Days 56, 70, and other follow-up time points.
Time Frame: Day 28 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
percentage of participants
  Day 28 | 10.1 [4.5 to 19.0] | 5.0 [0.6 to 16.9] | 2.6 [0.1 to 13.8] | 0 [0.0 to 9.5] | 4.9 [0.6 to 16.5] | 2.6 [0.1 to 13.5] | 9.0 [3.7 to 17.6] | 2.6 [0.1 to 13.5] | 0 [0.0 to 9.0] | 5.1 [0.6 to 17.3] | 2.6 [0.1 to 13.5] | 2.4 [0.1 to 12.9] | 5.1 [0.6 to 17.3]
  Day 56 | 6.4 [2.1 to 14.3] | 5.1 [0.6 to 17.3] | 0 [0.0 to 9.7] | 0 [0.0 to 9.7] | 2.5 [0.1 to 13.2] | 0 [0.0 to 8.8] | 5.1 [1.4 to 12.5] | 2.6 [0.1 to 13.5] | 0 [0.0 to 9.3] | 2.7 [0.1 to 14.2] | 2.6 [0.1 to 13.8] | 0 [0.0 to 8.8] | 5.1 [0.6 to 17.3]
  Day 70 | 9.2 [3.8 to 18.1] | 7.7 [1.6 to 20.9] | 0 [0.0 to 10.0] | 0 [0.0 to 9.7] | 7.5 [1.6 to 20.4] | 0 [0.0 to 8.8] | 6.6 [2.2 to 14.7] | 5.3 [0.6 to 17.7] | 0 [0.0 to 9.3] | 5.6 [0.7 to 18.7] | 2.7 [0.1 to 14.2] | 2.4 [0.1 to 12.9] | 5.3 [0.6 to 17.7]
  Day 84 | 3.9 [0.8 to 11.0] | 5.1 [0.6 to 17.3] | 0 [0.0 to 10.3] | 0 [0.0 to 10.0] | 2.6 [0.1 to 13.5] | 2.6 [0.1 to 13.8] | 2.6 [0.3 to 9.2] | 2.6 [0.1 to 13.8] | 0 [0.0 to 9.3] | 2.9 [0.1 to 15.3] | 0 [0.0 to 9.5] | 0 [0.0 to 8.6] | 2.6 [0.1 to 13.8]
  Day 182 | 2.7 [0.3 to 9.4] | 2.6 [0.1 to 13.5] | 0 [0.0 to 10.3] | 0 [0.0 to 10.0] | 2.6 [0.1 to 13.5] | 2.6 [0.1 to 13.8] | 2.7 [0.3 to 9.3] | 0 [0.0 to 9.5] | 0 [0.0 to 9.5] | 2.8 [0.1 to 14.5] | 0 [0.0 to 9.3] | 0 [0.0 to 9.0] | 2.6 [0.1 to 13.8]

23. Secondary Outcome: HAI Antibody Titers Specific for the HA Receptor Binding Domains of Vaccine Homologous Influenza A/Cambodia (H3N2 Subtype) Strain Expressed as SCR
Description: HAI antibody titers specific for the HA receptor binding domains of vaccine homologous Influenza A/Cambodia (H3N2 Subtype) strain(s) calculated as SCR defined as the proportion of participants in a given treatment group with either a baseline reciprocal (Day 0) titer of < 10 and a post-vaccination reciprocal titer ≥ 40, or a baseline reciprocal (Day 0) titer of ≥ 10 and a post-vaccination titer ≥ 4-fold higher than the baseline titer as measured on Days 56, 70, and other follow-up time points.
Time Frame: Day 28 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
percentage of participants
  Day 28 | 30.4 [20.5 to 41.8] | 22.5 [10.8 to 38.5] | 23.7 [11.4 to 40.2] | 13.5 [4.5 to 28.8] | 26.8 [14.2 to 42.9] | 20.0 [9.1 to 35.6] | 28.2 [18.6 to 39.5] | 12.8 [4.3 to 27.4] | 15.4 [5.9 to 30.5] | 41.0 [25.6 to 57.9] | 30.8 [17.0 to 47.6] | 19.5 [8.8 to 34.9] | 30.8 [17.0 to 47.6]
  Day 56 | 23.1 [14.3 to 34.0] | 17.9 [7.5 to 33.5] | 19.4 [8.2 to 36.0] | 11.1 [3.1 to 26.1] | 15.0 [5.7 to 29.8] | 12.5 [4.2 to 26.8] | 20.3 [12.0 to 30.8] | 10.3 [2.9 to 24.2] | 13.2 [4.4 to 28.1] | 35.1 [20.2 to 52.5] | 26.3 [13.4 to 43.1] | 15.0 [5.7 to 29.8] | 23.1 [11.1 to 39.3]
  Day 70 | 27.6 [18.0 to 39.1] | 30.8 [17.0 to 47.6] | 25.7 [12.5 to 43.3] | 13.9 [4.7 to 29.5] | 25.0 [12.7 to 41.2] | 22.5 [10.8 to 38.5] | 28.9 [19.1 to 40.5] | 18.4 [7.7 to 34.3] | 15.8 [6.0 to 31.3] | 36.1 [20.8 to 53.8] | 27.0 [13.8 to 44.1] | 17.1 [7.2 to 32.1] | 21.1 [9.6 to 37.3]
  Day 84 | 14.3 [7.4 to 24.1] | 15.4 [5.9 to 30.5] | 8.8 [1.9 to 23.7] | 5.7 [0.7 to 19.2] | 12.8 [4.3 to 27.4] | 13.2 [4.4 to 28.1] | 15.8 [8.4 to 26.0] | 13.2 [4.4 to 28.1] | 10.5 [2.9 to 24.8] | 23.5 [10.7 to 41.2] | 13.5 [4.5 to 28.8] | 12.2 [4.1 to 26.2] | 10.5 [2.9 to 24.8]
  Day 182 | 10.8 [4.8 to 20.2] | 17.9 [7.5 to 33.5] | 8.8 [1.9 to 23.7] | 5.7 [0.7 to 19.2] | 5.1 [0.6 to 17.3] | 10.5 [2.9 to 24.8] | 9.3 [3.8 to 18.3] | 5.4 [0.7 to 18.2] | 8.1 [1.7 to 21.9] | 11.1 [3.1 to 26.1] | 5.3 [0.6 to 17.7] | 5.1 [0.6 to 17.3] | 7.9 [1.7 to 21.4]

24. Secondary Outcome: HAI Antibody Titers Specific for the HA Receptor Binding Domains of Vaccine Homologous Influenza A/Hong Kong (H3N2 Subtype) Strain Expressed as SCR
Description: HAI antibody titers specific for the HA receptor binding domains of vaccine homologous Influenza A/Hong Kong (H3N2 Subtype)strain(s) calculated as SCR defined as the proportion of participants in a given treatment group with either a baseline reciprocal (Day 0) titer of < 10 and a post-vaccination reciprocal titer ≥ 40, or a baseline reciprocal (Day 0) titer of ≥ 10 and a post-vaccination titer ≥ 4-fold higher than the baseline titer as measured on Days 56, 70, and other follow-up time points.
Time Frame: Day 28 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
percentage of participants
  Day 28 | 21.5 [13.1 to 32.2] | 22.5 [10.8 to 38.5] | 13.2 [4.4 to 28.1] | 10.8 [3.0 to 25.4] | 17.1 [7.2 to 32.1] | 5.0 [0.6 to 16.9] | 25.6 [16.4 to 36.8] | 7.7 [1.6 to 20.9] | 17.9 [7.5 to 33.5] | 28.2 [15.0 to 44.9] | 25.6 [13.0 to 42.1] | 17.1 [7.2 to 32.1] | 20.5 [9.3 to 36.5]
  Day 56 | 19.2 [11.2 to 29.7] | 20.5 [9.3 to 36.5] | 13.9 [4.7 to 29.5] | 8.3 [1.8 to 22.5] | 10.0 [2.8 to 23.7] | 7.5 [1.6 to 20.4] | 19.0 [11.0 to 29.4] | 7.7 [1.6 to 20.9] | 10.5 [2.9 to 24.8] | 18.9 [8.0 to 35.2] | 10.5 [2.9 to 24.8] | 12.5 [4.2 to 26.8] | 15.4 [5.9 to 30.5]
  Day 70 | 25.0 [15.8 to 36.3] | 23.1 [11.1 to 39.3] | 17.1 [6.6 to 33.6] | 11.1 [3.1 to 26.1] | 12.5 [4.2 to 26.8] | 12.5 [4.2 to 26.8] | 21.1 [12.5 to 31.9] | 13.2 [4.4 to 28.1] | 18.4 [7.7 to 34.3] | 27.8 [14.2 to 45.2] | 18.9 [8.0 to 35.2] | 12.2 [4.1 to 26.2] | 13.2 [4.4 to 28.1]
  Day 84 | 11.7 [5.5 to 21.0] | 15.4 [5.9 to 30.5] | 11.8 [3.3 to 27.5] | 5.7 [0.7 to 19.2] | 10.3 [2.9 to 24.2] | 5.3 [0.6 to 17.7] | 15.8 [8.4 to 26.0] | 5.3 [0.6 to 17.7] | 10.5 [2.9 to 24.8] | 20.6 [8.7 to 37.9] | 13.5 [4.5 to 28.8] | 9.8 [2.7 to 23.1] | 13.2 [4.4 to 28.1]
  Day 182 | 6.8 [2.2 to 15.1] | 12.8 [4.3 to 27.4] | 5.9 [0.7 to 19.7] | 5.7 [0.7 to 19.2] | 5.1 [0.6 to 17.3] | 5.3 [0.6 to 17.7] | 9.3 [3.8 to 18.3] | 0 [0.0 to 9.5] | 0 [0.0 to 9.5] | 8.3 [1.8 to 22.5] | 2.6 [0.1 to 13.8] | 7.7 [1.6 to 20.9] | 10.5 [2.9 to 24.8]

25. Secondary Outcome: HAI Antibody Titers Specific for the HA Receptor Binding Domains of Vaccine Homologous Influenza B/Maryland (Victoria Subtype) Strain Expressed as SCR
Description: HAI antibody titers specific for the HA receptor binding domains of vaccine homologous Influenza B/Maryland (Victoria Subtype) strain(s) calculated as SCR defined as the proportion of participants in a given treatment group with either a baseline reciprocal (Day 0) titer of < 10 and a post-vaccination reciprocal titer ≥ 40, or a baseline reciprocal (Day 0) titer of ≥ 10 and a post-vaccination titer ≥ 4-fold higher than the baseline titer as measured on Days 56, 70, and other follow-up time points.
Time Frame: Day 28 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
percentage of participants
  Day 28 | 11.4 [5.3 to 20.5] | 17.5 [7.3 to 32.8] | 5.3 [0.6 to 17.7] | 5.4 [0.7 to 18.2] | 4.9 [0.6 to 16.5] | 5.0 [0.6 to 16.9] | 14.1 [7.3 to 23.8] | 0 [0.0 to 9.0] | 5.1 [0.6 to 17.3] | 10.3 [2.9 to 24.2] | 7.7 [1.6 to 20.9] | 4.9 [0.6 to 16.5] | 20.5 [9.3 to 36.5]
  Day 56 | 12.8 [6.3 to 22.3] | 7.7 [1.6 to 20.9] | 0 [0.0 to 9.7] | 2.8 [0.1 to 14.5] | 2.5 [0.1 to 13.2] | 5.0 [0.6 to 16.9] | 10.1 [4.5 to 19.0] | 0 [0.0 to 9.0] | 2.6 [0.1 to 13.8] | 5.4 [0.7 to 18.2] | 5.3 [0.6 to 17.7] | 0 [0.0 to 8.8] | 15.4 [5.9 to 30.5]
  Day 70 | 15.8 [8.4 to 26.0] | 12.8 [4.3 to 27.4] | 2.9 [0.1 to 14.9] | 8.3 [1.8 to 22.5] | 10.0 [2.8 to 23.7] | 7.5 [1.6 to 20.4] | 14.5 [7.5 to 24.4] | 2.6 [0.1 to 13.8] | 7.9 [1.7 to 21.4] | 8.3 [1.8 to 22.5] | 5.4 [0.7 to 18.2] | 7.3 [1.5 to 19.9] | 10.5 [2.9 to 24.8]
  Day 84 | 22.1 [13.4 to 33.0] | 12.8 [4.3 to 27.4] | 11.8 [3.3 to 27.5] | 8.6 [1.8 to 23.1] | 17.9 [7.5 to 33.5] | 7.9 [1.7 to 21.4] | 19.7 [11.5 to 30.5] | 2.6 [0.1 to 13.8] | 10.5 [2.9 to 24.8] | 11.8 [3.3 to 27.5] | 8.1 [1.7 to 21.9] | 4.9 [0.6 to 16.5] | 13.2 [4.4 to 28.1]
  Day 182 | 16.2 [8.7 to 26.6] | 10.3 [2.9 to 24.2] | 5.9 [0.7 to 19.7] | 8.6 [1.8 to 23.1] | 7.7 [1.6 to 20.9] | 2.6 [0.1 to 13.8] | 16.0 [8.6 to 26.3] | 0 [0.0 to 9.5] | 5.4 [0.7 to 18.2] | 0 [0.0 to 9.7] | 2.6 [0.1 to 13.8] | 2.6 [0.1 to 13.5] | 13.2 [4.4 to 28.1]

26. Secondary Outcome: HAI Antibody Titers Specific for the HA Receptor Binding Domains of Vaccine Homologous Influenza B/Phuket (Yamagata Subtype) Strain Expressed as SCR
Description: HAI antibody titers specific for the HA receptor binding domains of vaccine homologous Influenza B/Phuket (Yamagata Subtype) strain(s) calculated as SCR defined as the proportion of participants in a given treatment group with either a baseline reciprocal (Day 0) titer of < 10 and a post-vaccination reciprocal titer ≥ 40, or a baseline reciprocal (Day 0) titer of ≥ 10 and a post-vaccination titer ≥ 4-fold higher than the baseline titer as measured on Days 56, 70, and other follow-up time points.
Time Frame: Day 28 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
percentage of participants
  Day 28 | 20.3 [12.0 to 30.8] | 22.5 [10.8 to 38.5] | 2.6 [0.1 to 13.8] | 5.4 [0.7 to 18.2] | 22.0 [10.6 to 37.6] | 10.0 [2.8 to 23.7] | 17.9 [10.2 to 28.3] | 10.3 [2.9 to 24.2] | 10.3 [2.9 to 24.2] | 12.8 [4.3 to 27.4] | 15.4 [5.9 to 30.5] | 22.0 [10.6 to 37.6] | 43.6 [27.8 to 60.4]
  Day 56 | 16.7 [9.2 to 26.8] | 15.4 [5.9 to 30.5] | 5.6 [0.7 to 18.7] | 5.6 [0.7 to 18.7] | 10.0 [2.8 to 23.7] | 7.5 [1.6 to 20.4] | 11.4 [5.3 to 20.5] | 7.7 [1.6 to 20.9] | 2.6 [0.1 to 13.8] | 8.1 [1.7 to 21.9] | 10.5 [2.9 to 24.8] | 17.5 [7.3 to 32.8] | 38.5 [23.4 to 55.4]
  Day 70 | 25.0 [15.8 to 36.3] | 25.6 [13.0 to 42.1] | 17.1 [6.6 to 33.6] | 11.1 [3.1 to 26.1] | 37.5 [22.7 to 54.2] | 10.0 [2.8 to 23.7] | 21.1 [12.5 to 31.9] | 7.9 [1.7 to 21.4] | 7.9 [1.7 to 21.4] | 22.2 [10.1 to 39.2] | 13.5 [4.5 to 28.8] | 24.4 [12.4 to 40.3] | 34.2 [19.6 to 51.4]
  Day 84 | 29.9 [20.0 to 41.4] | 30.8 [17.0 to 47.6] | 17.6 [6.8 to 34.5] | 20.0 [8.4 to 36.9] | 33.3 [19.1 to 50.2] | 13.2 [4.4 to 28.1] | 34.2 [23.7 to 46.0] | 18.4 [7.7 to 34.3] | 7.9 [1.7 to 21.4] | 26.5 [12.9 to 44.4] | 27.0 [13.8 to 44.1] | 22.0 [10.6 to 37.6] | 42.1 [26.3 to 59.2]
  Day 182 | 20.3 [11.8 to 31.2] | 17.9 [7.5 to 33.5] | 11.8 [3.3 to 27.5] | 11.4 [3.2 to 26.7] | 17.9 [7.5 to 33.5] | 10.5 [2.9 to 24.8] | 18.7 [10.6 to 29.3] | 16.2 [6.2 to 32.0] | 5.4 [0.7 to 18.2] | 11.1 [3.1 to 26.1] | 7.9 [1.7 to 21.4] | 12.8 [4.3 to 27.4] | 21.1 [9.6 to 37.3]

27. Secondary Outcome: HAI Antibody Titers Specific for the HA Receptor Binding Domains of Vaccine Homologous Influenza B/Washington (Victoria Subtype) Strain Expressed as SCR
Description: HAI antibody titers specific for the HA receptor binding domains of vaccine homologous Influenza B/Washington (Victoria Subtype) calculated as SCR defined as the proportion of participants in a given treatment group with either a baseline reciprocal (Day 0) titer of < 10 and a post-vaccination reciprocal titer ≥ 40, or a baseline reciprocal (Day 0) titer of ≥ 10 and a post-vaccination titer ≥ 4-fold higher than the baseline titer as measured on Days 56, 70, and other follow-up time points.
Time Frame: Day 28 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
percentage of participants
  Day 28 | 5.1 [1.4 to 12.5] | 0 [0.0 to 8.8] | 0 [0.0 to 9.3] | 2.7 [0.1 to 14.2] | 4.9 [0.6 to 16.5] | 5.0 [0.6 to 16.9] | 6.4 [2.1 to 14.3] | 2.6 [0.1 to 13.5] | 2.6 [0.1 to 13.5] | 2.6 [0.1 to 13.5] | 7.7 [1.6 to 20.9] | 4.9 [0.6 to 16.5] | 15.4 [5.9 to 30.5]
  Day 56 | 6.4 [2.1 to 14.3] | 0 [0.0 to 9.0] | 0 [0.0 to 9.7] | 2.8 [0.1 to 14.5] | 2.5 [0.1 to 13.2] | 2.5 [0.1 to 13.2] | 3.8 [0.8 to 10.7] | 0 [0.0 to 9.0] | 2.6 [0.1 to 13.8] | 3.8 [0.1 to 14.2] | 2.6 [0.1 to 13.8] | 0 [0.0 to 8.8] | 15.4 [5.9 to 30.5]
  Day 70 | 6.6 [2.2 to 14.7] | 0 [0.0 to 9.0] | 0 [0.0 to 10.0] | 2.8 [0.1 to 14.5] | 7.5 [1.6 to 20.4] | 5.0 [0.6 to 16.9] | 5.3 [1.5 to 12.9] | 0 [0.0 to 9.3] | 0 [0.0 to 9.3] | 2.8 [0.1 to 14.5] | 8.1 [1.7 to 21.9] | 0 [0.0 to 8.6] | 13.2 [4.4 to 28.1]
  Day 84 | 1.3 [0.0 to 7.0] | 0 [0.0 to 9.0] | 0 [0.0 to 10.3] | 2.9 [0.1 to 14.9] | 2.6 [0.1 to 13.5] | 0 [0.0 to 9.3] | 1.3 [0.0 to 7.1] | 0 [0.0 to 9.3] | 2.6 [0.1 to 13.8] | 0 [0.0 to 10.3] | 2.7 [0.1 to 14.2] | 0 [0.0 to 8.6] | 7.9 [1.7 to 21.4]
  Day 182 | 2.7 [0.3 to 9.4] | 0 [0.0 to 9.0] | 0 [0.0 to 10.3] | 2.9 [0.1 to 14.9] | 2.6 [0.1 to 13.5] | 0 [0.0 to 9.3] | 0 [0.0 to 4.8] | 0 [0.0 to 9.5] | 2.7 [0.1 to 14.2] | 0 [0.0 to 9.7] | 2.6 [0.1 to 13.8] | 0 [0.0 to 9.0] | 5.3 [0.6 to 17.7]

28. Secondary Outcome: HAI Antibody Titers Specific for the HA Receptor Binding Domains of Vaccine Homologous Influenza A/Brisbane (H1N1 Subtype) Expressed as Geometric Mean Titer Ratio (GMTR)
Description: GMT ratio (GMTR) between select treatment arms at Days 28,56, 70, and other follow-up time points post-vaccination (adjusted for intergroup variation in baseline [pre-vaccination] titers)
Time Frame: Day 28 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric mean titer ratio
Groups:
- Group A and Group C - ICC Vaccine Formulation: 2 doses of Formulation 1. 1 dose each on Days 0 and Day 56. ...
- Group B -ICC Vaccine Formulation: 2 doses of Formulation 2. 1 dose each on Days 0 and Day 56. ...
- Group D - ICC Vaccine Formulation: 2 doses of Formulation 3. 1 dose each on Days 0 and Day 56. ...
- Group E - ICC Vaccine Formulation: 2 doses of Formulation 4. 1 dose each on Days 0 and Day 56. ...
- Group F- ICC Vaccine Formulation: 2 doses of Formulation 5. 1 dose each on Days 0 and Day 56. ...
- Group G- ICC Vaccine Formulation: 2 doses of Formulation 6. 1 dose each on Days 0 and Day 56. ...
- Group H and Group N- ICC Vaccine Formulation: 2 doses of Formulation 7. 1 dose each on Day 0 and Day 56. ...
- Group I- ICC Vaccine Formulation: 2 doses of Formulation 8. 1 dose each on Days 0 and Day 56. ...
- Group J -ICC Vaccine Formulation: 2 doses of Formulation 9. 1 dose each on Days 0 and Day 56. ...
- Group K - ICC Vaccine Formulation: 2 doses of Formulation 10. 1 dose each on Days 0 and Day 56. ...
- Group L - ICC Vaccine Formulation: 2 doses of Formulation 11. 1 dose each on Days 0 and Day 56. ...
- Group M -ICC Vaccine Formulation: 2 doses of Formulation 12. 1 dose each on Days 0 and Day 56. ...
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41
Geometric mean titer ratio
  Day 28 (Comparison to qNIV Reference [Group O] Day 28) | 1.04 [0.81 to 1.34] | 0.77 [0.55 to 1.07] | 0.73 [0.58 to 0.91] | 0.76 [0.61 to 0.94] | 0.83 [0.64 to 1.07] | 0.80 [0.64 to 1.01] | 0.98 [0.79 to 1.21] | 0.75 [0.59 to 0.96] | 0.65 [0.52 to 0.81] | 0.97 [0.76 to 1.25] | 0.87 [0.69 to 1.10] | 0.78 [0.63 to 0.98]
  Day 56 (Comparison to qNIV Reference [Group O] Day 56) | 1.08 [0.86 to 1.36] | 0.83 [0.61 to 1.13] | 0.83 [0.65 to 1.07] | 0.80 [0.65 to 0.99] | 0.81 [0.65 to 1.02] | 0.85 [0.68 to 1.06] | 0.95 [0.77 to 1.16] | 0.76 [0.60 to 0.97] | 0.68 [0.54 to 0.86] | 0.94 [0.72 to 1.23] | 0.83 [0.64 to 1.07] | 0.87 [0.69 to 1.08]
  Day 70 (Comparison to qNIV Reference [Group O] Day 70) | 1.22 [0.96 to 1.54] | 1.16 [0.85 to 1.58] | 1.09 [0.85 to 1.39] | 1.11 [0.87 to 1.42] | 1.08 [0.83 to 1.41] | 0.98 [0.80 to 1.21] | 1.11 [0.90 to 1.36] | 0.97 [0.78 to 1.22] | 0.85 [0.68 to 1.06] | 1.15 [0.90 to 1.46] | 1.09 [0.84 to 1.41] | 1.09 [0.89 to 1.34]
  Day 84 (Comparison to qNIV Reference [Group O] Day 84) | 1.17 [0.88 to 1.54] | 1.03 [0.72 to 1.48] | 1.17 [0.88 to 1.56] | 1.03 [0.79 to 1.35] | 1.07 [0.77 to 1.49] | 0.81 [0.60 to 1.09] | 1.14 [0.88 to 1.47] | 0.79 [0.60 to 1.04] | 0.87 [0.66 to 1.15] | 0.99 [0.73 to 1.36] | 1.08 [0.77 to 1.50] | 1.00 [0.75 to 1.32]
  Day 182 (Comparison to qNIV Reference [Group O] Day 182) | 1.28 [0.95 to 1.72] | 0.96 [0.65 to 1.40] | 1.18 [0.89 to 1.57] | 1.03 [0.78 to 1.35] | 1.01 [0.74 to 1.36] | 0.98 [0.72 to 1.31] | 1.07 [0.82 to 1.39] | 0.84 [0.63 to 1.11] | 0.92 [0.70 to 1.21] | 1.06 [0.76 to 1.49] | 1.02 [0.75 to 1.39] | 1.00 [0.75 to 1.35]
  Day70 (Comparison to qNIV Reference [Group O] Day 28)** | 1.09 [0.86 to 1.39] | 1.04 [0.76 to 1.42] | 0.98 [0.76 to 1.26] | 1.00 [0.78 to 1.30] | 0.98 [0.75 to 1.28] | 0.89 [0.71 to 1.11] | 1.00 [0.81 to 1.23] | 0.88 [0.70 to 1.11] | 0.77 [0.61 to 0.97] | 1.04 [0.81 to 1.33] | 0.99 [0.75 to 1.29] | 0.98 [0.79 to 1.22]

29. Secondary Outcome: HAI Antibody Titers Specific for the HA Receptor Binding Domains of Vaccine Homologous Influenza A/Kansas (H3N2 Subtype) Expressed as GMTR
Description: as for outcome 28
Time Frame: Day 28 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric mean titer ratio
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41
Geometric mean titer ratio
  Day 28 (Comparison to qNIV Reference [Group O] Day 28) | 0.76 [0.54 to 1.07] | 0.67 [0.40 to 1.12] | 0.48 [0.32 to 0.72] | 0.48 [0.32 to 0.71] | 0.69 [0.44 to 1.06] | 0.52 [0.35 to 0.77] | 0.74 [0.52 to 1.06] | 0.47 [0.32 to 0.69] | 0.46 [0.31 to 0.68] | 0.81 [0.51 to 1.28] | 0.75 [0.52 to 1.09] | 0.70 [0.47 to 1.05]
  Day 56 (Comparison to qNIV Reference [Group O] Day 56) | 0.88 [0.64 to 1.23] | 0.72 [0.45 to 1.15] | 0.67 [0.46 to 0.99] | 0.56 [0.39 to 0.80] | 0.67 [0.45 to 1.00] | 0.56 [0.39 to 0.79] | 0.87 [0.63 to 1.19] | 0.53 [0.37 to 0.75] | 0.59 [0.41 to 0.84] | 0.80 [0.53 to 1.20] | 0.79 [0.55 to 1.14] | 0.81 [0.64 to 1.23]
  Day 70 (Comparison to qNIV Reference [Group O] Day 70) | 1.06 [0.77 to 1.45] | 1.01 [0.63 to 1.63] | 0.83 [0.53 to 1.29] | 0.87 [0.60 to 1.25] | 1.01 [0.67 to 1.52] | 0.81 [0.56 to 1.18] | 1.12 [0.81 to 1.55] | 0.80 [0.56 to 1.16] | 0.73 [0.50 to 1.06] | 1.03 [0.66 to 1.61] | 0.92 [0.64 to 1.33] | 0.92 [0.62 to 1.35]
  Day 84 (Comparison to qNIV Reference [Group O] Day 84) | 1.12 [0.83 to 1.51] | 1.07 [0.70 to 1.63] | 1.01 [0.71 to 1.45] | 0.78 [0.56 to 1.09] | 1.09 [0.75 to 1.57] | 0.83 [0.57 to 1.18] | 1.19 [0.88 to 1.59] | 0.78 [0.56 to 1.08] | 0.78 [0.55 to 1.11] | 0.95 [0.67 to 1.35] | 0.98 [0.70 to 1.37] | 0.99 [0.83 to 1.51]
  Day 182 (Comparison to qNIV Reference [Group O] Day 182) | 1.24 [0.93 to 1.65] | 1.11 [0.74 to 1.67] | 1.05 [0.73 to 1.49] | 0.76 [0.56 to 1.03] | 1.09 [0.78 to 1.52] | 0.92 [0.64 to 1.32] | 1.16 [0.87 to 1.55] | 0.89 [0.65 to 1.22] | 0.96 [0.70 to 1.30] | 1.04 [0.75 to 1.44] | 1.01 [0.73 to 1.39] | 1.14 [0.82 to 1.59]
  Day70 (Comparison to qNIV Reference [Group O] Day 28)** | 0.83 [0.61 to 1.15] | 0.80 [0.49 to 1.29] | 0.64 [0.41 to 1.00] | 0.69 [0.47 to 1.00] | 0.80 [0.53 to 1.21] | 0.64 [0.44 to 0.94] | 0.88 [0.64 to 1.22] | 0.64 [0.44 to 0.93] | 0.58 [0.39 to 0.86] | 0.81 [0.52 to 1.27] | 0.73 [0.50 to 1.06] | 0.73 [0.49 to 1.07]

30. Secondary Outcome: HAI Antibody Titers Specific for the HA Receptor Binding Domains of Vaccine Homologous Influenza A/Wisconsin (H1N1 Subtype) Expressed as GMTR
Description: as for outcome 28
Time Frame: Day 28 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric mean titer ratio
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41
Geometric mean titer ratio
  Day 28 (Comparison to qNIV Reference [Group O] Day 28) | 1.07 [0.89 to 1.29] | 0.89 [0.72 to 1.11] | 0.83 [0.68 to 1.00] | 0.84 [0.71 to 1.00] | 0.99 [0.83 to 1.17] | 0.89 [0.75 to 1.06] | 1.02 [0.86 to 1.21] | 0.82 [0.68 to 0.99] | 0.82 [0.69 to 0.98] | 0.96 [0.78 to 1.19] | 0.92 [0.77 to 1.09] | 0.95 [0.79 to 1.14]
  Day 56 (Comparison to qNIV Reference [Group O] Day 56) | 1.08 [0.89 to 1.32] | 0.87 [0.68 to 1.12] | 0.85 [0.69 to 1.05] | 0.87 [0.72 to 1.05] | 0.94 [0.78 to 1.12] | 0.86 [0.72 to 1.04] | 0.95 [0.79 to 1.14] | 0.88 [0.72 to 1.08] | 0.83 [0.68 to 1.00] | 0.98 [0.79 to 1.21] | 0.92 [0.76 to 1.10] | 0.89 [0.74 to 1.08]
  Day 70 (Comparison to qNIV Reference [Group O] Day 70) | 1.20 [0.98 to 1.48] | 0.96 [0.76 to 1.22] | 0.96 [0.79 to 1.18] | 1.00 [0.83 to 1.20] | 1.17 [0.93 to 1.47] | 0.89 [0.74 to 1.07] | 1.08 [0.91 to 1.28] | 0.98 [0.80 to 1.21] | 0.86 [0.72 to 1.02] | 1.09 [0.87 to 1.35] | 1.01 [0.83 to 1.22] | 1.05 [0.87 to 1.26]
  Day 84 (Comparison to qNIV Reference [Group O] Day 84) | 1.27 [1.01 to 1.60] | 1.08 [0.81 to 1.43] | 0.97 [0.75 to 1.25] | 0.99 [0.77 to 1.28] | 1.22 [0.95 to 1.58] | 1.08 [0.80 to 1.44] | 1.22 [0.98 to 1.51] | 1.03 [0.80 to 1.33] | 0.82 [0.64 to 1.05] | 1.05 [0.77 to 1.41] | 1.03 [0.80 to 1.33] | 1.17 [0.92 to 1.49]
  Day 182 (Comparison to qNIV Reference [Group O] Day 182) | 1.23 [0.96 to 1.57] | 0.93 [0.70 to 1.22] | 0.93 [0.69 to 1.24] | 0.95 [0.72 to 1.25] | 1.14 [0.88 to 1.49] | 1.05 [0.78 to 1.41] | 1.08 [0.87 to 1.36] | 0.99 [0.76 to 1.29] | 0.80 [0.61 to 1.04] | 1.10 [0.83 to 1.48] | 0.95 [0.74 to 1.23] | 1.14 [0.88 to 1.47]
  Day70 (Comparison to qNIV Reference [Group O] Day 28)** | 1.14 [0.93 to 1.39] | 0.90 [0.71 to 1.12] | 0.90 [0.74 to 1.09] | 0.95 [0.79 to 1.13] | 1.10 [0.89 to 1.37] | 0.84 [0.70 to 1.00] | 1.03 [0.87 to 1.21] | 0.92 [0.76 to 1.11] | 0.81 [0.69 to 0.96] | 1.03 [0.84 to 1.27] | 0.96 [0.81 to 1.15] | 0.98 [0.83 to 1.17]

31. Secondary Outcome: HAI Antibody Titers Specific for the HA Receptor Binding Domains of Vaccine Homologous Influenza A/Cambodia (H3N2 Subtype) Expressed as GMTR
Description: as for outcome 28
Time Frame: Day 28 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric mean titer ratio
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41
Geometric mean titer ratio
  Day 28 (Comparison to qNIV Reference [Group O] Day 28) | 0.98 [0.72 to 1.33] | 0.94 [0.58 to 1.53] | 0.72 [0.51 to 1.02] | 0.72 [0.52 to 1.01] | 0.97 [0.65 to 1.44] | 0.82 [0.58 to 1.16] | 0.93 [0.69 to 1.26] | 0.71 [0.51 to 0.98] | 0.77 [0.55 to 1.08] | 1.02 [0.67 to 1.54] | 1.08 [0.77 to 1.54] | 0.79 [0.56 to 1.12]
  Day 56 (Comparison to qNIV Reference [Group O] Day 56) | 1.01 [0.75 to 1.36] | 0.96 [0.62 to 1.49] | 0.85 [0.61 to 1.18] | 0.79 [0.56 to 1.11] | 0.90 [0.63 to 1.29] | 0.83 [0.60 to 1.13] | 0.97 [0.73 to 1.30] | 0.77 [0.56 to 1.05] | 0.79 [0.56 to 1.10] | 1.14 [0.75 to 1.73] | 1.04 [0.74 to 1.47] | 0.83 [0.60 to 1.17]
  Day 70 (Comparison to qNIV Reference [Group O] Day 70) | 1.02 [0.77 to 1.34] | 1.05 [0.68 to 1.61] | 0.92 [0.67 to 1.27] | 0.83 [0.61 to 1.13] | 1.05 [0.74 to 1.48] | 0.91 [0.66 to 1.25] | 1.00 [0.76 to 1.32] | 0.92 [0.68 to 1.24] | 0.81 [0.59 to 1.11] | 1.15 [0.77 to 1.71] | 1.03 [0.74 to 1.43] | 0.90 [0.66 to 1.23]
  Day 84 (Comparison to qNIV Reference [Group O] Day 84) | 1.13 [0.85 to 1.52] | 1.36 [0.87 to 2.12] | 1.03 [0.72 to 1.46] | 0.94 [0.68 to 1.32] | 1.18 [0.82 to 1.70] | 1.06 [0.75 to 1.51] | 1.20 [0.89 to 1.61] | 1.06 [0.77 to 1.46] | 0.93 [0.66 to 1.32] | 1.40 [0.96 to 2.07] | 1.38 [1.00 to 1.90] | 0.99 [0.72 to 1.36]
  Day 182 (Comparison to qNIV Reference [Group O] Day 182) | 1.25 [0.94 to 1.66] | 1.42 [0.91 to 2.19] | 0.98 [0.68 to 1.42] | 0.85 [0.60 to 1.19] | 1.15 [0.82 to 1.62] | 1.03 [0.73 to 1.45] | 1.12 [0.83 to 1.51] | 1.10 [0.81 to 1.50] | 1.06 [0.77 to 1.46] | 1.39 [0.98 to 1.97] | 1.15 [0.83 to 1.61] | 1.01 [0.73 to 1.39]
  Day70 (Comparison to qNIV Reference [Group O] Day 28)** | 0.94 [0.70 to 1.26] | 0.96 [0.61 to 1.51] | 0.84 [0.59 to 1.20] | 0.76 [0.54 to 1.07] | 0.96 [0.66 to 1.38] | 0.84 [0.59 to 1.18] | 0.92 [0.69 to 1.23] | 0.85 [0.61 to 1.18] | 0.75 [0.53 to 1.06] | 1.04 [0.68 to 1.58] | 0.95 [0.67 to 1.36] | 0.83 [0.59 to 1.15]

32. Secondary Outcome: HAI Antibody Titers Specific for the HA Receptor Binding Domains of Vaccine Homologous Influenza A/Hong Kong (H3N2 Subtype) Expressed as GMTR
Description: as for outcome 28
Time Frame: Day 28 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric mean titer ratio
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41
Geometric mean titer ratio
  Day 28 (Comparison to qNIV Reference [Group O] Day 28) | 0.96 [0.73 to 1.26] | 0.94 [0.62 to 1.42] | 0.73 [0.53 to 1.00] | 0.73 [0.53 to 1.00] | 0.91 [0.63 to 1.30] | 0.77 [0.57 to 1.03] | 0.95 [0.72 to 1.25] | 0.76 [0.56 to 1.03] | 0.86 [0.63 to 1.18] | 0.99 [0.71 to 1.39] | 0.99 [0.70 to 1.39] | 0.88 [0.64 to 1.20]
  Day 56 (Comparison to qNIV Reference [Group O] Day 56) | 1.03 [0.78 to 1.34] | 0.97 [0.66 to 1.43] | 0.82 [0.61 to 1.11] | 0.80 [0.59 to 1.09] | 0.82 [0.60 to 1.12] | 0.87 [0.66 to 1.15] | 1.02 [0.79 to 1.33] | 0.78 [0.59 to 1.04] | 0.91 [0.68 to 1.21] | 0.99 [0.71 to 1.36] | 1.02 [0.74 to 1.40] | 0.94 [0.70 to 1.25]
  Day 70 (Comparison to qNIV Reference [Group O] Day 70) | 1.07 [0.83 to 1.38] | 1.14 [0.79 to 1.66] | 0.97 [0.73 to 1.28] | 0.91 [0.70 to 1.19] | 0.96 [0.72 to 1.28] | 0.92 [0.72 to 1.19] | 1.01 [0.80 to 1.29] | 0.84 [0.65 to 1.08] | 0.91 [0.70 to 1.19] | 1.07 [0.81 to 1.43] | 1.09 [0.81 to 1.47] | 0.94 [0.72 to 1.22]
  Day 84 (Comparison to qNIV Reference [Group O] Day 84) | 1.05 [0.78 to 1.41] | 1.20 [0.82 to 1.77] | 0.94 [0.66 to 1.34] | 0.93 [0.66 to 1.31] | 1.05 [0.75 to 1.48] | 0.95 [0.70 to 1.31] | 1.19 [0.89 to 1.60] | 0.94 [0.69 to 1.28] | 0.93 [0.66 to 1.30] | 1.19 [0.81 to 1.75] | 1.18 [0.85 to 1.65] | 1.14 [0.82 to 1.59]
  Day 182 (Comparison to qNIV Reference [Group O] Day 182) | 1.03 [0.78 to 1.37] | 1.18 [0.79 to 1.77] | 0.89 [0.63 to 1.25] | 0.87 [0.62 to 1.21] | 1.01 [0.73 to 1.41] | 0.92 [0.66 to 1.30] | 1.03 [0.78 to 1.36] | 0.94 [0.70 to 1.26] | 0.98 [0.72 to 1.33] | 1.19 [0.87 to 1.64] | 1.09 [0.80 to 1.50] | 1.06 [0.75 to 1.50]
  Day70 (Comparison to qNIV Reference [Group O] Day 28)** | 0.99 [0.74 to 1.31] | 1.05 [0.70 to 1.59] | 0.89 [0.63 to 1.24] | 0.84 [0.61 to 1.16] | 0.89 [0.64 to 1.25] | 0.86 [0.64 to 1.16] | 0.93 [0.71 to 1.21] | 0.78 [0.57 to 1.06] | 0.85 [0.61 to 1.17] | 0.97 [0.69 to 1.36] | 1.02 [0.72 to 1.44] | 0.86 [0.63 to 1.18]

33. Secondary Outcome: HAI Antibody Titers Specific for the HA Receptor Binding Domains of Vaccine Homologous Influenza B/Maryland (Victoria Subtype) Expressed as GMTR
Description: as for outcome 28
Time Frame: Day 28 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric mean titer ratio
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41
Geometric mean titer ratio
  Day 28 (Comparison to qNIV Reference [Group O] Day 28) | 0.96 [0.75 to 1.24] | 0.89 [0.65 to 1.22] | 0.62 [0.47 to 0.82] | 0.74 [0.55 to 0.99] | 0.83 [0.61 to 1.14] | 0.70 [0.53 to 0.94] | 0.90 [0.71 to 1.14] | 0.67 [0.51 to 0.87] | 0.65 [0.50 to 0.85] | 0.78 [0.59 to 1.04] | 0.78 [0.58 to 1.05] | 0.78 [0.60 to 1.03]
  Day 56 (Comparison to qNIV Reference [Group O] Day 56) | 1.04 [0.81 to 1.35] | 0.85 [0.65 to 1.11] | 0.75 [0.58 to 0.96] | 0.87 [0.67 to 1.13] | 0.74 [0.56 to 0.99] | 0.76 [0.60 to 0.98] | 0.95 [0.77 to 1.17] | 0.74 [0.59 to 0.94] | 0.70 [0.55 to 0.90] | 0.87 [0.67 to 1.14] | 0.76 [0.57 to 1.00] | 0.82 [0.65 to 1.04]
  Day 70 (Comparison to qNIV Reference [Group O] Day 70) | 1.18 [0.92 to 1.52] | 1.04 [0.79 to 1.38] | 0.84 [0.65 to 1.08] | 0.98 [0.76 to 1.27] | 1.04 [0.80 to 1.36] | 0.88 [0.70 to 1.12] | 1.05 [0.86 to 1.30] | 0.90 [0.71 to 1.14] | 0.82 [0.65 to 1.04] | 1.02 [0.79 to 1.33] | 0.95 [0.72 to 1.24] | 1.01 [0.80 to 1.27]
  Day 84 (Comparison to qNIV Reference [Group O] Day 84) | 1.10 [0.84 to 1.44] | 1.03 [0.82 to 1.31] | 0.90 [0.69 to 1.17] | 0.87 [0.67 to 1.12] | 1.02 [0.78 to 1.32] | 0.92 [0.73 to 1.17] | 1.15 [0.93 to 1.41] | 0.78 [0.61 to 0.98] | 0.79 [0.61 to 1.01] | 0.94 [0.73 to 1.22] | 0.99 [0.77 to 1.27] | 0.95 [0.75 to 1.21]
  Day 182 (Comparison to qNIV Reference [Group O] Day 182) | 1.15 [0.90 to 1.46] | 1.01 [0.81 to 1.26] | 0.88 [0.70 to 1.11] | 0.86 [0.66 to 1.11] | 0.97 [0.77 to 1.23] | 0.86 [0.69 to 1.07] | 1.08 [0.88 to 1.33] | 0.85 [0.68 to 1.06] | 0.88 [0.71 to 1.09] | 0.90 [0.71 to 1.14] | 0.89 [0.71 to 1.13] | 0.92 [0.73 to 1.15]
  Day70 (Comparison to qNIV Reference [Group O] Day 28)** | 1.03 [0.79 to 1.34] | 0.90 [0.66 to 1.22] | 0.72 [0.54 to 0.97] | 0.85 [0.63 to 1.14] | 0.90 [0.67 to 1.21] | 0.76 [0.58 to 1.00] | 0.91 [0.73 to 1.14] | 0.78 [0.59 to 1.02] | 0.71 [0.54 to 0.93] | 0.89 [0.66 to 1.19] | 0.82 [0.61 to 1.11] | 0.87 [0.67 to 1.14]

34. Secondary Outcome: HAI Antibody Titers Specific for the HA Receptor Binding Domains of Vaccine Homologous Influenza B/Phuket (Yamagata Subtype) Expressed as GMTR
Description: as for outcome 28
Time Frame: Day 28 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric mean titer ratio
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41
Geometric mean titer ratio
  Day 28 (Comparison to qNIV Reference [Group O] Day 28) | 0.76 [0.59 to 0.98] | 0.58 [0.44 to 0.77] | 0.44 [0.34 to 0.57] | 0.50 [0.39 to 0.65] | 0.68 [0.51 to 0.91] | 0.50 [0.39 to 0.65] | 0.64 [0.51 to 0.80] | 0.59 [0.46 to 0.76] | 0.49 [0.38 to 0.62] | 0.60 [0.46 to 0.77] | 0.60 [0.47 to 0.77] | 0.70 [0.53 to 0.92]
  Day 56 (Comparison to qNIV Reference [Group O] Day 56) | 0.81 [0.63 to 1.04] | 0.62 [0.48 to 0.81] | 0.53 [0.41 to 0.70] | 0.54 [0.42 to 0.70] | 0.69 [0.51 to 0.92] | 0.56 [0.44 to 0.72] | 0.68 [0.55 to 0.84] | 0.65 [0.52 to 0.83] | 0.52 [0.41 to 0.65] | 0.65 [0.51 to 0.85] | 0.61 [0.47 to 0.79] | 0.75 [0.57 to 0.97]
  Day 70 (Comparison to qNIV Reference [Group O] Day 70) | 1.02 [0.77 to 1.34] | 0.86 [0.66 to 1.13] | 0.69 [0.51 to 0.92] | 0.76 [0.59 to 0.99] | 1.00 [0.74 to 1.36] | 0.72 [0.56 to 0.91] | 0.86 [0.68 to 1.08] | 0.79 [0.61 to 1.02] | 0.66 [0.51 to 0.84] | 0.84 [0.63 to 1.13] | 0.79 [0.60 to 1.03] | 0.89 [0.69 to 1.16]
  Day 84 (Comparison to qNIV Reference [Group O] Day 84) | 0.95 [0.74 to 1.22] | 0.82 [0.65 to 1.02] | 0.73 [0.57 to 0.92] | 0.72 [0.56 to 0.92] | 1.00 [0.77 to 1.29] | 0.73 [0.58 to 0.91] | 0.90 [0.72 to 1.12] | 0.73 [0.58 to 0.91] | 0.68 [0.54 to 0.85] | 0.86 [0.67 to 1.12] | 0.87 [0.68 to 1.11] | 0.88 [0.70 to 1.12]
  Day 182 (Comparison to qNIV Reference [Group O] Day 182) | 1.11 [0.86 to 1.43] | 0.91 [0.74 to 1.11] | 0.80 [0.63 to 1.02] | 0.82 [0.64 to 1.05] | 1.05 [0.81 to 1.35] | 0.80 [0.64 to 1.00] | 0.90 [0.74 to 1.10] | 0.83 [0.67 to 1.04] | 0.80 [0.65 to 0.99] | 0.93 [0.75 to 1.14] | 0.84 [0.67 to 1.05] | 0.94 [0.74 to 1.20]
  Day70 (Comparison to qNIV Reference [Group O] Day 28)** | 0.86 [0.65 to 1.13] | 0.73 [0.56 to 0.95] | 0.57 [0.43 to 0.76] | 0.64 [0.50 to 0.83] | 0.85 [0.63 to 1.14] | 0.60 [0.48 to 0.76] | 0.72 [0.58 to 0.91] | 0.56 [0.44 to 0.71] | 0.56 [0.44 to 0.71] | 0.71 [0.54 to 0.94] | 0.66 [0.51 to 0.86] | 0.75 [0.58 to 0.97]

35. Secondary Outcome: HAI Antibody Titers Specific for the HA Receptor Binding Domains of Vaccine Homologous Influenza B/Washington (Victoria Subtype)Expressed as GMTR
Description: as for outcome 28
Time Frame: Day 28 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric mean titer ratio
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41
Geometric mean titer ratio
  Day 28 (Comparison to qNIV Reference [Group O] Day 28) | 0.93 [0.76 to 1.14] | 0.82 [0.65 to 1.03] | 0.75 [0.59 to 0.96] | 0.79 [0.61 to 1.03] | 0.85 [0.66 to 1.10] | 0.77 [0.60 to 0.99] | 0.85 [0.68 to 1.06] | 0.74 [0.58 to 0.93] | 0.74 [0.58 to 0.94] | 0.83 [0.65 to 1.06] | 0.80 [0.60 to 1.06] | 0.82 [0.64 to 1.06]
  Day 56 (Comparison to qNIV Reference [Group O] Day 56) | 0.91 [0.74 to 1.11] | 0.87 [0.70 to 1.09] | 0.72 [0.57 to 0.91] | 0.85 [0.66 to 1.09] | 0.78 [0.62 to 0.99] | 0.76 [0.60 to 0.96] | 0.88 [0.73 to 1.07] | 0.76 [0.61 to 0.95] | 0.80 [0.64 to 1.00] | 0.82 [0.64 to 1.04] | 0.80 [0.62 to 1.04] | 0.86 [0.69 to 1.07]
  Day 70 (Comparison to qNIV Reference [Group O] Day 70) | 1.01 [0.83 to 1.24] | 0.88 [0.70 to 1.12] | 0.82 [0.64 to 1.05] | 0.91 [0.71 to 1.17] | 0.91 [0.70 to 1.17] | 0.80 [0.63 to 1.01] | 0.90 [0.74 to 1.10] | 0.79 [0.63 to 0.99] | 0.79 [0.62 to 1.00] | 0.96 [0.75 to 1.23] | 0.85 [0.64 to 1.12] | 0.85 [0.68 to 1.06]
  Day 84 (Comparison to qNIV Reference [Group O] Day 84) | 0.86 [0.68 to 1.10] | 0.88 [0.68 to 1.15] | 0.74 [0.56 to 0.98] | 0.80 [0.60 to 1.06] | 0.90 [0.68 to 1.20] | 0.73 [0.56 to 0.94] | 0.92 [0.73 to 1.16] | 0.73 [0.55 to 0.99] | 0.71 [0.53 to 0.95] | 0.84 [0.63 to 1.13] | 0.88 [0.65 to 1.18] | 0.84 [0.65 to 1.11]
  Day 182 (Comparison to qNIV Reference [Group O] Day 182) | 0.91 [0.72 to 1.15] | 0.83 [0.64 to 1.09] | 0.73 [0.55 to 0.97] | 0.81 [0.60 to 1.08] | 0.83 [0.64 to 1.07] | 0.72 [0.54 to 0.94] | 0.86 [0.68 to 1.08] | 0.78 [0.59 to 1.01] | 0.79 [0.60 to 1.03] | 0.90 [0.69 to 1.16] | 0.75 [0.57 to 0.99] | 0.86 [0.67 to 1.11]
  Day70 (Comparison to qNIV Reference [Group O] Day 28)** | 0.99 [0.80 to 1.21] | 0.86 [0.67 to 1.11] | 0.81 [0.62 to 1.04] | 0.88 [0.68 to 1.15] | 0.87 [0.67 to 1.12] | 0.77 [0.60 to 0.98] | 0.88 [0.72 to 1.08] | 0.76 [0.60 to 0.96] | 0.77 [0.60 to 0.98] | 0.93 [0.72 to 1.19] | 0.83 [0.63 to 1.11] | 0.83 [0.66 to 1.05]

36. Secondary Outcome: Percentage of Participants With a Reciprocal HAI Titer ≥ 40 Specific for the HA Receptor Binding Domains of Vaccine Homologous Influenza A/Brisbane (H1N1 Subtype) Expressed as Seroprotection Rate (SPR).
Description: Percentage of participants with a reciprocal HAI titer ≥ 40 specific for the HA receptor binding domains of vaccine homologous Influenza A/Brisbane (H1N1 Subtype) on Days 56, 70, and other follow-up time points.
Time Frame: Day 28 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Number (95% Confidence Interval); unit: percentage of participants(SPR)
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
percentage of participants(SPR)
  Day 28 | 96.3 [89.4 to 99.2] | 85.0 [70.2 to 94.3] | 94.7 [82.3 to 99.4] | 94.6 [81.8 to 99.3] | 92.7 [80.1 to 98.5] | 85.4 [70.8 to 94.4] | 98.7 [93.1 to 100.0] | 92.3 [79.1 to 98.4] | 87.2 [72.6 to 95.7] | 92.3 [79.1 to 98.4] | 94.9 [82.7 to 99.4] | 95.1 [83.5 to 99.4] | 100.0 [91.0 to 100.0]
  Day 56 | 96.2 [89.3 to 99.2] | 87.2 [72.6 to 95.7] | 97.2 [85.5 to 99.9] | 91.7 [77.5 to 98.2] | 87.5 [73.2 to 95.8] | 87.5 [73.2 to 95.8] | 94.9 [87.5 to 98.6] | 89.7 [75.8 to 97.1] | 84.2 [68.7 to 94.0] | 91.9 [78.1 to 98.3] | 92.1 [78.6 to 98.3] | 97.5 [86.8 to 99.9] | 100.0 [91.0 to 100.0]
  Day 70 | 97.4 [90.9 to 99.7] | 94.9 [82.7 to 99.4] | 94.3 [80.8 to 99.3] | 97.2 [85.5 to 99.9] | 95.0 [83.1 to 99.4] | 95.0 [83.1 to 99.4] | 98.7 [92.9 to 100.0] | 97.4 [86.2 to 99.9] | 92.1 [78.6 to 98.3] | 97.2 [85.5 to 99.9] | 97.3 [85.8 to 99.9] | 100.0 [91.4 to 100.0] | 100.0 [90.7 to 100.0]
  Day 84 | 94.9 [87.4 to 98.6] | 89.7 [75.8 to 97.1] | 94.1 [80.3 to 99.3] | 94.3 [80.8 to 99.3] | 87.2 [72.6 to 95.7] | 78.9 [62.7 to 90.4] | 92.1 [83.6 to 97.0] | 97.4 [86.2 to 99.9] | 89.5 [75.2 to 97.1] | 94.1 [80.3 to 99.3] | 91.9 [78.1 to 98.3] | 95.1 [83.5 to 99.4] | 94.7 [82.3 to 99.4]
  Day 182 | 90.7 [81.7 to 96.2] | 82.1 [66.5 to 92.5] | 85.3 [68.9 to 95.0] | 85.7 [69.7 to 95.2] | 79.5 [63.5 to 90.7] | 68.4 [51.3 to 82.5] | 82.7 [72.2 to 90.4] | 75.7 [58.8 to 88.2] | 78.4 [61.8 to 90.2] | 83.3 [67.2 to 93.6] | 81.6 [65.7 to 92.3] | 82.1 [66.5 to 92.5] | 78.9 [62.7 to 90.4]

37. Secondary Outcome: Percentage of Participants With a Reciprocal HAI Titer ≥ 40 Specific for the HA Receptor Binding Domains of Vaccine Homologous Influenza A/Kansas (H3N2 Subtype) Expressed as SPR
Description: Percentage of participants with a reciprocal HAI titer ≥ 40 specific for the HA receptor binding domains of vaccine homologous Influenza A/Kansas (H3N2 Subtype) on Days 56, 70, and other follow-up time points.
Time Frame: Day 28 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Number (95% Confidence Interval); unit: percentage of participants(SPR)
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
percentage of participants(SPR)
  Day 28 | 93.8 [86.0 to 97.9] | 75.0 [58.8 to 87.3] | 73.7 [56.9 to 86.6] | 78.4 [61.8 to 90.2] | 87.8 [73.8 to 95.9] | 85.4 [70.8 to 94.4] | 89.7 [80.8 to 95.5] | 79.5 [63.5 to 90.7] | 89.7 [75.8 to 97.1] | 87.2 [72.6 to 95.7] | 92.3 [79.1 to 98.4] | 90.2 [76.9 to 97.3] | 92.3 [79.1 to 98.4]
  Day 56 | 89.9 [81.0 to 95.5] | 71.8 [55.1 to 85.0] | 77.8 [60.8 to 89.9] | 75.0 [57.8 to 87.9] | 85.0 [70.2 to 94.3] | 85.0 [70.2 to 94.3] | 91.1 [82.6 to 96.4] | 79.5 [63.5 to 90.7] | 89.5 [75.2 to 97.1] | 83.8 [68.0 to 93.8] | 81.6 [65.7 to 92.3] | 85.0 [70.2 to 94.3] | 89.7 [75.8 to 97.1]
  Day 70 | 98.7 [93.0 to 100.0] | 89.7 [75.8 to 97.1] | 85.7 [69.7 to 95.2] | 97.2 [85.5 to 99.9] | 90.0 [76.3 to 97.2] | 95.0 [83.1 to 99.4] | 94.7 [87.1 to 98.5] | 94.7 [82.3 to 99.4] | 92.1 [78.6 to 98.3] | 83.3 [67.2 to 93.6] | 91.9 [78.1 to 98.3] | 87.8 [73.8 to 95.9] | 89.5 [75.2 to 97.1]
  Day 84 | 94.9 [87.4 to 98.6] | 89.7 [75.8 to 97.1] | 82.4 [65.5 to 93.2] | 91.4 [76.9 to 98.2] | 94.9 [82.7 to 99.4] | 92.1 [78.6 to 98.3] | 96.1 [88.9 to 99.2] | 92.1 [78.6 to 98.3] | 94.7 [82.3 to 99.4] | 85.3 [68.9 to 95.0] | 91.9 [78.1 to 98.3] | 87.8 [73.8 to 95.9] | 86.8 [71.9 to 95.6]
  Day 182 | 86.7 [76.8 to 93.4] | 79.5 [63.5 to 90.7] | 73.5 [55.7 to 87.1] | 77.1 [59.9 to 89.6] | 92.3 [79.1 to 98.4] | 81.6 [65.7 to 92.3] | 90.7 [81.7 to 96.2] | 83.8 [68.0 to 93.8] | 97.3 [85.8 to 99.9] | 83.3 [67.2 to 93.6] | 86.8 [71.9 to 95.6] | 84.6 [69.5 to 94.1] | 81.6 [65.7 to 92.3]

38. Secondary Outcome: Percentage of Participants With a Reciprocal HAI Titer ≥ 40 Specific for the HA Receptor Binding Domains of Vaccine Homologous Influenza A/Wisconsin (H1N1 Subtype) Expressed as SPR
Description: Percentage of participants with a reciprocal HAI titer ≥ 40 specific for the HA receptor binding domains of vaccine homologous Influenza A/Wisconsin (H1N1 Subtype) on Days 56, 70, and other follow-up time points.
Time Frame: Day 28 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
percentage of participants
  Day 28 | 98.8 [93.2 to 100.0] | 100.0 [91.2 to 100.0] | 100.0 [90.7 to 100.0] | 100.0 [90.5 to 100.0] | 100.0 [91.4 to 100.0] | 97.6 [87.1 to 99.9] | 100.0 [95.4 to 100.0] | 100.0 [91.0 to 100.0] | 100.0 [91.0 to 100.0] | 97.4 [86.5 to 99.9] | 100.0 [91.0 to 100.0] | 97.6 [87.1 to 99.9] | 100.0 [91.0 to 100.0]
  Day 56 | 97.5 [91.2 to 99.7] | 97.4 [86.5 to 99.9] | 100.0 [90.3 to 100.0] | 97.2 [85.5 to 99.9] | 97.5 [86.8 to 99.9] | 95.0 [83.1 to 99.4] | 98.7 [93.1 to 100.0] | 100.0 [91.0 to 100.0] | 97.4 [86.2 to 99.9] | 100.0 [90.5 to 100.0] | 100.0 [90.7 to 100.0] | 97.5 [86.8 to 99.9] | 97.4 [86.5 to 99.9]
  Day 70 | 98.7 [93.0 to 100.0] | 100.0 [91.0 to 100.0] | 100.0 [90.0 to 100.0] | 100.0 [90.3 to 100.0] | 100.0 [91.2 to 100.0] | 97.5 [86.8 to 99.9] | 98.7 [92.9 to 100.0] | 100.0 [90.7 to 100.0] | 100.0 [90.7 to 100.0] | 100.0 [90.3 to 100.0] | 97.3 [85.8 to 99.9] | 100.0 [91.4 to 100.0] | 100.0 [90.7 to 100.0]
  Day 84 | 93.6 [85.7 to 97.9] | 89.7 [75.8 to 97.1] | 88.2 [72.5 to 96.7] | 88.6 [73.3 to 96.8] | 87.2 [72.6 to 95.7] | 86.8 [71.9 to 95.6] | 90.8 [81.9 to 96.2] | 89.5 [75.2 to 97.1] | 81.6 [65.7 to 92.3] | 88.2 [72.5 to 96.7] | 89.2 [74.6 to 97.0] | 92.7 [80.1 to 98.5] | 86.8 [71.9 to 95.6]
  Day 182 | 89.3 [80.1 to 95.3] | 79.5 [63.5 to 90.7] | 88.2 [72.5 to 96.7] | 77.1 [59.9 to 89.6] | 87.2 [72.6 to 95.7] | 76.3 [59.8 to 88.6] | 86.7 [76.8 to 93.4] | 75.7 [58.8 to 88.2] | 73.0 [55.9 to 86.2] | 83.3 [67.2 to 93.6] | 73.7 [56.9 to 86.6] | 89.7 [75.8 to 97.1] | 86.8 [71.9 to 95.6]

39. Secondary Outcome: Percentage of Participants With a Reciprocal HAI Titer ≥ 40 Specific for the HA Receptor Binding Domains of Vaccine Homologous Influenza A/Cambodia (H3N2 Subtype) Expressed as SPR
Description: Percentage of participants with a reciprocal HAI titer ≥ 40 specific for the HA receptor binding domains of vaccine homologous Influenza A/Cambodia (H3N2 Subtype) on Days 56, 70, and other follow-up time points.
Time Frame: Day 28 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
percentage of participants
  Day 28 | 90.0 [81.2 to 95.6] | 77.5 [61.5 to 89.2] | 71.1 [54.1 to 84.6] | 89.2 [74.6 to 97.0] | 90.2 [76.9 to 97.3] | 87.8 [73.8 to 95.9] | 87.2 [77.7 to 93.7] | 82.1 [66.5 to 92.5] | 87.2 [72.6 to 95.7] | 76.9 [60.7 to 88.9] | 94.9 [82.7 to 99.4] | 85.4 [70.8 to 94.4] | 100.0 [91.0 to 100.0]
  Day 56 | 86.1 [76.5 to 92.8] | 79.5 [63.5 to 90.7] | 72.2 [54.8 to 85.8] | 77.8 [60.8 to 89.9] | 87.5 [73.2 to 95.8] | 82.5 [67.2 to 92.7] | 82.3 [72.1 to 90.0] | 74.4 [57.9 to 87.0] | 78.9 [62.7 to 90.4] | 75.7 [58.8 to 88.2] | 76.3 [59.8 to 88.6] | 75.0 [58.8 to 87.3] | 89.7 [75.8 to 97.1]
  Day 70 | 90.9 [82.2 to 96.3] | 84.6 [69.5 to 94.1] | 80.0 [63.1 to 91.6] | 88.9 [73.9 to 96.9] | 95.0 [83.1 to 99.4] | 85.0 [70.2 to 94.3] | 92.1 [83.6 to 97.0] | 84.2 [68.7 to 94.0] | 81.6 [65.7 to 92.3] | 80.6 [64.0 to 91.8] | 89.2 [74.6 to 97.0] | 92.7 [80.1 to 98.5] | 97.4 [86.2 to 99.9]
  Day 84 | 73.1 [61.8 to 82.5] | 71.8 [55.1 to 85.0] | 64.7 [46.5 to 80.3] | 62.9 [44.9 to 78.5] | 76.9 [60.7 to 88.9] | 68.4 [51.3 to 82.5] | 71.1 [59.5 to 80.9] | 71.1 [54.1 to 84.6] | 63.2 [46.0 to 78.2] | 61.8 [43.6 to 77.8] | 75.7 [58.8 to 88.2] | 61.0 [44.5 to 75.8] | 78.9 [62.7 to 90.4]
  Day 182 | 66.7 [54.8 to 77.1] | 71.8 [55.1 to 85.0] | 50.0 [32.4 to 67.6] | 45.7 [28.8 to 63.4] | 66.7 [49.8 to 80.9] | 63.2 [46.0 to 78.2] | 57.3 [45.4 to 68.7] | 62.2 [44.8 to 77.5] | 64.9 [47.5 to 79.8] | 55.6 [38.1 to 72.1] | 63.2 [46.0 to 78.2] | 56.4 [39.6 to 72.2] | 65.8 [48.6 to 80.4]

40. Secondary Outcome: Percentage of Participants With a Reciprocal HAI Titer ≥ 40 Specific for the HA Receptor Binding Domains of Vaccine Homologous Influenza A/Hong Kong (H3N2 Subtype) Expressed as SPR
Description: Percentage of participants with a reciprocal HAI titer ≥ 40 specific for the HA receptor binding domains of vaccine homologous Influenza A/Hong Kong (H3N2 Subtype)on Days 56, 70, and other follow-up time points.
Time Frame: Day 28 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Number (95% Confidence Interval); unit: percentage of participants(SPR)
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
percentage of participants(SPR)
  Day 28 | 98.8 [93.2 to 100.0] | 92.5 [79.6 to 98.4] | 97.4 [86.2 to 99.9] | 91.9 [78.1 to 98.3] | 95.1 [83.5 to 99.4] | 97.6 [87.1 to 99.9] | 100.0 [95.4 to 100.0] | 100.0 [91.0 to 100.0] | 100.0 [91.0 to 100.0] | 97.4 [86.5 to 99.9] | 100.0 [91.0 to 100.0] | 95.1 [83.5 to 99.4] | 97.4 [86.5 to 99.9]
  Day 56 | 97.5 [91.2 to 99.7] | 89.7 [75.8 to 97.1] | 97.2 [85.5 to 99.9] | 88.9 [73.9 to 96.9] | 95.0 [83.1 to 99.4] | 95.0 [83.1 to 99.4] | 97.5 [91.2 to 99.7] | 92.3 [79.1 to 98.4] | 100.0 [90.7 to 100.0] | 97.3 [85.8 to 99.9] | 100.0 [90.7 to 100.0] | 95.0 [83.1 to 99.4] | 100.0 [91.0 to 100.0]
  Day 70 | 97.4 [90.9 to 99.7] | 94.9 [82.7 to 99.4] | 100.0 [90.0 to 100.0] | 97.2 [85.5 to 99.9] | 97.5 [86.8 to 99.9] | 97.5 [86.8 to 99.9] | 100.0 [95.3 to 100.0] | 100.0 [90.7 to 100.0] | 97.4 [86.2 to 99.9] | 97.2 [85.5 to 99.9] | 100.0 [90.5 to 100.0] | 97.6 [87.1 to 99.9] | 100.0 [90.7 to 100.0]
  Day 84 | 88.5 [79.2 to 94.6] | 84.6 [69.5 to 94.1] | 85.3 [68.9 to 95.0] | 82.9 [66.4 to 93.4] | 92.3 [79.1 to 98.4] | 86.8 [71.9 to 95.6] | 88.2 [78.7 to 94.4] | 86.8 [71.9 to 95.6] | 81.6 [65.7 to 92.3] | 88.2 [72.5 to 96.7] | 89.2 [74.6 to 97.0] | 87.8 [73.8 to 95.9] | 89.5 [75.2 to 97.1]
  Day 182 | 84.0 [73.7 to 91.4] | 82.1 [66.5 to 92.5] | 73.5 [55.6 to 87.1] | 77.1 [59.9 to 89.6] | 84.6 [69.5 to 94.1] | 78.9 [62.7 to 90.4] | 85.3 [75.3 to 92.4] | 86.5 [71.2 to 95.5] | 86.5 [71.2 to 95.5] | 88.9 [73.9 to 96.9] | 81.6 [65.7 to 92.3] | 84.6 [69.5 to 94.1] | 86.8 [71.9 to 95.6]

41. Secondary Outcome: Percentage of Participants With a Reciprocal HAI Titer ≥ 40 Specific for the HA Receptor Binding Domains of Vaccine Homologous Influenza B/Maryland (Victoria Subtype) Expressed as SPR
Description: Percentage of participants with a reciprocal HAI titer ≥ 40 specific for the HA receptor binding domains of vaccine homologous Influenza B/Maryland (Victoria Subtype) on Days 56, 70, and other follow-up time points.
Time Frame: Day 28 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
percentage of participants
  Day 28 | 90.0 [81.2 to 95.6] | 77.5 [61.5 to 89.2] | 73.7 [56.9 to 86.6] | 75.7 [58.8 to 88.2] | 78.0 [62.4 to 89.4] | 73.2 [57.1 to 85.8] | 83.3 [73.2 to 90.8] | 76.9 [60.7 to 88.9] | 66.7 [49.8 to 80.9] | 82.1 [66.5 to 92.5] | 76.9 [60.7 to 88.9] | 80.5 [65.1 to 91.2] | 87.2 [72.6 to 95.7]
  Day 56 | 87.3 [78.0 to 93.8] | 74.4 [57.9 to 87.0] | 66.7 [49.0 to 81.4] | 83.3 [67.2 to 93.6] | 67.5 [50.9 to 81.4] | 70.0 [53.5 to 83.4] | 79.7 [69.2 to 88.0] | 74.4 [57.9 to 87.0] | 65.8 [48.6 to 80.4] | 83.8 [68.0 to 93.8] | 71.1 [54.1 to 84.6] | 85.0 [70.2 to 94.3] | 76.9 [60.7 to 88.9]
  Day 70 | 92.2 [83.8 to 97.1] | 82.1 [66.5 to 92.5] | 74.3 [56.7 to 87.5] | 88.9 [73.9 to 96.9] | 77.5 [61.5 to 89.2] | 77.5 [61.5 to 89.2] | 88.2 [78.7 to 94.4] | 81.6 [65.7 to 92.3] | 76.3 [59.8 to 88.6] | 88.9 [73.9 to 96.9] | 81.1 [64.8 to 92.0] | 87.8 [73.8 to 95.9] | 84.2 [68.7 to 94.0]
  Day 84 | 85.9 [76.2 to 92.7] | 89.7 [75.8 to 97.1] | 82.4 [65.5 to 93.2] | 88.6 [73.3 to 96.8] | 84.6 [69.5 to 94.1] | 81.6 [65.7 to 92.3] | 89.5 [80.3 to 95.3] | 76.3 [59.8 to 88.6] | 78.9 [62.7 to 90.4] | 85.3 [68.9 to 95.0] | 91.9 [78.1 to 98.3] | 85.4 [70.8 to 94.4] | 86.8 [71.9 to 95.6]
  Day 182 | 88.0 [78.4 to 94.0] | 89.7 [75.8 to 97.1] | 73.5 [55.6 to 87.1] | 80.0 [63.1 to 91.6] | 84.6 [69.5 to 94.1] | 76.3 [59.8 to 88.6] | 84.0 [73.7 to 91.4] | 73.0 [55.9 to 86.2] | 81.1 [64.8 to 92.0] | 75.0 [57.8 to 87.9] | 76.3 [59.8 to 88.6] | 79.5 [63.5 to 90.7] | 84.2 [68.7 to 94.0]

42. Secondary Outcome: Percentage of Participants With a Reciprocal HAI Titer ≥ 40 Specific for the HA Receptor Binding Domains of Vaccine Homologous Influenza B/Phuket (Yamagata Subtype) Expressed as SPR
Description: Percentage of participants with a reciprocal HAI titer ≥ 40 specific for the HA receptor binding domains of vaccine homologous Influenza B/Phuket (Yamagata Subtype) on Days 56, 70, and other follow-up time points.
Time Frame: Day 28 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Number (95% Confidence Interval); unit: percentage of participants(SPR)
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
percentage of participants(SPR)
  Day 28 | 90.0 [81.2 to 95.6] | 80.0 [64.4 to 90.9] | 57.9 [40.8 to 73.7] | 67.6 [50.2 to 82.0] | 92.7 [80.1 to 98.5] | 73.2 [57.1 to 85.8] | 83.3 [73.2 to 90.8] | 87.2 [72.6 to 95.7] | 74.4 [57.9 to 87.0] | 89.7 [75.8 to 97.1] | 79.5 [63.5 to 90.7] | 85.4 [70.8 to 94.4] | 97.4 [86.5 to 99.9]
  Day 56 | 89.9 [81.0 to 95.5] | 76.9 [60.7 to 88.9] | 55.6 [38.1 to 72.1] | 66.7 [49.0 to 81.4] | 85.0 [70.2 to 94.3] | 75.0 [58.8 to 87.3] | 77.2 [66.4 to 85.9] | 89.7 [75.8 to 97.1] | 68.4 [51.3 to 82.5] | 89.2 [74.6 to 97.0] | 73.7 [56.9 to 86.6] | 85.0 [70.2 to 94.3] | 97.4 [86.5 to 99.9]
  Day 70 | 90.9 [82.2 to 96.3] | 87.2 [72.6 to 95.7] | 62.9 [44.9 to 78.5] | 80.6 [64.0 to 91.8] | 90.0 [76.3 to 97.2] | 82.5 [67.2 to 92.7] | 88.2 [78.7 to 94.4] | 89.5 [75.2 to 97.1] | 84.2 [68.7 to 94.0] | 91.7 [77.5 to 98.2] | 86.5 [71.2 to 95.5] | 92.7 [80.1 to 98.5] | 94.7 [82.3 to 99.4]
  Day 84 | 94.9 [87.4 to 98.6] | 94.9 [82.7 to 99.4] | 73.5 [55.6 to 87.1] | 80.0 [63.1 to 91.6] | 97.4 [86.5 to 99.9] | 89.5 [75.2 to 97.1] | 92.1 [83.6 to 97.0] | 92.1 [78.6 to 98.1] | 86.8 [71.9 to 95.6] | 88.2 [72.5 to 96.7] | 89.2 [74.6 to 97.0] | 90.2 [76.9 to 97.3] | 100.0 [90.7 to 100.0]
  Day 182 | 92.0 [83.4 to 97.0] | 87.2 [72.6 to 95.7] | 73.5 [55.6 to 87.1] | 77.1 [59.9 to 89.6] | 89.7 [75.8 to 97.1] | 76.3 [59.8 to 88.6] | 82.7 [72.2 to 90.4] | 89.2 [74.6 to 97.0] | 83.8 [68.0 to 93.8] | 88.9 [73.9 to 96.9] | 78.9 [62.7 to 90.4] | 89.7 [75.8 to 97.1] | 92.1 [78.6 to 98.3]

43. Secondary Outcome: Percentage of Participants With a Reciprocal HAI Titer ≥ 40 Specific for the HA Receptor Binding Domains of Vaccine Homologous Influenza B/Washington (Victoria Subtype) Expressed as SPR
Description: Percentage of participants with a reciprocal HAI titer ≥ 40 specific for the HA receptor binding domains of vaccine homologous Influenza B/Washington (Victoria Subtype) on Days 56, 70, and other follow-up time points.
Time Frame: Day 28 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Number (95% Confidence Interval); unit: percentage of participants(SPR)
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
percentage of participants(SPR)
  Day 28 | 97.5 [91.3 to 99.7] | 100.0 [91.2 to 100.0] | 97.4 [86.2 to 99.9] | 100.0 [90.5 to 100.0] | 95.1 [83.5 to 99.4] | 92.7 [80.1 to 98.5] | 96.2 [89.2 to 99.2] | 92.3 [79.1 to 98.4] | 94.9 [82.7 to 99.4] | 97.4 [86.5 to 99.9] | 94.9 [82.7 to 99.4] | 95.1 [83.5 to 99.4] | 97.4 [86.5 to 99.9]
  Day 56 | 98.7 [93.1 to 100.0] | 97.4 [86.5 to 99.9] | 91.7 [77.5 to 98.2] | 97.2 [85.5 to 99.9] | 90.0 [76.3 to 97.2] | 90.0 [76.3 to 97.2] | 97.5 [91.2 to 99.7] | 89.7 [75.8 to 97.1] | 97.4 [86.2 to 99.9] | 97.3 [85.8 to 99.9] | 94.7 [82.3 to 99.4] | 95.0 [83.1 to 99.4] | 97.4 [86.5 to 99.9]
  Day 70 | 98.7 [93.0 to 100.0] | 97.4 [86.5 to 99.9] | 97.1 [85.1 to 99.9] | 100.0 [90.3 to 100.0] | 92.5 [79.6 to 98.4] | 90.0 [76.3 to 97.2] | 98.7 [92.9 to 100.0] | 94.7 [82.3 to 99.4] | 94.7 [82.3 to 99.4] | 100.0 [90.3 to 100.0] | 94.6 [81.8 to 99.3] | 97.6 [87.1 to 99.9] | 97.4 [86.2 to 99.9]
  Day 84 | 83.3 [73.2 to 90.8] | 84.6 [69.5 to 94.1] | 79.4 [62.1 to 91.3] | 82.9 [66.4 to 93.6] | 82.1 [66.5 to 92.5] | 78.9 [62.7 to 90.4] | 85.5 [75.6 to 92.5] | 71.1 [54.1 to 84.6] | 73.7 [56.9 to 86.6] | 82.4 [65.5 to 93.2] | 91.9 [78.1 to 98.3] | 85.4 [70.8 to 94.4] | 78.9 [62.7 to 90.4]
  Day 182 | 82.7 [72.2 to 90.4] | 82.1 [66.5 to 92.5] | 76.5 [58.8 to 89.3] | 77.1 [59.9 to 89.6] | 79.5 [63.5 to 90.7] | 71.1 [54.1 to 84.6] | 82.7 [72.2 to 90.4] | 70.3 [53.0 to 84.1] | 81.1 [64.8 to 92.0] | 80.6 [64.0 to 91.8] | 73.7 [56.9 to 86.6] | 82.1 [66.5 to 92.5] | 78.9 [62.7 to 90.4]

44. Secondary Outcome: MN50 GMTs to the SARS-CoV-2 Wuhan Strain Expressed as Geometric Mean Titers (GMT)
Description: MN50 GMTs to the SARS-CoV-2 Wuhan Strain from the matched vaccine construct (and mismatched variant if available), at Days 0, 56, 70, and other follow-up time points.
Time Frame: Day 0 to Day 182
Population: Per Protocol Analysis Set population
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean titer
Groups:
- SARS-CoV-2 rS With Matrix-M1 Adjuvant: 2 doses of Formulation 14. 1 dose each on Days 0 and Day 56. ...
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | SARS-CoV-2 rS With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 40
geometric mean titer
  Day 0 | 127.7 [97.2 to 167.8] | 123.4 [75.5 to 201.6] | 112.1 [82.0 to 153.4] | 140.3 [105.3 to 187.1] | 126.3 [91.8 to 173.8] | 114.1 [79.6 to 163.5] | 158.6 [124.6 to 201.8] | 95.6 [69.9 to 130.6] | 124.8 [93.4 to 166.6] | 116.2 [83.6 to 161.5] | 136.3 [96.3 to 193.0] | 125.5 [87.5 to 180.0] | 106.3 [78.1 to 144.7]
  Day 28 | 476.7 [385.0 to 590.2] | 293.4 [188.3 to 457.4] | 377.1 [275.1 to 516.9] | 729.7 [536.6 to 992.2] | 378.9 [282.8 to 507.8] | 568.6 [419.1 to 771.4] | 331.7 [271.8 to 404.8] | 331.6 [239.4 to 459.3] | 356.0 [274.4 to 462.0] | 469.4 [353.4 to 623.4] | 245.1 [171.1 to 351.1] | 367.6 [262.3 to 515.1] | 617.7 [470.3 to 811.1]
  Day 56 | 328.5 [264.0 to 408.9] | 168.8 [110.2 to 258.5] | 290.6 [221.9 to 380.6] | 419.0 [316.1 to 555.4] | 259.9 [192.2 to 351.6] | 452.5 [315.1 to 649.9] | 232.4 [182.1 to 296.5] | 232.4 [167.2 to 323.1] | 226.3 [172.1 to 297.6] | 332.6 [237.6 to 465.4] | 169.0 [124.4 to 229.5] | 226.3 [168.9 to 303.2] | 432.9 [338.4 to 553.7]
  Day 70 | 554.2 [442.7 to 693.6] | 298.0 [223.9 to 396.7] | 430.7 [315.1 to 588.7] | 665.1 [524.5 to 843.4] | 407.9 [316.5 to 525.7] | 607.6 [462.8 to 797.6] | 286.4 [223.6 to 366.8] | 338.0 [246.6 to 463.2] | 292.1 [216.3 to 394.5] | 579.7 [405.8 to 828.1] | 224.2 [168.4 to 298.5] | 325.6 [245.7 to 431.5] | 956.0 [747.3 to 1223.1]
  Day 84 | 731.3 [580.5 to 921.2] | 403.2 [294.2 to 552.4] | 452.5 [364.4 to 562.1] | 932.4 [714.1 to 1217.5] | 535.8 [416.8 to 688.7] | 905.1 [674.7 to 1214.1] | 430.1 [347.0 to 533.2] | 478.0 [353.2 to 646.9] | 428.4 [333.0 to 551.2] | 518.8 [365.5 to 736.3] | 320.0 [239.9 to 426.9] | 460.5 [345.1 to 614.3] | 1280.0 [977.0 to 1676.9]
  Day 182 | 711.7 [501.7 to 1009.7] | 823.5 [498.3 to 1360.7] | 702.0 [447.8 to 1100.4] | 1000.9 [649.0 to 1543.6] | 535.5 [347.2 to 826.1] | 895.6 [604.0 to 1328.2] | 610.9 [421.0 to 886.4] | 721.2 [449.4 to 1157.5] | 699.9 [406.1 to 1206.1] | 752.4 [519.5 to 1089.6] | 503.9 [287.7 to 882.7] | 452.5 [248.6 to 823.7] | 1403.9 [940.5 to 2095.7]

45. Secondary Outcome: MN50 GMTs to the SARS-CoV-2 Omicron BA.1 Variant Expressed as GMT
Description: MN50 GMTs to the SARS-CoV-2 Omicron BA.1 Variant from the matched vaccine construct (and mismatched variant if available), at Days 0, 56, 70, and other follow-up time points.
Time Frame: Day 0 to Day 70
Population: Per Protocol Analysis Set population
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean titer
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | SARS-CoV-2 rS With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 40
geometric mean titer
  Day 0 | 10.7 [10.1 to 11.4] | 11.9 [9.3 to 15.3] | 10.2 [9.8 to 10.6] | 10.2 [9.8 to 10.6] | 10.3 [9.9 to 10.8] | 10.0 [10 to 10] | 10.8 [10.0 to 11.7] | 10.0 [10 to 10] | 10.7 [9.6 to 12.0] | 10.4 [9.9 to 10.9] | 10.4 [9.9 to 10.9] | 10.9 [9.4 to 12.6] | 10.7 [9.7 to 11.9]
  Day 28 | 17.0 [14.5 to 19.9] | 12.3 [9.8 to 15.4] | 13.1 [11.0 to 15.7] | 16.6 [13.7 to 20.1] | 12.9 [11.2 to 14.8] | 20.7 [15.7 to 27.3] | 12.4 [11.3 to 13.7] | 13.3 [10.9 to 16.2] | 12.4 [10.7 to 14.3] | 16.4 [12.6 to 21.3] | 11.1 [10.2 to 12.1] | 13.4 [11.1 to 16.2] | 19.0 [14.6 to 24.7]
  Day 56 | 15.0 [13.3 to 16.9] | 10.9 [9.4 to 12.7] | 13.3 [11.2 to 15.8] | 14.4 [11.8 to 17.6] | 12.3 [10.8 to 14.1] | 18.3 [15.0 to 22.4] | 11.7 [10.7 to 12.8] | 12.2 [10.7 to 13.8] | 11.8 [10.5 to 13.2] | 13.9 [11.3 to 17.0] | 10.6 [9.9 to 11.2] | 13.7 [11.3 to 16.6] | 15.6 [12.5 to 19.5]
  Day 70 | 24.2 [20.1 to 29.0] | 14.8 [12.1 to 18.0] | 19.6 [15.7 to 24.4] | 23.8 [18.1 to 31.2] | 17.1 [13.9 to 21.1] | 24.2 [18.7 to 31.3] | 15.4 [13.4 to 17.8] | 17.6 [13.8 to 22.4] | 15.8 [13.1 to 19.0] | 21.6 [16.0 to 29.3] | 13.2 [11.4 to 15.4] | 16.2 [13.3 to 19.9] | 36.5 [27.6 to 48.4]

46. Secondary Outcome: MN50 GMTs to the SARS-CoV-2 Wuhan Strain Expressed as Geometric Mean Fold Rise (GMFR)
Description: as for outcome 44
Time Frame: Day 28 to Day 182
Population: Per Protocol Analysis Set population
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean fold rise
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | SARS-CoV-2 rS With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 40
geometric mean fold rise
  Day 28 | 3.7 [3.1 to 4.6] | 2.4 [1.8 to 3.1] | 3.4 [2.6 to 4.4] | 5.2 [3.8 to 7.1] | 3.0 [2.1 to 4.3] | 5.0 [3.8 to 6.5] | 2.1 [1.8 to 2.5] | 3.5 [2.6 to 4.6] | 2.9 [2.2 to 3.7] | 4.1 [3.0 to 5.7] | 1.8 [1.3 to 2.5] | 2.9 [2.1 to 4.0] | 5.8 [4.3 to 7.9]
  Day 56 | 2.5 [2.0 to 3.2] | 1.5 [1.2 to 2.0] | 2.5 [1.8 to 3.3] | 3.0 [2.2 to 4.0] | 2.1 [1.6 to 2.9] | 3.7 [2.8 to 5.0] | 1.5 [1.2 to 1.8] | 2.4 [1.9 to 3.2] | 1.8 [1.4 to 2.5] | 3.0 [2.2 to 4.1] | 1.3 [0.9 to 1.8] | 1.8 [1.3 to 2.4] | 4.1 [3.0 to 5.4]
  Day 70 | 4.2 [3.2 to 5.4] | 2.7 [2.0 to 3.7] | 3.4 [2.5 to 4.6] | 4.8 [3.6 to 6.3] | 3.3 [2.4 to 4.5] | 5.0 [3.6 to 6.9] | 1.8 [1.5 to 2.2] | 3.5 [2.5 to 4.9] | 2.4 [1.7 to 3.3] | 5.5 [3.7 to 8.1] | 1.6 [1.2 to 2.2] | 2.6 [1.9 to 3.6] | 9.1 [6.5 to 12.6]
  Day 84 | 5.6 [4.4 to 7.1] | 3.7 [2.6 to 5.1] | 4.0 [3.0 to 5.3] | 6.8 [4.8 to 9.7] | 4.1 [2.9 to 5.9] | 7.4 [5.4 to 10.3] | 2.8 [2.2 to 3.5] | 5.0 [3.6 to 6.9] | 3.5 [2.4 to 5.0] | 4.8 [3.4 to 6.8] | 2.3 [1.8 to 2.9] | 3.7 [2.5 to 5.3] | 12.2 [8.8 to 16.8]
  Day 182 | 5.5 [3.9 to 7.8] | 6.0 [3.2 to 11.1] | 5.2 [3.1 to 8.7] | 7.2 [4.8 to 10.7] | 4.2 [2.5 to 7.1] | 7.4 [4.6 to 11.7] | 3.8 [2.6 to 5.6] | 7.4 [4.4 to 12.6] | 6.0 [3.4 to 10.4] | 7.0 [4.4 to 11.0] | 3.5 [2.0 to 6.2] | 3.3 [2.6 to 5.6] | 13.3 [8.0 to 22.2]

47. Secondary Outcome: MN50 GMTs to the SARS-CoV-2 Omicron BA.1 Variant Expressed as GMFR
Description: as for outcome 45
Time Frame: Day 28 to Day 70
Population: Per Protocol Analysis Set population
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean fold rise
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | SARS-CoV-2 rS With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 40
geometric mean fold rise
  Day 28 | 1.6 [1.4 to 1.8] | 1.0 [1.0 to 1.1] | 1.3 [1.1 to 1.5] | 1.6 [1.3 to 2.0] | 1.2 [1.1 to 1.4] | 2.1 [1.6 to 2.7] | 1.1 [1.1 to 1.2] | 1.3 [1.1 to 1.6] | 1.2 [1.0 to 1.3] | 1.6 [1.2 to 2.0] | 1.1 [1.0 to 1.2] | 1.2 [1.0 to 1.5] | 1.8 [1.4 to 2.2]
  Day 56 | 1.4 [1.3 to 1.5] | 1.0 [1.0 to 1.1] | 1.3 [1.1 to 1.5] | 1.4 [1.2 to 1.7] | 1.2 [1.0 to 1.4] | 1.8 [1.5 to 2.2] | 1.1 [1.0 to 1.2] | 1.2 [1.1 to 1.4] | 1.1 [1.0 to 1.2] | 1.3 [1.1 to 1.6] | 1.0 [1.0 to 1.1] | 1.3 [1.1 to 1.5] | 1.5 [1.2 to 1.8]
  Day 70 | 2.2 [1.9 to 2.7] | 1.4 [1.2 to 1.6] | 1.9 [1.5 to 2.4] | 2.3 [1.8 to 3.0] | 1.7 [1.3 to 2.0] | 2.4 [1.9 to 3.1] | 1.4 [1.2 to 1.6] | 1.8 [1.4 to 2.2] | 1.5 [1.2 to 1.7] | 2.1 [1.6 to 2.8] | 1.3 [1.1 to 1.5] | 1.5 [1.2 to 1.8] | 3.4 [2.5 to 4.5]

48. Secondary Outcome: MN50 GMTs to the SARS-CoV-2 Wuhan Strain Expressed as SCR
Description: as for outcome 44
Time Frame: Day 28 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | SARS-CoV-2 rS With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 40
Percentage of participants
  Day 28 | 67.5 [56.1 to 77.6] | 42.5 [27.0 to 59.1] | 55.3 [38.3 to 71.4] | 70.3 [53.0 to 84.1] | 41.5 [26.3 to 57.9] | 82.9 [67.9 to 92.8] | 36.4 [25.7 to 48.1] | 61.5 [44.6 to 76.6] | 51.3 [34.8 to 67.6] | 60.5 [43.4 to 76.0] | 28.2 [15.0 to 44.9] | 52.5 [36.1 to 68.5] | 76.9 [60.7 to 88.9]
  Day 56 | 44.3 [33.1 to 55.9] | 17.9 [7.5 to 33.5] | 44.4 [27.9 to 61.9] | 44.4 [27.9 to 61.9] | 37.5 [22.7 to 54.2] | 62.5 [45.8 to 77.3] | 23.1 [14.3 to 34.0] | 33.3 [19.1 to 50.2] | 28.9 [15.4 to 45.9] | 52.8 [35.5 to 69.6] | 10.5 [2.9 to 24.8] | 27.5 [14.6 to 43.9] | 61.5 [44.6 to 76.6]
  Day 70 | 64.9 [53.2 to 75.5] | 48.7 [32.4 to 65.2] | 54.3 [36.6 to 71.2] | 69.4 [51.9 to 83.7] | 52.5 [36.1 to 68.5] | 75.0 [58.8 to 87.3] | 29.3 [19.4 to 41.0] | 55.3 [38.3 to 71.4] | 39.5 [24.0 to 56.6] | 74.3 [56.7 to 87.5] | 29.7 [15.9 to 47.0] | 50.0 [33.8 to 66.2] | 86.8 [71.9 to 95.6]
  Day 84 | 75.6 [64.6 to 84.7] | 61.5 [44.6 to 76.6] | 67.6 [49.5 to 82.6] | 77.1 [59.9 to 89.6] | 53.8 [37.2 to 69.9] | 84.2 [68.7 to 94.0] | 52.0 [40.2 to 63.7] | 71.1 [54.1 to 84.6] | 52.6 [35.8 to 69.0] | 69.7 [51.3 to 84.4] | 35.1 [20.2 to 52.5] | 57.5 [40.9 to 73.0] | 94.7 [82.3 to 99.4]
  Day 182 | 69.4 [56.3 to 80.4] | 60.6 [42.1 to 77.1] | 66.7 [47.2 to 82.7] | 80.6 [62.5 to 92.5] | 54.3 [36.6 to 71.2] | 81.8 [64.5 to 93.0] | 56.7 [44.0 to 68.8] | 72.4 [52.8 to 87.3] | 67.7 [48.6 to 83.3] | 86.7 [69.3 to 96.2] | 65.5 [45.7 to 82.1] | 45.2 [27.3 to 64.0] | 86.7 [69.3 to 96.2]

49. Secondary Outcome: MN50 GMTs to the SARS-CoV-2 Omicron BA.1 Variant Expressed as SCR
Description: as for outcome 45
Time Frame: Day 28 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | SARS-CoV-2 rS With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 40
Percentage of participants
  Day 28 | 21.3 [12.9 to 31.8] | 0 [0.0 to 8.8] | 13.2 [4.4 to 28.1] | 21.6 [9.8 to 38.2] | 7.3 [1.5 to 19.9] | 29.3 [16.1 to 45.5] | 2.6 [0.3 to 9.1] | 12.8 [4.3 to 27.4] | 7.7 [1.6 to 20.9] | 21.1 [9.6 to 37.3] | 0 [0.0 to 9.0] | 15.0 [5.7 to 29.8] | 17.9 [7.5 to 33.5]
  Day 56 | 8.9 [3.6 to 17.4] | 0 [0.0 to 9.0] | 11.1 [3.1 to 26.1] | 16.7 [6.4 to 32.8] | 7.5 [1.6 to 20.4] | 22.5 [10.8 to 38.5] | 2.6 [0.3 to 9.0] | 5.1 [0.6 to 17.3] | 2.6 [0.1 to 13.8] | 13.9 [4.7 to 29.5] | 0 [0.0 to 9.3] | 10.0 [2.8 to 23.7] | 12.8 [4.3 to 27.4]
  Day 70 | 32.5 [22.2 to 44.1] | 10.3 [2.9 to 24.2] | 28.6 [14.6 to 46.3] | 41.7 [25.5 to 59.2] | 22.5 [10.8 to 38.5] | 45.0 [29.3 to 61.5] | 14.7 [7.6 to 24.7] | 23.7 [11.4 to 40.2] | 13.2 [4.4 to 28.1] | 31.4 [16.9 to 49.3] | 8.1 [1.7 to 21.9] | 17.5 [7.3 to 32.8] | 63.2 [46.0 to 78.2]

50. Secondary Outcome: MN50 GMTs to the SARS-CoV-2 Wuhan Strain Expressed as GMTR
Description: as for outcome 44
Time Frame: Day 28 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric mean titer ratio
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41
Geometric mean titer ratio
  Day 28 (Comparison to SARS-CoV-2 Reference [Group P]) | 0.70 [0.53 to 0.93] | 0.43 [0.30 to 0.61] | 0.60 [0.42 to 0.84] | 1.05 [0.73 to 1.51] | 0.58 [0.40 to 0.84] | 0.89 [0.64 to 1.23] | 0.44 [0.34 to 0.58] | 0.57 [0.40 to 0.81] | 0.54 [0.39 to 0.74] | 0.74 [0.52 to 1.05] | 0.35 [0.24 to 0.51] | 0.55 [0.38 to 0.79]
  Day 56 (Comparison to SARS-CoV-2 Reference [Group P]) | 0.69 [0.52 to 0.92] | 0.38 [0.27 to 0.53] | 0.64 [0.47 to 0.88] | 0.86 [0.62 to 1.20] | 0.56 [0.40 to 0.79] | 0.97 [0.68 to 1.38] | 0.42 [0.31 to 0.57] | 0.57 [0.41 to 0.79] | 0.49 [0.36 to 0.68] | 0.75 [0.53 to 1.06] | 0.36 [0.26 to 0.50] | 0.69 [0.52 to 0.92]
  Day 70 (Comparison to SARS-CoV-2 Reference [Group P]0) | 0.53 [0.39 to 0.73] | 0.31 [0.22 to 0.42] | 0.42 [0.29 to 0.60] | 0.64 [0.46 to 0.87] | 0.41 [0.29 to 0.56] | 0.61 [0.43 to 0.85] | 0.24 [0.17 to 0.34] | 0.36 [0.25 to 0.53] | 0.29 [0.20 to 0.42] | 0.61 [0.41 to 0.90] | 0.21 [0.15 to 0.30] | 0.53 [0.39 to 0.73]
  Day 84 (Comparison to SARS-CoV-2 Reference [Group P]) | 0.52 [0.38 to 0.72] | 0.31 [0.22 to 0.43] | 0.34 [0.25 to 0.47] | 0.67 [0.47 to 0.96] | 0.40 [0.28 to 0.56] | 0.67 [0.47 to 0.95] | 0.28 [0.21 to 0.39] | 0.39 [0.27 to 0.56] | 0.32 [0.23 to 0.46] | 0.40 [0.28 to 0.59] | 0.22 [0.16 to 0.30] | 0.34 [0.24 to 0.49]
  Day 182 (Comparison to SARS-CoV-2 Reference [Group P]) | 0.47 [0.27 to 0.80] | 0.56 [0.30 to 1.07] | 0.48 [0.27 to 0.87] | 0.64 [0.37 to 1.13] | 0.37 [0.21 to 0.67] | 0.62 [0.36 to 1.06] | 0.38 [0.21 to 0.69] | 0.52 [0.29 to 0.95] | 0.48 [0.25 to 0.93] | 0.53 [0.32 to 0.90] | 0.32 [0.17 to 0.62] | 0.28 [0.15 to 0.52]

51. Secondary Outcome: MN50 GMTs to the SARS-CoV-2 Omicron BA.1 Expressed as GMTR
Description: MN50 GMTs to the SARS-CoV-2 Omicron BA.1 from the matched vaccine construct (and mismatched variant if available), at Days 0, 56, 70, and other follow-up time points.
Time Frame: Day 28 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric mean titer ratio
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41
Geometric mean titer ratio
  Day 28 (Comparison to SARS-CoV-2 Reference [Group P]) | 0.90 [0.69 to 1.17] | 0.59 [0.46 to 0.76] | 0.73 [0.54 to 0.99] | 0.93 [0.68 to 1.26] | 0.71 [0.54 to 0.92] | 1.18 [0.81 to 1.71] | 0.65 [0.53 to 0.79] | 0.76 [0.55 to 1.04] | 0.65 [0.50 to 0.86] | 0.91 [0.65 to 1.27] | 0.61 [0.47 to 0.78] | 0.70 [0.52 to 0.93]
  Day 56 (Comparison to SARS-CoV-2 Reference [Group P]) | 0.96 [0.78 to 1.18] | 0.70 [0.57 to 0.87] | 0.89 [0.68 to 1.17] | 0.96 [0.72 to 1.28] | 0.81 [0.64 to 1.03] | 1.24 [0.92 to 1.66] | 0.75 [0.63 to 0.90] | 0.82 [0.64 to 1.05] | 0.75 [0.60 to 0.96] | 0.92 [0.70 to 1.21] | 0.70 [0.56 to 0.86] | 0.87 [0.67 to 1.13]
  Day 70 (Comparison to SARS-CoV-2 Reference [Group P]0) | 0.66 [0.48 to 0.91] | 0.41 [0.30 to 0.56] | 0.55 [0.38 to 0.78] | 0.67 [0.45 to 0.98] | 0.48 [0.34 to 0.67] | 0.42 [0.32 to 0.55] | 0.75 [0.63 to 0.90] | 0.49 [0.34 to 0.72] | 0.43 [0.31 to 0.60] | 0.61 [0.41 to 0.91] | 0.37 [0.27 to 0.50] | 0.44 [0.32 to 0.61]

52. Secondary Outcome: Microneutralization (MN50) Antibody Responses Specific to Vaccine Homologous Wild-type Influenza A/Brisbane (H1N1 Subtype) Expressed as GMT
Description: Microneutralization (MN50) antibody responses: neutralizing antibody titers specific to vaccine homologous wild-type Influenza A/Brisbane (H1N1 Subtype) and/or antigenically-drifted influenza strains, as measured by an MN assay, expressed as GMT.
Time Frame: Day 0 to Day 182
Population: Per Protocol Analysis Set population
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean titer
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
geometric mean titer
  Day 0 | 844.5 [593.8 to 1200.9] | 561.5 [350.8 to 898.9] | 737.2 [467.1 to 1163.5] | 737.0 [443.4 to 1225.0] | 723.6 [453.9 to 1153.6] | 865.1 [528.4 to 1416.4] | 746.4 [515.7 to 1080.5] | 806.4 [462.7 to 1405.3] | 794.3 [473.6 to 1332.2] | 837.0 [501.5 to 1396.8] | 1197.5 [678.2 to 2114.6] | 761.1 [493.8 to 1173.2] | 923.8 [524.3 to 1627.7]
  Day 28 | 1597.5 [1225.6 to 2082.1] | 1043.8 [692.5 to 1573.3] | 1099.4 [796.1 to 1518.3] | 1065.2 [689.3 to 1646.0] | 1225.2 [833.6 to 1800.6] | 1088.6 [744.0 to 1592.8] | 1426.2 [1042.0 to 1952.2] | 1102.0 [685.5 to 1771.7] | 971.8 [629.8 to 1499.4] | 1426.2 [858.4 to 2228.9] | 1617.1 [1012.2 to 2583.6] | 1173.6 [839.5 to 1640.8] | 1935.2 [1278.7 to 2929.0]
  Day 56 | 1503.2 [1148.5 to 1967.5] | 947.1 [607.6 to 1476.4] | 1078.1 [772.7 to 1504.0] | 1000.7 [632.7 to 1582.8] | 1514.7 [733.9 to 1616.7] | 952.5 [632.1 to 1435.2] | 1139.6 [829.2 to 1566.1] | 954.7 [598.4 to 1523.2] | 831.2 [536.6 to 1287.7] | 1229.2 [750.0 to 2014.5] | 1514.7 [952.2 to 2409.5] | 1093.0 [775.8 to 1539.8] | 1637.7 [1018.5 to 2633.5]
  Day 70 | 2022.0 [1538.7 to 2656.9] | 1462.2 [995.2 to 2148.6] | 1482.5 [1079.9 to 2035.3] | 1768.3 [1219.8 to 2563.3] | 1750.8 [1213.7 to 2525.8] | 1316.3 [916.8 to 1889.8] | 1570.6 [1158.4 to 2129.4] | 1463.6 [971.7 to 2204.6] | 1062.2 [695.6 to 1622.1] | 1756.8 [1134.3 to 2720.9] | 2095.7 [1346.2 to 3262.4] | 1600.4 [1164.6 to 2199.3] | 1381.8 [894.1 to 2135.6]
  Day 84 | 4673.3 [3529.7 to 6187.4] | 3767.7 [2509.4 to 5656.7] | 3539.2 [2480.9 to 5049.0] | 3530.8 [2308.5 to 5400.3] | 4025.5 [2712.5 to 5974.2] | 2248.0 [1478.4 to 3418.2] | 3979.8 [2961.8 to 5347.8] | 3938.5 [2499.2 to 6206.5] | 2636.7 [1774.8 to 3917.4] | 5100.1 [3166.7 to 8213.9] | 4844.1 [3089.4 to 7595.6] | 3887.2 [2577.5 to 5862.3] | 3576.7 [2299.3 to 5563.7]
  Day 182 | 3339.6 [2470.1 to 4515.3] | 2097.3 [1424.6 to 3087.6] | 2368.2 [1634.0 to 3432.5] | 2287.1 [1526.9 to 3425.8] | 2646.0 [1739.3 to 4025.4] | 1882.2 [1169.0 to 3030.5] | 2846.0 [2099.5 to 3857.9] | 2341.7 [1486.1 to 3689.9] | 1660.1 [1062.9 to 2592.8] | 3172.3 [1940.1 to 5187.0] | 2407.0 [1310.2 to 4421.9] | 2684.6 [1789.3 to 4027.8] | 2849.4 [1747.4 to 4646.5]

53. Secondary Outcome: Microneutralization (MN50) Antibody Responses Specific to Vaccine Homologous Wild-type Influenza A/Kansas (H3N2 Subtype) Expressed as GMT
Description: Microneutralization (MN50) antibody responses: neutralizing antibody titers specific to vaccine homologous wild-type Influenza A/Kansas (H3N2 Subtype) and/or antigenically-drifted influenza strains, as measured by an MN assay, expressed as GMT.
Time Frame: Day 0 to Day 182
Population: Per Protocol Analysis Set population
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean titer
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
geometric mean titer
  Day 0 | 184.4 [144.2 to 235.8] | 220.6 [153.2 to 317.4] | 153.5 [98.9 to 238.2] | 178.9 [126.7 to 252.5] | 177.5 [130.4 to 241.7] | 203.9 [142.7 to 291.3] | 185.3 [148.8 to 230.8] | 185.7 [123.0 to 280.4] | 276.6 [181.4 to 422.0] | 156.4 [114.1 to 214.4] | 220.0 [154.4 to 313.5] | 218.2 [158.2 to 301.0] | 162.5 [105.9 to 249.4]
  Day 28 | 794.0 [615.3 to 1024.5] | 749.1 [416.2 to 1348.3] | 416.9 [272.4 to 638.1] | 550.5 [370.5 to 817.9] | 654.0 [441.1 to 969.9] | 583.6 [414.4 to 821.9] | 764.3 [577.2 to 1012.0] | 461.8 [318.7 to 669.0] | 607.2 [399.6 to 922.7] | 713.9 [577.2 to 1012.0] | 790.6 [521.2 to 1199.2] | 781.7 [524.9 to 1164.2] | 1013.1 [714.1 to 1437.1]
  Day 56 | 682.7 [531.1 to 877.5] | 613.1 [339.6 to 1106.7] | 416.9 [272.4 to 638.1] | 550.5 [370.5 to 817.9] | 654.0 [441.1 to 969.9] | 583.6 [414.4 to 821.9] | 764.3 [577.2 to 1012.0] | 394.5 [273.2 to 569.7] | 561.4 [368.2 to 856.0] | 544.4 [359.7 to 823.8] | 650.7 [419.5 to 1009.3] | 688.7 [464.4 to 1021.2] | 788.9 [552.7 to 1126.0]
  Day 70 | 917.5 [754.7 to 1115.3] | 922.9 [534.9 to 1592.2] | 588.6 [392.8 to 882.1] | 812.2 [573.8 to 1149.6] | 736.1 [537.4 to 1008.3] | 722.8 [500.4 to 1044.1] | 899.2 [705.9 to 1145.3] | 614.5 [443.2 to 852.0] | 772.9 [525.0 to 1137.9] | 691.4 [455.9 to 1048.5] | 884.9 [608.1 to 1287.7] | 866.1 [605.8 to 1238.2] | 747.7 [519.9 to 1075.3]
  Day 84 | 874.0 [717.5 to 1064.5] | 810.7 [475.0 to 1383.9] | 617.5 [408.6 to 933.2] | 664.6 [457.6 to 965.4] | 802.3 [560.7 to 1148.0] | 637.5 [431.8 to 941.1] | 907.2 [727.8 to 1130.9] | 681.8 [487.6 to 953.5] | 768.0 [537.2 to 1098.1] | 714.4 [470.5 to 1084.8] | 865.7 [608.7 to 1231.1] | 902.3 [629.0 to 1294.3] | 754.5 [515.2 to 1104.7]
  Day 182 | 611.6 [487.9 to 766.6] | 520.7 [315.5 to 859.2] | 339.1 [224.4 to 512.4] | 449.5 [308.6 to 654.9] | 539.1 [384.3 to 756.2] | 436.4 [301.2 to 632.4] | 563.7 [444.7 to 714.7] | 415.6 [296.7 to 582.0] | 528.7 [372.2 to 751.0] | 486.3 [328.4 to 720.2] | 497.1 [344.6 to 717.0] | 547.9 [376.6 to 797.1] | 510.1 [356.1 to 730.6]

54. Secondary Outcome: Microneutralization (MN50) Antibody Responses Specific to Vaccine Homologous Wild-type Influenza A/Wisconsin (H1N1 Subtype) Expressed as GMT
Description: Microneutralization (MN50) antibody responses: neutralizing antibody titers specific to vaccine homologous wild-type Influenza A/Wisconsin (H1N1 Subtype) and/or antigenically-drifted influenza strains, as measured by an MN assay, expressed as GMT.
Time Frame: Day 0 to Day 182
Population: Per Protocol Analysis Set population
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean titer
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
geometric mean titer
  Day 0 | 88.8 [66.5 to 118.7] | 64.3 [53.4 to 99.0] | 56.0 [43.2 to 74.6] | 71.9 [54.0 to 100.8] | 74.9 [55.2 to 111.4] | 74.9 [55.2 to 117.3] | 80.5 [69.6 to 126.0] | 84.3 [50.6 to 123.6] | 87.2 [52.9 to 110.4] | 76.7 [74.6 to 150.7] | 95.5 [61.4 to 152.7] | 71.8 [49.7 to 103.7] | 99.8 [64.7 to 153.8]
  Day 28 | 103.9 [78.6 to 137.2] | 72.7 [53.4 to 99.0] | 56.7 [43.2 to 74.6] | 73.8 [54.0 to 100.8] | 78.4 [55.2 to 111.4] | 80.4 [55.2 to 117.3] | 93.7 [69.6 to 126.0] | 79.1 [50.6 to 123.6] | 76.4 [52.9 to 110.4] | 106.0 [74.6 to 150.7] | 96.8 [61.4 to 152.7] | 79.0 [54.2 to 115.1] | 112.5 [73.4 to 172.4]
  Day 56 | 95.3 [72.7 to 125.1] | 68.0 [50.6 to 91.5] | 58.2 [43.6 to 77.7] | 67.5 [50.1 to 91.1] | 73.4 [51.7 to 104.3] | 68.9 [48.1 to 98.8] | 78.9 [59.9 to 104.0] | 76.0 [49.9 to 115.9] | 69.5 [49.5 to 97.5] | 87.9 [62.5 to 123.6] | 85.0 [54.1 to 133.6] | 77.4 [53.4 to 112.4] | 106.7 [69.2 to 164.4]
  Day 70 | 122.6 [92.2 to 163.1] | 78.1 [56.1 to 108.8] | 74.4 [54.3 to 102.1] | 96.3 [68.9 to 134.8] | 97.5 [65.8 to 144.3] | 77.2 [53.0 to 112.5] | 102.7 [75.8 to 139.0] | 90.5 [58.3 to 140.4] | 74.6 [52.5 to 105.9] | 114.8 [81.0 to 162.6] | 113.3 [73.2 to 175.3] | 94.0 [64.7 to 136.7] | 109.8 [71.8 to 168.1]
  Day 84 | 135.6 [102.8 to 178.9] | 87.5 [62.9 to 121.8] | 87.1 [61.6 to 123.2] | 100.0 [70.4 to 142.0] | 115.5 [76.9 to 173.3] | 79.9 [54.8 to 116.5] | 115.9 [85.1 to 157.9] | 101.8 [64.7 to 160.2] | 81.1 [57.1 to 115.1] | 154.7 [101.0 to 236.8] | 129.5 [82.1 to 204.3] | 113.6 [76.8 to 168.0] | 126.1 [81.4 to 195.4]
  Day 182 | 97.4 [74.8 to 126.7] | 66.0 [50.0 to 87.3] | 64.6 [47.6 to 87.6] | 81.1 [59.0 to 111.6] | 86.3 [58.0 to 128.5] | 68.9 [47.3 to 100.2] | 92.9 [68.9 to 125.1] | 80.1 [51.8 to 123.8] | 66.3 [48.2 to 91.3] | 115.3 [81.2 to 163.8] | 95.8 [62.0 to 148.1] | 89.9 [62.6 to 129.3] | 104.1 [67.2 to 161.4]

55. Secondary Outcome: Microneutralization (MN50) Antibody Responses Specific to Vaccine Homologous Wild-type Influenza A/Cambodia (H3N2 Subtype) Expressed as GMT
Description: Microneutralization (MN50) antibody responses: neutralizing antibody titers specific to vaccine homologous wild-type Influenza A/Cambodia (H3N2 Subtype) and/or antigenically-drifted influenza strains, as measured by an MN assay, expressed as GMT.
Time Frame: Day 0 to Day 182
Population: Per Protocol Analysis Set population
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean titer
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
geometric mean titer
  Day 0 | 29.1 [24.9 to 33.9] | 31.6 [25.7 to 38.9] | 29.0 [21.8 to 38.4] | 30.3 [23.2 to 39.4] | 28.4 [22.6 to 35.7] | 30.8 [23.5 to 40.5] | 26.7 [22.4 to 31.7] | 32.7 [23.9 to 44.8] | 27.5 [21.0 to 36.1] | 24.6 [19.0 to 32.1] | 30.6 [23.1 to 40.5] | 24.2 [19.6 to 29.8] | 28.5 [22.1 to 36.8]
  Day 28 | 56.5 [44.6 to 71.4] | 64.3 [39.9 to 103.8] | 43.7 [30.4 to 62.7] | 50.8 [36.1 to 71.4] | 61.6 [41.4 to 91.8] | 45.9 [33.5 to 62.8] | 48.4 [37.5 to 62.5] | 45.2 [31.4 to 64.9] | 40.5 [28.5 to 57.5] | 63.4 [42.3 to 95.1] | 59.4 [39.2 to 89.8] | 39.2 [27.4 to 56.2] | 51.2 [36.9 to 70.9]
  Day 56 | 51.1 [40.9 to 63.9] | 56.9 [35.2 to 91.9] | 42.1 [28.9 to 61.3] | 45.7 [33.0 to 63.5] | 46.6 [32.2 to 67.5] | 40.7 [29.7 to 55.8] | 43.3 [34.2 to 54.9] | 41.3 [28.6 to 59.6] | 37.8 [26.1 to 54.6] | 49.7 [33.0 to 74.8] | 51.6 [35.2 to 75.7] | 36.5 [26.4 to 50.5] | 42.9 [30.9 to 59.5]
  Day 70 | 57.8 [46.1 to 72.3] | 71.2 [43.9 to 115.2] | 51.7 [34.6 to 77.2] | 56.6 [40.1 to 79.8] | 63.2 [43.6 to 91.5] | 50.8 [35.6 to 72.4] | 51.9 [40.3 to 66.8] | 51.0 [34.7 to 75.0] | 43.5 [29.9 to 63.2] | 55.6 [35.6 to 86.6] | 63.1 [42.2 to 94.4] | 43.1 [30.6 to 60.7] | 39.5 [28.3 to 54.9]
  Day 84 | 51.4 [40.9 to 64.7] | 64.5 [39.7 to 104.8] | 49.3 [32.7 to 74.4] | 54.5 [38.9 to 76.4] | 54.7 [36.8 to 81.3] | 44.6 [30.5 to 65.4] | 45.9 [35.8 to 58.7] | 48.9 [33.4 to 71.7] | 41.9 [28.7 to 61.2] | 66.4 [42.0 to 104.8] | 62.4 [42.0 to 92.9] | 39.3 [28.3 to 54.5] | 39.0 [28.8 to 52.9]
  Day 182 | 40.4 [32.7 to 50.0] | 48.2 [30.6 to 76.0] | 38.6 [26.8 to 55.5] | 42.1 [31.0 to 57.1] | 40.5 [28.5 to 57.6] | 37.1 [25.3 to 54.3] | 35.5 [28.4 to 44.4] | 39.6 [27.2 to 57.6] | 32.9 [23.0 to 47.2] | 44.7 [29.7 to 67.3] | 45.9 [31.9 to 65.9] | 32.2 [24.1 to 43.1] | 34.6 [25.8 to 46.2]

56. Secondary Outcome: Microneutralization (MN50) Antibody Responses Specific to Vaccine Homologous Wild-type Influenza A/Hong Kong (H3N2 Subtype) Expressed as GMT
Description: Microneutralization (MN50) antibody responses: neutralizing antibody titers specific to vaccine homologous wild-type Influenza A/Hong Kong (H3N2 Subtype) and/or antigenically-drifted influenza strains, as measured by an MN assay, expressed as GMT.
Time Frame: Day 0 to Day 182
Population: Per Protocol Analysis Set population
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean titer
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
geometric mean titer
  Day 0 | 74.6 [57.1 to 97.5] | 64.4 [43.3 to 95.8] | 64.4 [40.6 to 102.2] | 60.9 [40.6 to 91.4] | 67.3 [45.5 to 99.7] | 77.0 [48.4 to 122.4] | 57.0 [43.7 to 74.5] | 69.6 [44.3 to 109.3] | 71.1 [43.5 to 116.3] | 50.0 [33.4 to 74.8] | 89.4 [55.8 to 143.4] | 55.9 [37.9 to 82.5] | 68.7 [44.4 to 106.2]
  Day 28 | 162.5 [120.4 to 219.5] | 167.7 [86.8 to 324.2] | 113.1 [67.5 to 189.5] | 123.0 [77.9 to 194.3] | 154.2 [89.9 to 264.5] | 141.7 [88.8 to 226.2] | 152.9 [111.7 to 209.5] | 110.7 [70.6 to 173.5] | 136.1 [79.6 to 232.8] | 157.2 [96.6 to 256.1] | 209.5 [117.4 to 373.6] | 128.7 [81.1 to 204.2] | 165.8 [105.5 to 260.5]
  Day 56 | 141.2 [104.5 to 190.6] | 141.8 [74.7 to 269.2] | 100.6 [59.6 to 169.8] | 102.6 [64.1 to 164.4] | 116.7 [70.7 to 192.8] | 120.8 [75.8 to 192.4] | 120.2 [86.7 to 166.5] | 98.4 [64.2 to 150.9] | 128.4 [74.1 to 222.6] | 112.3 [68.3 to 184.6] | 182.5 [104.0 to 320.4] | 104.6 [65.9 to 165.9] | 135.9 [85.4 to 216.2]
  Day 70 | 174.2 [129.6 to 234.2] | 194.0 [100.7 to 373.8] | 145.0 [87.3 to 240.6] | 139.8 [89.8 to 217.7] | 165.5 [99.9 to 274.3] | 163.2 [101.1 to 263.4] | 160.0 [117.2 to 218.3] | 129.3 [81.9 to 204.1] | 155.5 [92.0 to 262.7] | 129.7 [78.6 to 214.0] | 225.9 [129.2 to 395.0] | 142.6 [90.6 to 224.5] | 133.6 [81.8 to 218.3]
  Day 84 | 154.8 [114.2 to 209.7] | 202.2 [106.1 to 385.5] | 143.1 [84.6 to 241.9] | 130.0 [82.2 to 205.7] | 157.2 [94.2 to 262.4] | 143.5 [84.8 to 242.9] | 150.2 [110.5 to 204.1] | 144.5 [90.3 to 231.3] | 161.5 [96.4 to 270.5] | 150.9 [92.2 to 246.9] | 212.1 [121.4 to 370.7] | 130.0 [82.3 to 205.5] | 122.4 [76.9 to 194.8]
  Day 182 | 113.5 [82.3 to 156.6] | 138.0 [74.8 to 254.5] | 92.7 [55.1 to 156.0] | 101.2 [64.2 to 159.6] | 119.3 [71.7 to 198.5] | 109.3 [67.2 to 177.8] | 98.5 [72.1 to 134.5] | 101.9 [65.5 to 158.5] | 118.3 [70.0 to 199.8] | 102.5 [62.7 to 167.6] | 134.7 [78.8 to 230.3] | 103.2 [65.3 to 163.2] | 101.4 [65.0 to 158.1]

57. Secondary Outcome: Microneutralization (MN50) Antibody Responses Specific to Vaccine Homologous Wild-type Influenza B/Phuket (Yamagata Subtype) Expressed as GMT
Description: Microneutralization (MN50) antibody responses: neutralizing antibody titers specific to vaccine homologous wild-type Influenza B/Phuket (Yamagata Subtype) and/or antigenically-drifted influenza strains, as measured by an MN assay, expressed as GMT.
Time Frame: Day 0 to Day 182
Population: Per Protocol Analysis Set population
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean titer
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
geometric mean titer
  Day 0 | 69.4 [57.9 to 83.2] | 76.9 [57.7 to 102.5] | 57.8 [44.0 to 75.9] | 65.0 [50.0 to 84.7] | 60.8 [49.0 to 75.3] | 69.9 [53.5 to 91.2] | 61.3 [52.5 to 71.6] | 66.4 [53.1 to 83.1] | 62.1 [48.7 to 79.1] | 69.0 [53.7 to 88.5] | 67.6 [52.6 to 86.9] | 63.0 [49.1 to 80.9] | 65.2 [50.8 to 83.5]
  Day 28 | 118.4 [95.0 to 147.5] | 97.7 [70.7 to 134.9] | 63.3 [48.5 to 82.4] | 79.7 [59.1 to 107.6] | 97.5 [69.0 to 137.7] | 87.8 [66.9 to 115.3] | 89.6 [74.0 to 108.4] | 85.1 [65.6 to 110.5] | 73.1 [57.1 to 93.6] | 111.9 [82.4 to 152.1] | 89.9 [66.9 to 120.9] | 99.0 [71.5 to 136.9] | 111.5 [83.8 to 148.4]
  Day 56 | 110.2 [87.4 to 138.9] | 86.4 [62.5 to 119.4] | 63.0 [47.7 to 83.1] | 76.3 [56.3 to 103.3] | 89.9 [63.1 to 127.9] | 84.2 [64.7 to 109.6] | 81.3 [67.5 to 98.0] | 79.4 [61.7 to 102.4] | 70.0 [54.5 to 89.9] | 92.8 [66.5 to 129.6] | 84.2 [61.7 to 114.8] | 91.5 [66.3 to 126.3] | 102.0 [75.8 to 137.3]
  Day 70 | 132.3 [105.0 to 166.7] | 110.8 [78.5 to 156.2] | 73.9 [54.7 to 100.0] | 100.3 [73.0 to 137.8] | 118.6 [84.6 to 166.2] | 95.5 [71.1 to 128.2] | 96.0 [77.8 to 118.5] | 98.3 [75.5 to 127.9] | 82.3 [62.7 to 108.1] | 135.9 [97.3 to 189.9] | 93.4 [67.8 to 128.8] | 109.8 [79.5 to 151.6] | 95.3 [71.3 to 127.4]
  Day 84 | 195.6 [155.4 to 246.2] | 137.8 [97.4 to 194.9] | 120.1 [89.5 to 161.2] | 143.5 [101.7 to 202.6] | 159.5 [115.2 to 220.7] | 117.2 [87.0 to 157.9] | 144.9 [117.7 to 178.4] | 135.9 [102.7 to 179.8] | 120.7 [89.8 to 162.1] | 187.7 [125.0 to 282.0] | 129.6 [92.6 to 181.5] | 187.5 [133.9 to 262.6] | 135.0 [103.6 to 176.0]
  Day 182 | 158.7 [125.9 to 200.2] | 100.0 [72.1 to 138.8] | 83.0 [60.1 to 114.8] | 121.0 [85.8 to 170.7] | 125.7 [92.2 to 171.4] | 96.3 [72.8 to 127.3] | 108.4 [87.9 to 133.7] | 101.4 [77.6 to 132.5] | 91.9 [69.5 to 121.6] | 142.5 [99.2 to 204.7] | 106.2 [79.5 to 142.0] | 128.1 [92.6 to 177.3] | 118.3 [90.3 to 155.1]

58. Secondary Outcome: Microneutralization (MN50) Antibody Responses Specific to Vaccine Homologous Wild-type Influenza B/Maryland (Victoria Subtype) Expressed as GMT
Description: Microneutralization (MN50) antibody responses: neutralizing antibody titers specific to vaccine homologous wild-type Influenza B/Maryland (Victoria Subtype) and/or antigenically-drifted influenza strains, as measured by an MN assay, expressed as GMT.
Time Frame: Day 0 to Day 182
Population: Per Protocol Analysis Set population
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean titer
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
geometric mean titer
  Day 0 | 153.4 [127.0 to 185.3] | 153.1 [113.5 to 206.4] | 136.2 [103.3 to 179.7] | 125.9 [93.7 to 169.1] | 145.0 [114.3 to 183.9] | 148.2 [115.9 to 189.4] | 163.7 [138.0 to 194.2] | 167.2 [128.2 to 218.1] | 162.5 [123.5 to 213.9] | 176.9 [132.4 to 236.4] | 152.1 [121.2 to 191.0] | 148.6 [111.5 to 198.0] | 129.4 [97.4 to 171.8]
  Day 28 | 265.9 [225.4 to 313.7] | 236.3 [178.5 to 312.9] | 173.3 [130.1 to 230.8] | 183.1 [130.7 to 256.6] | 249.0 [196.9 to 314.9] | 184.7 [148.1 to 230.3] | 270.0 [226.9 to 321.1] | 207.8 [165.9 to 260.3] | 196.5 [151.3 to 255.4] | 261.9 [199.1 to 344.6] | 229.4 [177.4 to 296.7] | 218.7 [168.1 to 284.6] | 280.6 [215.8 to 364.7]
  Day 56 | 242.3 [205.0 to 286.5] | 209.6 [157.2 to 279.5] | 168.8 [128.1 to 222.2] | 165.3 [119.9 to 227.8] | 215.9 [173.0 to 269.4] | 179.1 [142.0 to 225.9] | 243.7 [204.8 to 290.1] | 197.1 [157.0 to 247.4] | 193.0 [149.1 to 249.7] | 236.4 [182.1 to 307.0] | 210.9 [161.2 to 275.8] | 205.6 [155.7 to 271.5] | 246.7 [182.8 to 333.0]
  Day 70 | 284.8 [239.2 to 339.0] | 266.5 [198.8 to 357.1] | 194.0 [149.1 to 252.6] | 199.4 [144.1 to 276.0] | 267.4 [213.7 to 334.7] | 203.2 [162.8 to 253.8] | 274.2 [229.9 to 326.9] | 209.2 [158.6 to 275.8] | 212.9 [164.6 to 275.3] | 271.3 [198.5 to 370.7] | 242.7 [188.6 to 312.4] | 245.1 [192.1 to 312.7] | 219.4 [163.6 to 294.2]
  Day 84 | 508.5 [425.0 to 608.4] | 396.5 [288.0 to 546.1] | 330.6 [245.8 to 444.7] | 364.4 [265.1 to 500.8] | 390.7 [298.3 to 511.7] | 310.1 [238.6 to 403.0] | 464.3 [383.2 to 562.5] | 365.9 [274.7 to 487.4] | 335.4 [249.0 to 451.7] | 521.9 [362.2 to 752.1] | 381.4 [271.2 to 536.3] | 477.2 [350.6 to 649.7] | 364.1 [261.8 to 506.4]
  Day 182 | 433.4 [359.3 to 522.7] | 300.7 [221.0 to 409.2] | 267.3 [197.4 to 361.9] | 302.6 [219.1 to 417.8] | 302.7 [235.7 to 388.9] | 278.6 [215.6 to 360.1] | 384.4 [311.2 to 474.8] | 272.3 [206.5 to 359.0] | 284.5 [208.8 to 387.8] | 407.3 [301.5 to 550.3] | 306.6 [220.2 to 426.8] | 337.3 [250.6 to 453.9] | 312.4 [226.0 to 431.8]

59. Secondary Outcome: Microneutralization (MN50) Antibody Responses Specific to Vaccine Homologous Wild-type Influenza B/Washington (Victoria Subtype)Expressed as GMT
Description: Microneutralization (MN50) antibody responses: neutralizing antibody titers specific to vaccine homologous wild-type Influenza B/Washington (Victoria Subtype) and/or antigenically-drifted influenza strains, as measured by an MN assay, expressed as GMT.
Time Frame: Day 0 to Day 182
Population: Per Protocol Analysis Set population
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean titer
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
geometric mean titer
  Day 0 | 155.0 [125.0 to 192.2] | 131.8 [91.6 to 189.6] | 148.6 [106.0 to 208.2] | 131.1 [95.5 to 179.9] | 136.5 [97.9 to 190.1] | 143.9 [112.5 to 184.2] | 149.2 [120.6 to 189.0] | 158.6 [112.4 to 223.8] | 131.6 [96.2 to 179.9] | 173.0 [120.6 to 248.0] | 147.1 [106.1 to 204.1] | 148.8 [102.1 to 216.6] | 124.4 [91.4 to 169.4]
  Day 28 | 269.6 [220.9 to 328.9] | 221.3 [160.1 to 306.0] | 177.5 [130.7 to 241.0] | 210.5 [150.9 to 293.6] | 242.5 [175.4 to 335.3] | 194.5 [149.1 to 253.8] | 252.7 [202.8 to 314.9] | 206.7 [149.4 to 286.1] | 161.9 [117.8 to 222.5] | 246.3 [175.7 to 345.3] | 239.2 [170.1 to 336.4] | 219.0 [157.1 to 305.2] | 282.0 [199.5 to 398.8]
  Day 56 | 245.2 [200.4 to 299.9] | 191.9 [137.1 to 268.5] | 168.2 [120.4 to 234.8] | 180.9 [132.4 to 247.1] | 204.2 [148.7 to 280.4] | 180.7 [136.9 to 238.5] | 223.3 [179.4 to 277.8] | 184.3 [132.3 to 256.7] | 162.9 [118.7 to 223.5] | 215.2 [156.4 to 296.0] | 225.3 [160.2 to 316.8] | 214.6 [145.3 to 316.8] | 238.1 [171.4 to 331.0]
  Day 70 | 285.7 [232.5 to 351.2] | 238.8 [167.9 to 339.7] | 199.8 [147.8 to 270.1] | 217.7 [157.1 to 301.9] | 250.5 [181.4 to 345.8] | 210.8 [161.9 to 274.4] | 250.9 [202.5 to 310.9] | 204.3 [146.3 to 285.4] | 183.9 [132.1 to 256.1] | 246.1 [171.9 to 352.2] | 253.9 [193.1 to 333.9] | 237.1 [173.8 to 323.3] | 285.7 [232.5 to 351.2]
  Day 84 | 297.3 [245.1 to 360.7] | 240.2 [171.1 to 337.3] | 236.2 [177.6 to 314.2] | 259.5 [189.5 to 355.2] | 259.0 [180.2 to 372.2] | 200.4 [149.2 to 269.2] | 270.6 [218.8 to 334.5] | 217.8 [159.3 to 297.9] | 216.5 [155.9 to 300.7] | 320.5 [226.0 to 454.5] | 280.0 [197.0 to 398.0] | 268.8 [193.8 to 372.8] | 241.5 [169.7 to 343.8]
  Day 182 | 247.3 [200.0 to 305.8] | 178.3 [129.2 to 246.1] | 176.1 [127.1 to 244.0] | 219.9 [159.2 to 303.6] | 192.1 [135.6 to 272.1] | 176.6 [132.6 to 235.1] | 235.9 [188.3 to 295.7] | 173.5 [127.0 to 236.9] | 179.4 [128.2 to 251.1] | 245.3 [176.0 to 341.9] | 227.5 [158.0 to 327.5] | 203.3 [144.4 to 286.2] | 196.7 [140.8 to 274.9]

60. Secondary Outcome: Microneutralization (MN50) Antibody Responses Influenza A/Brisbane (H1N1 Subtype) Expressed as GMFR
Description: Microneutralization (MN50) antibody responses: neutralizing antibody titers specific to vaccine Influenza A/Brisbane (H1N1 Subtype) antigenically-drifted influenza strains, as measured by a MN assay, expressed as GMFR.
Time Frame: Day 28 to Day 182
Population: Per Protocol Analysis Set population
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean fold rise
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
geometric mean fold rise
  Day 28 | 1.9 [1.4 to 2.4] | 1.9 [1.2 to 3.0] | 1.5 [1.2 to 2.0] | 1.7 [1.3 to 2.2] | 1.7 [1.3 to 2.2] | 1.2 [1.0 to 1.4] | 1.9 [1.5 to 2.3] | 1.4 [1.1 to 1.8] | 1.2 [1.0 to 1.4] | 1.7 [1.3 to 2.3] | 1.4 [1.0 to 1.7] | 1.5 [1.2 to 1.9] | 2.1 [1.6 to 2.8]
  Day 56 | 1.8 [1.4 to 2.3] | 1.6 [1.0 to 2.8] | 1.3 [1.0 to 1.7] | 1.4 [1.1 to 1.7] | 1.4 [1.2 to 1.7] | 1.1 [0.9 to 1.3] | 1.5 [1.2 to 1.9] | 1.2 [0.9 to 1.5] | 1.1 [1.0 to 1.3] | 1.4 [1.1 to 1.9] | 1.3 [1.0 to 1.6] | 1.5 [1.2 to 1.9] | 1.8 [1.3 to 2.4]
  Day 70 | 2.4 [1.8 to 3.2] | 2.5 [1.5 to 4.3] | 1.8 [1.3 to 2.5] | 2.4 [1.6 to 3.6] | 2.3 [1.6 to 3.2] | 1.5 [1.2 to 2.0] | 2.1 [1.7 to 2.7] | 1.8 [1.3 to 2.5] | 1.5 [1.1 to 1.9] | 2.0 [1.4 to 3.0] | 1.7 [1.2 to 2.4] | 2.1 [1.6 to 2.8] | 1.6 [1.3 to 2.2]
  Day 84 | 5.5 [4.1 to 7.4] | 6.6 [3.7 to 11.7] | 4.2 [2.8 to 6.2] | 5.0 [3.4 to 7.5] | 5.2 [3.5 to 7.8] | 2.8 [2.1 to 3.7] | 5.5 [4.3 to 7.0] | 4.8 [3.3 to 7.0] | 3.6 [2.7 to 4.9] | 5.7 [3.6 to 9.0] | 3.8 [2.5 to 5.8] | 5.1 [3.8 to 6.8] | 4.3 [3.2 to 5.8]
  Day 182 | 4.1 [3.1 to 5.5] | 3.6 [2.1 to 6.3] | 2.7 [2.0 to 3.8] | 3.3 [2.3 to 4.7] | 3.4 [2.4 to 4.8] | 2.2 [1.7 to 2.9] | 3.8 [2.9 to 4.9] | 2.9 [2.1 to 4.0] | 2.3 [1.8 to 2.9] | 3.7 [2.5 to 5.4] | 2.0 [1.2 to 3.3] | 3.5 [2.6 to 4.9] | 3.4 [2.6 to 4.4]

61. Secondary Outcome: Microneutralization (MN50) Antibody Responses Influenza A/Kansas (H3N2 Subtype) Expressed as GMFR
Description: Microneutralization (MN50) antibody responses: neutralizing antibody titers specific to vaccine Influenza A/Kansas (H3N2 Subtype) antigenically-drifted influenza strains, as measured by a MN assay, expressed as GMFR.
Time Frame: Day 28 to Day 182
Population: Per Protocol Analysis Set population
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean fold rise
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
geometric mean fold rise
  Day 28 | 4.3 [3.4 to 5.4] | 3.4 [2.1 to 5.5] | 2.7 [2.1 to 3.6] | 3.1 [2.3 to 4.1] | 3.7 [2.5 to 5.4] | 2.8 [2.1 to 3.8] | 4.1 [3.3 to 5.2] | 2.5 [1.9 to 3.3] | 2.2 [1.6 to 2.9] | 4.7 [3.2 to 7.0] | 3.6 [2.7 to 4.7] | 3.6 [2.6 to 5.0] | 6.2 [4.1 to 9.4]
  Day 56 | 3.7 [2.9 to 4.7] | 2.7 [1.7 to 4.5] | 2.3 [1.7 to 3.1] | 2.6 [2.0 to 3.4] | 2.7 [1.9 to 3.7] | 2.5 [1.8 to 3.4] | 3.4 [2.8 to 4.3] | 2.1 [1.6 to 2.8] | 2.0 [1.5 to 2.7] | 3.6 [2.5 to 5.2] | 3.1 [2.3 to 4.1] | 3.2 [2.3 to 4.5] | 4.9 [3.2 to 7.3]
  Day 70 | 5.0 [3.9 to 6.4] | 4.1 [2.5 to 6.7] | 3.6 [2.6 to 5.1] | 4.4 [3.3 to 5.8] | 4.1 [3.0 to 5.6] | 3.5 [2.5 to 5.0] | 4.9 [3.9 to 6.0] | 3.1 [2.2 to 4.2] | 2.7 [2.0 to 3.7] | 4.7 [3.2 to 6.9] | 3.9 [2.9 to 5.3] | 4.0 [2.9 to 5.3] | 4.7 [3.2 to 7.1]
  Day 84 | 4.8 [3.8 to 6.2] | 3.6 [2.3 to 5.7] | 3.7 [2.5 to 5.4] | 3.6 [2.6 to 5.0] | 4.2 [2.9 to 6.3] | 3.0 [2.2 to 4.3] | 5.0 [4.0 to 6.2] | 3.4 [2.5 to 4.7] | 2.7 [2.0 to 3.6] | 5.0 [3.2 to 7.6] | 3.9 [2.8 to 5.3] | 4.1 [3.1 to 5.5] | 4.8 [3.0 to 7.6]
  Day 182 | 3.3 [2.6 to 4.3] | 2.3 [1.5 to 3.6] | 2.1 [1.5 to 3.0] | 2.4 [1.8 to 3.3] | 2.9 [2.1 to 3.9] | 2.2 [1.6 to 3.1] | 3.2 [2.6 to 3.9] | 2.1 [1.6 to 2.9] | 1.8 [1.3 to 2.3] | 3.3 [2.3 to 4.8] | 2.3 [1.7 to 3.2] | 2.7 [2.0 to 3.6] | 3.2 [2.2 to 4.6]

62. Secondary Outcome: Microneutralization (MN50) Antibody Responses Influenza A/Wisconsin (H1N1 Subtype) Expressed as GMFR
Description: Microneutralization (MN50) antibody responses: neutralizing antibody titers specific to vaccine Influenza A/Wisconsin (H1N1 Subtype) antigenically-drifted influenza strains, as measured by a MN assay, expressed as GMFR.
Time Frame: Day 28 to Day 182
Population: Per Protocol Analysis Set population
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean fold rise
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
geometric mean fold rise
  Day 28 | 1.2 [1.0 to 1.3] | 1.1 [0.9 to 1.4] | 1.1 [0.9 to 1.2] | 1.0 [0.9 to 1.1] | 1.0 [1.0 to 1.1] | 1.0 [0.9 to 1.1] | 1.2 [1.0 to 1.3] | 0.9 [0.9 to 1.0] | 0.9 [0.8 to 1.0] | 1.4 [1.1 to 1.7] | 1.0 [0.9 to 1.1] | 1.1 [0.9 to 1.3] | 1.1 [0.9 to 1.3]
  Day 56 | 1.1 [0.9 to 1.2] | 1.0 [0.9 to 1.3] | 1.0 [0.9 to 1.1] | 0.9 [0.8 to 1.0] | 1.0 [0.9 to 1.1] | 0.9 [0.8 to 1.0] | 1.0 [0.8 to 1.1] | 0.9 [0.8 to 1.0] | 0.9 [0.8 to 1.0] | 1.1 [0.9 to 1.3] | 0.9 [0.8 to 1.0] | 1.1 [0.9 to 1.3] | 1.1 [0.9 to 1.3]
  Day 70 | 1.4 [1.1 to 1.6] | 1.2 [1.0 to 1.5] | 1.3 [1.0 to 1.5] | 1.3 [1.1 to 1.5] | 1.3 [1.1 to 1.5] | 1.0 [0.9 to 1.2] | 1.3 [1.1 to 1.5] | 1.0 [0.9 to 1.3] | 0.9 [0.8 to 1.1] | 1.4 [1.1 to 1.8] | 1.2 [1.0 to 1.4] | 1.3 [1.1 to 1.6] | 1.1 [0.9 to 1.4]
  Day 84 | 1.5 [1.3 to 1.8] | 1.3 [1.1 to 1.7] | 1.4 [1.2 to 1.8] | 1.4 [1.1 to 1.7] | 1.5 [1.2 to 1.8] | 1.2 [1.0 to 1.4] | 1.4 [1.2 to 1.7] | 1.2 [1.0 to 1.4] | 1.0 [0.9 to 1.2] | 1.8 [1.3 to 2.4] | 1.4 [1.1 to 1.7] | 1.6 [1.3 to 2.0] | 1.3 [1.0 to 1.6]
  Day 182 | 1.2 [1.0 to 1.4] | 1.0 [0.8 to 1.2] | 1.1 [0.9 to 1.2] | 1.1 [1.0 to 1.3] | 1.1 [1.0 to 1.3] | 1.0 [0.9 to 1.1] | 1.2 [1.0 to 1.3] | 0.9 [0.8 to 1.1] | 0.8 [0.7 to 1.0] | 1.4 [1.0 to 1.8] | 1.0 [0.9 to 1.2] | 1.3 [1.0 to 1.5] | 1.1 [0.9 to 1.3]

63. Secondary Outcome: Microneutralization (MN50) Antibody Responses Influenza A/Cambodia (H3N2 Subtype) Expressed as GMFR
Description: Microneutralization (MN50) antibody responses: neutralizing antibody titers specific to vaccine Influenza A/Cambodia (H3N2 Subtype) antigenically-drifted influenza strains, as measured by a MN assay, expressed as GMFR.
Time Frame: Day 28 to Day 182
Population: Per Protocol Analysis Set population
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean fold rise
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
geometric mean fold rise
  Day 28 | 1.9 [1.6 to 2.3] | 2.0 [1.4 to 3.0] | 1.5 [1.2 to 1.8] | 1.7 [1.3 to 2.2] | 2.2 [1.5 to 3.1] | 1.5 [1.2 to 1.8] | 1.8 [1.5 to 2.2] | 1.4 [1.2 to 1.6] | 1.5 [1.2 to 1.8] | 2.6 [1.8 to 3.7] | 1.9 [1.4 to 2.6] | 1.6 [1.2 to 2.2] | 1.8 [1.4 to 2.3]
  Day 56 | 1.7 [1.5 to 2.1] | 1.8 [1.2 to 2.7] | 1.5 [1.1 to 1.9] | 1.5 [1.2 to 1.9] | 1.6 [1.2 to 2.2] | 1.3 [1.1 to 1.6] | 1.6 [1.4 to 1.9] | 1.3 [1.1 to 1.5] | 1.4 [1.1 to 1.7] | 2.2 [1.5 to 3.1] | 1.7 [1.3 to 2.2] | 1.6 [1.2 to 2.0] | 1.5 [1.2 to 1.9]
  Day 70 | 2.0 [1.7 to 2.3] | 2.2 [1.5 to 3.3] | 1.8 [1.4 to 2.3] | 1.8 [1.4 to 2.4] | 2.2 [1.6 to 3.0] | 1.6 [1.3 to 2.1] | 1.9 [1.6 to 2.3] | 1.5 [1.3 to 1.9] | 1.6 [1.2 to 2.0] | 2.4 [1.6 to 3.5] | 2.1 [1.5 to 2.8] | 1.8 [1.4 to 2.3] | 1.4 [1.1 to 1.7]
  Day 84 | 1.8 [1.5 to 2.1] | 2.0 [1.3 to 3.1] | 1.7 [1.3 to 2.2] | 1.7 [1.3 to 2.4] | 1.9 [1.3 to 2.7] | 1.4 [1.1 to 1.9] | 1.7 [1.4 to 2.1] | 1.5 [1.2 to 1.8] | 1.5 [1.2 to 2.0] | 2.8 [1.8 to 4.3] | 2.1 [1.5 to 2.8] | 1.6 [1.3 to 2.1] | 1.3 [1.1 to 1.7]
  Day 182 | 1.4 [1.2 to 1.6] | 1.5 [1.0 to 2.3] | 1.3 [1.0 to 1.7] | 1.3 [1.0 to 1.8] | 1.4 [1.0 to 1.9] | 1.2 [0.9 to 1.5] | 1.3 [1.1 to 1.6] | 1.2 [1.0 to 1.4] | 1.2 [0.9 to 1.5] | 1.9 [1.3 to 2.8] | 1.5 [1.2 to 2.0] | 1.3 [1.1 to 1.7] | 1.2 [1.0 to 1.5]

64. Secondary Outcome: Microneutralization (MN50) Antibody Responses Influenza A/Hong Kong (H3N2 Subtype) Expressed as GMFR
Description: Microneutralization (MN50) antibody responses: neutralizing antibody titers specific to vaccine Influenza A/Hong Kong (H3N2 Subtype) antigenically-drifted influenza strains, as measured by a MN assay, expressed as GMFR.
Time Frame: Day 28 to Day 182
Population: Per Protocol Analysis Set population
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean fold rise
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
geometric mean fold rise
  Day 28 | 2.2 [1.8 to 2.7] | 2.6 [1.6 to 4.3] | 1.7 [1.3 to 2.2] | 2.0 [1.5 to 2.7] | 2.3 [1.5 to 3.5] | 1.8 [1.4 to 2.5] | 2.6 [2.1 to 3.3] | 1.6 [1.3 to 2.0] | 1.9 [1.5 to 2.5] | 3.2 [2.3 to 4.5] | 2.3 [1.7 to 3.3] | 2.3 [1.6 to 3.2] | 2.4 [1.7 to 3.4]
  Day 56 | 1.9 [1.6 to 2.3] | 2.1 [1.3 to 3.4] | 1.5 [1.2 to 2.0] | 1.6 [1.2 to 2.2] | 1.7 [1.2 to 2.5] | 1.6 [1.2 to 2.0] | 2.1 [1.7 to 2.6] | 1.4 [1.1 to 1.7] | 1.8 [1.4 to 2.3] | 2.4 [1.8 to 3.2] | 2.1 [1.5 to 2.9] | 2.0 [1.4 to 2.7] | 2.0 [1.4 to 2.7]
  Day 70 | 2.3 [1.9 to 2.8] | 2.9 [1.8 to 4.8] | 2.2 [1.6 to 3.0] | 2.2 [1.6 to 3.0] | 2.5 [1.7 to 3.5] | 2.1 [1.5 to 2.9] | 2.7 [2.2 to 3.4] | 1.8 [1.3 to 2.4] | 2.2 [1.6 to 2.9] | 2.8 [2.1 to 3.8] | 2.5 [1.8 to 3.4] | 2.6 [1.8 to 3.5] | 1.9 [1.3 to 2.7]
  Day 84 | 2.1 [1.7 to 2.6] | 3.0 [1.9 to 4.9] | 2.0 [1.5 to 2.9] | 2.0 [1.5 to 2.8] | 2.2 [1.5 to 3.3] | 1.8 [1.2 to 2.6] | 2.6 [2.1 to 3.2] | 2.0 [1.5 to 2.6] | 2.2 [1.6 to 3.1] | 3.2 [2.2 to 4.5] | 2.3 [1.7 to 3.3] | 2.3 [1.7 to 3.2] | 1.7 [1.2 to 2.6]
  Day 182 | 1.5 [1.3 to 1.9] | 2.1 [1.3 to 3.3] | 1.4 [1.0 to 1.9] | 1.6 [1.1 to 2.2] | 1.7 [1.2 to 2.4] | 1.5 [1.0 to 2.2] | 1.8 [1.5 to 2.2] | 1.4 [1.1 to 1.8] | 1.6 [1.2 to 2.1] | 2.2 [1.6 to 3.1] | 1.6 [1.1 to 2.1] | 1.8 [1.3 to 2.6] | 1.4 [1.1 to 2.0]

65. Secondary Outcome: Microneutralization (MN50) Antibody Responses Influenza B/Maryland (Victoria Subtype) Expressed as GMFR
Description: Microneutralization (MN50) antibody responses: neutralizing antibody titers specific to vaccine Influenza B/Maryland (Victoria Subtype) antigenically-drifted influenza strains, as measured by a MN assay, expressed as GMFR.
Time Frame: Day 28 to Day 182
Population: Per Protocol Analysis Set population
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean fold rise
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
geometric mean fold rise
  Day 28 | 1.7 [1.5 to 2.0] | 1.5 [1.3 to 1.9] | 1.3 [1.1 to 1.5] | 1.5 [1.2 to 1.8] | 1.7 [1.4 to 2.2] | 1.3 [1.1 to 1.5] | 1.6 [1.4 to 1.9] | 1.2 [1.1 to 1.4] | 1.2 [1.1 to 1.4] | 1.5 [1.2 to 1.9] | 1.5 [1.2 to 1.8] | 1.5 [1.2 to 1.8] | 2.2 [1.5 to 3.0]
  Day 56 | 1.6 [1.4 to 1.9] | 1.3 [1.1 to 1.7] | 1.2 [1.1 to 1.4] | 1.3 [1.1 to 1.7] | 1.5 [1.2 to 1.8] | 1.2 [1.1 to 1.4] | 1.5 [1.3 to 1.7] | 1.2 [1.1 to 1.3] | 1.2 [1.0 to 1.3] | 1.4 [1.1 to 1.8] | 1.4 [1.1 to 1.7] | 1.4 [1.2 to 1.7] | 1.9 [1.4 to 2.7]
  Day 70 | 1.9 [1.6 to 2.2] | 1.7 [1.4 to 2.1] | 1.4 [1.2 to 1.7] | 1.6 [1.3 to 2.0] | 1.8 [1.5 to 2.2] | 1.4 [1.2 to 1.6] | 1.7 [1.5 to 1.9] | 1.3 [1.1 to 1.5] | 1.3 [1.1 to 1.4] | 1.6 [1.2 to 2.1] | 1.6 [1.3 to 1.9] | 1.6 [1.4 to 1.9] | 1.7 [1.2 to 2.4]
  Day 84 | 3.4 [2.9 to 4.1] | 2.5 [2.0 to 3.3] | 2.4 [1.9 to 3.0] | 3.0 [2.2 to 4.1] | 2.7 [2.0 to 3.6] | 2.1 [1.7 to 2.7] | 2.8 [2.4 to 3.3] | 2.2 [1.9 to 2.7] | 2.0 [1.7 to 2.3] | 3.2 [2.4 to 4.4] | 2.5 [1.9 to 3.2] | 3.2 [2.6 to 4.0] | 2.8 [2.0 to 4.0]
  Day 182 | 2.9 [2.4 to 3.4] | 1.9 [1.5 to 2.5] | 1.9 [1.6 to 2.3] | 2.5 [1.8 to 3.4] | 2.1 [1.6 to 2.6] | 1.9 [1.5 to 2.3] | 2.3 [1.9 to 2.7] | 1.7 [1.4 to 2.0] | 1.7 [1.4 to 1.9] | 2.4 [1.8 to 3.2] | 2.0 [1.6 to 2.6] | 2.4 [2.0 to 2.9] | 2.4 [1.7 to 3.4]

66. Secondary Outcome: Microneutralization (MN50) Antibody Responses Influenza B/Phuket (Yamagata Subtype) Expressed as GMFR
Description: Microneutralization (MN50) antibody responses: neutralizing antibody titers specific to vaccine Influenza B/Phuket (Yamagata Subtype) antigenically-drifted influenza strains, as measured by a MN assay, expressed as GMFR.
Time Frame: Day 28 to Day 182
Population: Per Protocol Analysis Set population
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean fold rise
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
geometric mean fold rise
  Day 28 | 1.7 [1.4 to 2.0] | 1.3 [1.1 to 1.5] | 1.1 [0.9 to 1.3] | 1.2 [1.0 to 1.4] | 1.6 [1.2 to 2.2] | 1.2 [1.1 to 1.4] | 1.5 [1.3 to 1.7] | 1.3 [1.1 to 1.5] | 1.2 [1.1 to 1.3] | 1.6 [1.3 to 2.0] | 1.3 [1.1 to 1.6] | 1.6 [1.3 to 1.9] | 1.7 [1.3 to 2.2]
  Day 56 | 1.6 [1.3 to 1.9] | 1.1 [1.0 to 1.3] | 1.1 [0.9 to 1.2] | 1.2 [1.0 to 1.4] | 1.5 [1.1 to 2.0] | 1.2 [1.1 to 1.4] | 1.3 [1.2 to 1.5] | 1.2 [1.0 to 1.4] | 1.1 [1.0 to 1.2] | 1.4 [1.1 to 1.7] | 1.3 [1.1 to 1.5] | 1.5 [1.2 to 1.8] | 1.6 [1.2 to 2.0]
  Day 70 | 1.9 [1.6 to 2.3] | 1.4 [1.2 to 1.7] | 1.2 [1.0 to 1.5] | 1.5 [1.3 to 1.8] | 1.9 [1.4 to 2.6] | 1.4 [1.2 to 1.6] | 1.6 [1.4 to 1.8] | 1.5 [1.2 to 1.7] | 1.3 [1.1 to 1.5] | 2.0 [1.6 to 2.6] | 1.4 [1.2 to 1.7] | 1.7 [1.4 to 2.1] | 1.5 [1.2 to 1.9]
  Day 84 | 2.9 [2.3 to 3.5] | 1.8 [1.4 to 2.2] | 2.0 [1.5 to 2.6] | 2.1 [1.7 to 2.7] | 2.6 [1.9 to 3.5] | 1.6 [1.4 to 1.9] | 2.4 [2.0 to 2.8] | 2.0 [1.7 to 2.4] | 1.9 [1.5 to 2.4] | 2.9 [2.1 to 4.0] | 1.9 [1.5 to 2.4] | 3.0 [2.4 to 3.8] | 2.1 [1.7 to 2.7]
  Day 182 | 2.3 [1.9 to 2.8] | 1.3 [1.1 to 1.5] | 1.4 [1.1 to 1.7] | 1.8 [1.5 to 2.2] | 2.0 [1.5 to 2.7] | 1.3 [1.1 to 1.6] | 1.8 [1.5 to 2.1] | 1.5 [1.3 to 1.8] | 1.4 [1.2 to 1.7] | 2.1 [1.6 to 2.8] | 1.6 [1.3 to 2.0] | 2.2 [1.7 to 2.7] | 1.8 [1.5 to 2.3]

67. Secondary Outcome: Microneutralization (MN50) Antibody Responses Influenza B/Washington (Victoria Subtype) Expressed as GMFR
Description: Microneutralization (MN50) antibody responses: neutralizing antibody titers specific to vaccine Influenza B/Washington (Victoria Subtype) antigenically-drifted influenza strains, as measured by a MN assay, expressed as GMFR.
Time Frame: Day 28 to Day 182
Population: Per Protocol Analysis Set population
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean fold rise
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
geometric mean fold rise
  Day 28 | 1.7 [1.5 to 2.1] | 1.7 [1.3 to 2.1] | 1.2 [1.0 to 1.5] | 1.6 [1.2 to 2.1] | 1.8 [1.4 to 2.3] | 1.4 [1.1 to 1.6] | 1.7 [1.4 to 2.0] | 1.3 [1.1 to 1.5] | 1.2 [1.1 to 1.4] | 1.5 [1.2 to 2.0] | 1.6 [1.3 to 2.1] | 1.5 [1.2 to 1.8] | 2.3 [1.5 to 3.3]
  Day 56 | 1.6 [1.4 to 1.9] | 1.4 [1.2 to 1.8] | 1.1 [0.9 to 1.3] | 1.4 [1.1 to 1.8] | 1.5 [1.2 to 1.8] | 1.3 [1.1 to 1.5] | 1.5 [1.3 to 1.7] | 1.2 [1.0 to 1.3] | 1.2 [1.0 to 1.4] | 1.4 [1.1 to 1.7] | 1.5 [1.2 to 1.9] | 1.4 [1.1 to 1.8] | 1.9 [1.3 to 2.7]
  Day 70 | 1.9 [1.6 to 2.2] | 1.8 [1.4 to 2.3] | 1.3 [1.0 to 1.6] | 1.7 [1.3 to 2.1] | 1.8 [1.5 to 2.2] | 1.5 [1.2 to 1.8] | 1.7 [1.4 to 1.9] | 1.3 [1.1 to 1.5] | 1.4 [1.2 to 1.6] | 1.6 [1.2 to 2.0] | 1.6 [1.2 to 2.0] | 1.6 [1.4 to 1.9] | 1.8 [1.3 to 2.5]
  Day 84 | 2.0 [1.6 to 2.3] | 1.8 [1.4 to 2.4] | 1.5 [1.2 to 2.0] | 2.1 [1.6 to 2.7] | 1.9 [1.5 to 2.4] | 1.5 [1.1 to 1.9] | 1.8 [1.5 to 2.1] | 1.4 [1.1 to 1.7] | 1.6 [1.3 to 1.9] | 2.1 [1.6 to 2.8] | 1.7 [1.3 to 2.2] | 1.8 [1.4 to 2.3] | 1.9 [1.3 to 2.8]
  Day 182 | 1.6 [1.3 to 1.9] | 1.3 [1.0 to 1.7] | 1.1 [0.9 to 1.3] | 1.7 [1.3 to 2.3] | 1.4 [1.1 to 1.7] | 1.2 [1.0 to 1.5] | 1.6 [1.3 to 1.8] | 1.1 [0.9 to 1.4] | 1.3 [1.1 to 1.6] | 1.6 [1.2 to 2.0] | 1.5 [1.2 to 1.9] | 1.4 [1.2 to 1.7] | 1.6 [1.1 to 2.2]

68. Secondary Outcome: Microneutralization (MN50) Antibody Responses of Vaccine Homologous Influenza A/Brisbane (H1N1 Subtype) Strain Expressed as SCR
Description: Microneutralization (MN50) antibody responses: neutralizing antibody titers specific to vaccine of vaccine homologous Influenza A/Brisbane (H1N1 Subtype) strain expressed as SCR and/or antigenically-drifted influenza strains, as measured by a MN assay, expressed as SCR.
Time Frame: Day 28 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
Percentage of participants
  Day 28 | 12.7 [6.2 to 22.0] | 12.5 [4.2 to 26.8] | 13.2 [4.4 to 28.1] | 5.4 [0.7 to 18.2] | 9.8 [2.7 to 23.1] | 2.5 [0.1 to 13.2] | 12.8 [6.3 to 22.3] | 7.7 [1.6 to 20.9] | 5.1 [0.6 to 17.3] | 17.9 [7.5 to 33.5] | 10.3 [2.9 to 24.2] | 9.8 [2.7 to 23.1] | 10.3 [2.9 to 24.2]
  Day 56 | 11.5 [5.4 to 20.8] | 10.3 [2.9 to 24.2] | 11.1 [3.1 to 26.1] | 5.6 [0.7 to 18.7] | 2.5 [0.1 to 13.2] | 0 [0.0 to 8.8] | 10.1 [4.5 to 19.0] | 5.1 [0.6 to 17.3] | 2.6 [0.1 to 13.8] | 10.8 [3.0 to 25.4] | 5.3 [0.6 to 17.7] | 10.0 [2.8 to 23.7] | 10.3 [2.9 to 24.2]
  Day 70 | 18.4 [10.5 to 29.0] | 12.8 [4.3 to 27.4] | 14.3 [4.8 to 30.3] | 22.2 [10.1 to 39.2] | 17.5 [7.3 to 32.8] | 10.0 [2.8 to 23.7] | 21.1 [12.5 to 31.9] | 18.4 [7.7 to 34.3] | 5.3 [0.6 to 17.7] | 19.4 [8.2 to 36.0] | 13.5 [4.5 to 28.8] | 12.2 [4.1 to 26.2] | 7.9 [1.7 to 21.4]
  Day 84 | 51.9 [40.3 to 63.5] | 53.8 [37.2 to 69.9] | 38.2 [22.2 to 56.4] | 54.3 [36.6 to 71.2] | 46.2 [30.1 to 62.8] | 31.6 [17.5 to 48.7] | 52.6 [40.8 to 64.2] | 47.4 [31.0 to 64.2] | 42.1 [26.3 to 59.2] | 50.0 [32.4 to 67.6] | 29.7 [15.9 to 47.0] | 63.4 [46.9 to 77.9] | 44.7 [28.6 to 61.7]
  Day 182 | 40.5 [29.3 to 52.6] | 28.2 [15.0 to 44.9] | 26.5 [12.9 to 44.4] | 28.6 [14.6 to 46.3] | 38.5 [23.4 to 55.4] | 21.1 [9.6 to 37.3] | 37.3 [26.4 to 49.3] | 21.6 [9.8 to 38.2] | 21.6 [9.8 to 38.2] | 38.9 [23.1 to 56.5] | 21.1 [9.6 to 37.3] | 33.3 [19.1 to 50.2] | 28.9 [15.4 to 45.9]

69. Secondary Outcome: Microneutralization (MN50) Antibody Responses of Vaccine Homologous Influenza A/Kansas (H3N2 Subtype) Strain Expressed as SCR
Description: Microneutralization (MN50) antibody responses: neutralizing antibody titers specific to vaccine of vaccine homologous Influenza A/Kansas (H3N2 Subtype) strain expressed as SCR and/or antigenically-drifted influenza strains, as measured by a MN assay, expressed as SCR.
Time Frame: Day 28 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
Percentage of participants
  Day 28 | 45.6 [34.3 to 57.2] | 27.5 [14.6 to 43.9] | 28.9 [15.4 to 45.9] | 27.0 [13.8 to 44.1] | 31.7 [18.1 to 48.1] | 20.0 [9.1 to 35.6] | 43.6 [32.4 to 55.3] | 25.6 [13.0 to 42.1] | 25.6 [13.0 to 42.1] | 46.2 [30.1 to 62.8] | 38.5 [23.4 to 55.4] | 36.6 [22.1 to 53.1] | 53.8 [37.2 to 69.9]
  Day 56 | 38.5 [27.7 to 50.2] | 28.2 [15.0 to 44.9] | 22.2 [10.1 to 39.2] | 27.8 [14.2 to 45.2] | 27.5 [14.2 to 45.2] | 27.5 [14.6 to 43.9] | 39.2 [28.4 to 50.9] | 23.1 [11.1 to 39.3] | 21.1 [9.6 to 37.3] | 40.5 [24.8 to 50.9] | 28.9 [15.4 to 45.9] | 30.0 [16.6 to 46.5] | 48.7 [32.4 to 65.2]
  Day 70 | 51.3 [39.6 to 63.0] | 38.5 [23.4 to 55.4] | 48.6 [31.4 to 66.0] | 55.6 [38.1 to 72.1] | 47.5 [31.5 to 63.9] | 32.5 [18.6 to 49.1] | 56.6 [44.7 to 67.9] | 31.6 [17.5 to 48.7] | 28.9 [15.4 to 45.9] | 50.0 [32.9 to 67.1] | 40.5 [24.8 to 57.9] | 43.9 [28.5 to 60.3] | 47.4 [31.0 to 64.2]
  Day 84 | 48.1 [36.5 to 59.7] | 38.5 [23.4 to 55.4] | 52.9 [35.1 to 70.2] | 45.7 [28.8 to 63.4] | 48.7 [32.4 to 65.2] | 31.6 [17.5 to 48.7] | 55.3 [43.4 to 66.7] | 34.2 [19.6 to 51.4] | 26.3 [13.4 to 43.1] | 47.1 [29.8 to 64.9] | 32.4 [18.0 to 49.8] | 41.5 [26.3 to 57.9] | 52.6 [35.8 to 69.0]
  Day 182 | 36.5 [25.6 to 48.5] | 25.6 [13.0 to 42.1] | 26.5 [12.9 to 44.4] | 22.9 [10.4 to 40.1] | 25.6 [13.0 to 42.1] | 26.3 [13.4 to 43.1] | 38.7 [27.6 to 50.6] | 21.6 [9.8 to 38.2] | 16.2 [6.2 to 32.0] | 30.6 [16.3 to 48.1] | 13.2 [4.4 to 28.1] | 28.2 [15.0 to 44.9] | 39.5 [24.0 to 56.6]

70. Secondary Outcome: Microneutralization (MN50) Antibody Responses of Vaccine Homologous Influenza A/Wisconsin (H1N1 Subtype) Strain Expressed as SCR
Description: Microneutralization (MN50) antibody responses: neutralizing antibody titers specific to vaccine of vaccine homologous Influenza A/Wisconsin (H1N1 Subtype) strain expressed as SCR and/or antigenically-drifted influenza strains, as measured by a MN assay, expressed as SCR.
Time Frame: Day 28 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
Percentage of participants
  Day 28 | 3.8 [0.8 to 10.7] | 7.5 [1.6 to 20.4] | 2.6 [0.1 to 13.8] | 0 [0.0 to 9.5] | 0 [0.0 to 8.6] | 0 [0.0 to 8.8] | 1.3 [0.0 to 6.9] | 0 [0.0 to 9.0] | 0 [0.0 to 9.0] | 12.8 [4.3 to 27.4] | 0 [0.0 to 9.0] | 4.9 [0.6 to 16.5] | 2.6 [0.1 to 13.5]
  Day 56 | 1.3 [0.0 to 6.9] | 5.1 [0.6 to 17.3] | 0 [0.0 to 9.7] | 0 [0.0 to 9.7] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 1.3 [0.0 to 6.9] | 0 [0.0 to 9.0] | 0 [0.0 to 9.3] | 8.1 [1.7 to 21.9] | 0 [0.0 to 9.3] | 5.0 [0.6 to 16.9] | 2.6 [0.1 to 13.5]
  Day 70 | 6.6 [2.2 to 14.7] | 7.7 [1.6 to 20.9] | 2.9 [0.1 to 14.9] | 2.8 [0.1 to 14.5] | 2.5 [0.1 to 13.2] | 2.5 [0.1 to 13.2] | 7.9 [3.0 to 16.4] | 2.6 [0.1 to 13.8] | 0 [0.0 to 9.3] | 11.1 [3.1 to 26.1] | 2.7 [0.1 to 14.2] | 4.9 [0.6 to 16.5] | 2.6 [0.1 to 13.8]
  Day 84 | 13.0 [6.4 to 22.6] | 12.8 [4.3 to 27.4] | 2.9 [0.1 to 15.3] | 2.9 [0.1 to 14.9] | 7.7 [1.6 to 20.9] | 0 [0.0 to 9.3] | 11.8 [5.6 to 21.3] | 5.3 [0.6 to 17.7] | 2.6 [0.1 to 13.8] | 20.6 [8.7 to 37.9] | 2.7 [0.1 to 14.2] | 14.6 [5.6 to 29.2] | 5.3 [0.6 to 17.7]
  Day 182 | 5.4 [1.5 to 13.3] | 5.1 [0.6 to 17.3] | 0 [0.0 to 10.3] | 2.9 [0.1 to 14.9] | 2.6 [0.1 to 13.5] | 0 [0.0 to 9.3] | 5.3 [1.5 to 13.1] | 2.7 [0.1 to 14.2] | 0 [0.0 to 9.5] | 13.9 [4.7 to 29.5] | 2.6 [0.1 to 13.8] | 2.6 [0.1 to 13.5] | 5.3 [0.6 to 17.7]

71. Secondary Outcome: Microneutralization (MN50) Antibody Responses of Vaccine Homologous Influenza A/Cambodia (H3N2 Subtype) Strain Expressed as SCR
Description: Microneutralization (MN50) antibody responses: neutralizing antibody titers specific to vaccine of vaccine homologous Influenza A/Cambodia (H3N2 Subtype) strain expressed as SCR and/or antigenically-drifted influenza strains, as measured by a MN assay, expressed as SCR.
Time Frame: Day 28 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
Percentage of participants
  Day 28 | 10.3 [2.9 to 24.2] | 17.5 [7.3 to 32.8] | 13.2 [4.4 to 28.1] | 10.8 [3.0 to 25.4] | 14.6 [5.6 to 29.2] | 10.0 [2.8 to 23.7] | 15.4 [8.2 to 25.3] | 5.1 [0.6 to 17.3] | 10.3 [2.9 to 24.2] | 30.8 [17.0 to 47.6] | 17.9 [7.5 to 33.5] | 14.6 [5.6 to 29.2] | 10.3 [2.9 to 24.2]
  Day 56 | 14.1 [7.3 to 23.8] | 15.4 [5.9 to 30.5] | 8.3 [1.8 to 22.5] | 5.6 [0.7 to 18.7] | 10.0 [2.8 to 23.7] | 10.0 [2.8 to 23.7] | 12.7 [6.2 to 22.0] | 2.6 [0.1 to 13.5] | 10.5 [2.9 to 24.8] | 21.6 [9.8 to 38.2] | 18.4 [7.7 to 34.3] | 10.0 [2.8 to 23.7] | 10.3 [2.9 to 24.2]
  Day 70 | 18.4 [10.5 to 29.0] | 23.1 [11.1 to 39.3] | 22.9 [10.4 to 40.1] | 16.7 [6.4 to 32.8] | 20.0 [9.1 to 35.6] | 17.5 [7.3 to 32.8] | 15.8 [8.4 to 26.0] | 7.9 [1.7 to 21.4] | 15.8 [6.0 to 31.3] | 30.6 [16.3 to 48.1] | 21.6 [9.8 to 38.2] | 12.2 [4.1 to 26.2] | 10.5 [2.9 to 24.8]
  Day 84 | 15.6 [8.3 to 25.6] | 20.5 [9.3 to 36.5] | 20.6 [8.7 to 37.9] | 14.3 [4.8 to 30.3] | 15.4 [5.9 to 30.5] | 10.5 [2.9 to 24.8] | 17.1 [9.4 to 27.5] | 2.6 [0.1 to 13.8] | 13.2 [4.4 to 28.1] | 38.2 [22.2 to 56.4] | 24.3 [11.8 to 41.2] | 17.1 [7.2 to 32.1] | 7.9 [1.7 to 21.4]
  Day 182 | 8.1 [3.0 to 16.8] | 17.9 [7.5 to 33.5] | 2.9 [0.1 to 15.3] | 8.6 [1.8 to 23.1] | 10.3 [2.9 to 24.2] | 5.3 [0.6 to 17.7] | 8.0 [3.0 to 16.6] | 2.7 [0.1 to 14.2] | 8.1 [1.7 to 21.9] | 19.4 [8.2 to 36.0] | 10.5 [2.9 to 24.8] | 7.7 [1.6 to 20.9] | 5.3 [0.6 to 17.7]

72. Secondary Outcome: Microneutralization (MN50) Antibody Responses of Vaccine Homologous Influenza A/Hong Kong (H3N2 Subtype) Strain Expressed as SCR
Description: Microneutralization (MN50) antibody responses: neutralizing antibody titers specific to vaccine of vaccine homologous Influenza A/Hong Kong (H3N2 Subtype) strain expressed as SCR and/or antigenically-drifted influenza strains, as measured by a MN assay, expressed as SCR.
Time Frame: Day 28 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
Percentage of participants
  Day 28 | 16.5 [9.1 to 26.5] | 27.5 [14.6 to 43.9] | 15.8 [6.0 to 31.3] | 16.2 [6.2 to 32.0] | 17.1 [7.2 to 32.1] | 17.5 [7.3 to 32.8] | 26.9 [17.5 to 38.2] | 10.3 [2.9 to 24.2] | 23.1 [11.1 to 39.3] | 35.9 [21.2 to 52.8] | 28.2 [15.0 to 44.9] | 29.3 [16.1 to 45.5] | 25.6 [13.0 to 42.1]
  Day 56 | 14.1 [7.3 to 23.8] | 25.6 [13.0 to 42.1] | 16.7 [6.4 to 32.8] | 11.1 [3.1 to 26.1] | 15.0 [5.7 to 29.8] | 15.0 [5.7 to 29.8] | 22.8 [14.1 to 33.6] | 7.7 [1.6 to 20.9] | 15.8 [6.0 to 31.3] | 27.0 [13.8 to 44.1] | 23.7 [11.4 to 40.2] | 22.5 [10.8 to 38.5] | 23.1 [11.1 to 39.3]
  Day 70 | 15.8 [8.4 to 26.0] | 33.3 [19.1 to 50.2] | 22.9 [10.4 to 40.1] | 22.2 [10.1 to 39.2] | 25.0 [12.7 to 41.2] | 20.0 [9.1 to 35.6] | 30.3 [20.2 to 41.9] | 18.4 [7.7 to 34.3] | 31.6 [17.5 to 48.7] | 30.6 [16.3 to 48.1] | 18.9 [8.0 to 35.2] | 26.8 [14.2 to 42.9] | 26.3 [13.4 to 43.1]
  Day 84 | 18.2 [10.3 to 28.6] | 28.2 [15.0 to 44.9] | 26.5 [12.9 to 44.4] | 14.3 [4.8 to 30.3] | 17.9 [7.5 to 33.5] | 26.3 [13.4 to 43.1] | 34.2 [23.7 to 46.0] | 23.7 [11.4 to 40.2] | 28.9 [15.4 to 45.9] | 32.4 [17.4 to 50.5] | 27.0 [13.8 to 44.1] | 26.8 [14.2 to 42.9] | 18.4 [7.7 to 34.3]
  Day 182 | 10.8 [4.8 to 20.2] | 20.5 [9.3 to 36.5] | 14.7 [5.0 to 31.1] | 17.1 [6.6 to 33.6] | 15.4 [5.9 to 30.5] | 15.8 [6.0 to 31.3] | 16.0 [8.6 to 26.3] | 5.4 [0.7 to 18.2] | 13.5 [4.5 to 28.8] | 16.7 [6.4 to 32.8] | 7.9 [1.7 to 21.4] | 20.5 [9.3 to 36.5] | 10.5 [4.8 to 20.2]

73. Secondary Outcome: Microneutralization (MN50) Antibody Responses of Vaccine Homologous Influenza B/Maryland (Victoria Subtype) Strain Expressed as SCR
Description: Microneutralization (MN50) antibody responses: neutralizing antibody titers specific to vaccine of vaccine homologous Influenza B/Maryland (Victoria Subtype) strain expressed as SCR and/or antigenically-drifted influenza strains, as measured by a MN assay, expressed as SCR.
Time Frame: Day 28 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
Percentage of participants
  Day 28 | 10.1 [4.5 to 19.0] | 10.0 [2.8 to 23.7] | 2.6 [0.1 to 13.8] | 2.7 [0.1 to 14.2] | 4.9 [0.6 to 16.5] | 2.5 [0.1 to 13.2] | 5.1 [1.4 to 12.6] | 0 [0.0 to 9.0] | 2.6 [0.1 to 13.5] | 7.7 [1.6 to 20.9] | 7.7 [1.6 to 20.9] | 9.8 [2.7 to 23.1] | 17.9 [7.5 to 33.5]
  Day 56 | 10.3 [4.5 to 19.2] | 7.7 [1.6 to 20.9] | 2.8 [0.1 to 14.5] | 2.8 [0.1 to 14.5] | 2.5 [0.1 to 13.2] | 2.5 [0.1 to 13.2] | 5.1 [1.4 to 12.5] | 0 [0.0 to 9.0] | 0 [0.0 to 9.3] | 8.1 [1.7 to 21.9] | 5.3 [0.6 to 17.7] | 5.0 [0.6 to 16.9] | 15.4 [5.9 to 30.5]
  Day 70 | 13.2 [6.5 to 22.9] | 10.3 [2.9 to 24.2] | 5.7 [0.7 to 19.2] | 5.6 [0.7 to 18.7] | 2.5 [0.1 to 13.2] | 5.0 [0.6 to 16.9] | 5.3 [1.5 to 12.9] | 2.6 [0.1 to 13.8] | 2.6 [0.1 to 13.8] | 8.3 [1.8 to 22.5] | 10.8 [3.0 to 25.4] | 4.9 [0.6 to 16.5] | 13.2 [4.4 to 28.1]
  Day 84 | 35.1 [24.5 to 46.8] | 23.1 [11.1 to 39.3] | 20.6 [8.7 to 37.9] | 20.0 [8.4 to 36.9] | 20.5 [9.3 to 36.5] | 21.1 [9.6 to 37.3] | 25.0 [15.8 to 36.3] | 15.8 [6.0 to 31.3] | 10.5 [2.9 to 24.8] | 38.2 [22.2 to 56.4] | 16.2 [6.2 to 32.0] | 31.7 [18.1 to 48.1] | 21.1 [9.6 to 37.3]
  Day 182 | 13.2 [4.4 to 28.1] | 15.4 [5.9 to 30.5] | 2.9 [0.1 to 15.3] | 20.0 [8.4 to 36.9] | 15.4 [5.9 to 30.5] | 13.2 [4.4 to 28.1] | 17.3 [9.6 to 27.8] | 5.4 [0.7 to 18.2] | 2.7 [0.1 to 14.2] | 22.2 [10.1 to 39.2] | 7.9 [1.7 to 21.4] | 20.5 [9.3 to 36.5] | 13.2 [4.4 to 28.1]

74. Secondary Outcome: Microneutralization (MN50) Antibody Responses of Vaccine Homologous Influenza B/Phuket (Yamagata Subtype) Strain Expressed as SCR
Description: Microneutralization (MN50) antibody responses: neutralizing antibody titers specific to vaccine of vaccine homologous Influenza B/Phuket (Yamagata Subtype) strain expressed as SCR and/or antigenically-drifted influenza strains, as measured by a MN assay, expressed as SCR.
Time Frame: Day 28 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
Percentage of participants
  Day 28 | 7.6 [2.8 to 15.8] | 5.0 [0.6 to 16.9] | 2.6 [0.1 to 13.8] | 5.4 [0.7 to 18.2] | 9.8 [2.7 to 23.1] | 0 [0.0 to 8.8] | 5.1 [1.4 to 12.6] | 5.1 [0.6 to 17.3] | 0 [0.0 to 9.0] | 5.1 [0.6 to 17.3] | 2.6 [0.1 to 13.5] | 7.3 [1.5 to 19.9] | 15.4 [5.9 to 30.5]
  Day 56 | 9.0 [3.7 to 17.6] | 5.1 [0.6 to 17.3] | 0 [0.0 to 9.7] | 5.6 [0.7 to 18.7] | 10.0 [2.8 to 23.7] | 2.5 [0.1 to 13.2] | 3.8 [0.8 to 10.7] | 2.6 [0.1 to 13.5] | 0 [0.0 to 9.3] | 5.4 [0.7 to 18.2] | 2.6 [0.1 to 13.8] | 10.0 [2.8 to 23.7] | 12.8 [4.3 to 27.4]
  Day 70 | 10.5 [4.7 to 19.7] | 5.1 [0.6 to 17.3] | 5.7 [0.7 to 19.2] | 8.3 [1.8 to 22.5] | 12.5 [4.2 to 26.8] | 0 [0.0 to 8.8] | 9.2 [3.8 to 18.1] | 5.3 [0.6 to 17.7] | 2.6 [0.1 to 13.8] | 13.9 [4.7 to 29.5] | 5.4 [0.7 to 18.2] | 9.8 [2.7 to 23.1] | 13.2 [4.4 to 28.1]
  Day 84 | 24.7 [15.6 to 35.7] | 10.3 [2.9 to 24.2] | 14.7 [5.0 to 31.1] | 20.0 [8.4 to 36.9] | 33.3 [19.1 to 50.2] | 5.3 [0.6 to 17.7] | 19.7 [11.5 to 30.5] | 15.8 [6.0 to 31.3] | 10.5 [2.9 to 24.8] | 35.3 [19.7 to 53.5] | 13.5 [4.5 to 28.8] | 29.3 [16.1 to 45.5] | 18.4 [7.7 to 34.3]
  Day 182 | 10.8 [4.8 to 20.2] | 5.1 [0.6 to 17.3] | 8.8 [1.9 to 23.7] | 11.4 [3.2 to 26.7] | 17.9 [7.5 to 33.5] | 2.6 [0.1 to 13.8] | 9.3 [3.8 to 18.3] | 5.4 [0.7 to 18.2] | 2.7 [0.1 to 14.2] | 16.7 [6.4 to 32.8] | 7.9 [1.7 to 21.4] | 23.1 [11.1 to 39.3] | 15.8 [6.0 to 31.3]

75. Secondary Outcome: Microneutralization (MN50) Antibody Responses of Vaccine Homologous Influenza B/Washington (Victoria Subtype) Strain Expressed as SCR
Description: Microneutralization (MN50) antibody responses: neutralizing antibody titers specific to vaccine of vaccine homologous Influenza B/Washington (Victoria Subtype) strain expressed as SCR and/or antigenically-drifted influenza strains, as measured by a MN assay, expressed as SCR.
Time Frame: Day 28 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 39
Percentage of participants
  Day 28 | 8.9 [3.6 to 17.4] | 12.5 [4.2 to 26.8] | 2.6 [0.1 to 13.8] | 8.1 [1.7 to 21.9] | 9.8 [2.7 to 23.1] | 7.5 [1.6 to 20.4] | 9.0 [3.7 to 17.6] | 5.1 [0.6 to 17.3] | 5.1 [0.6 to 17.3] | 10.3 [2.9 to 24.2] | 15.4 [5.9 to 30.5] | 9.8 [2.7 to 23.1] | 23.1 [11.1 to 39.3]
  Day 56 | 7.7 [2.9 to 16.0] | 10.3 [2.9 to 24.2] | 0 [0.0 to 9.7] | 5.6 [0.7 to 18.7] | 5.0 [0.6 to 16.9] | 5.0 [0.6 to 16.9] | 6.3 [2.1 to 14.2] | 0 [0.0 to 9.0] | 2.6 [0.1 to 13.8] | 8.1 [1.7 to 21.9] | 7.9 [1.7 to 21.4] | 7.5 [1.6 to 20.4] | 17.9 [7.5 to 33.5]
  Day 70 | 9.2 [3.8 to 18.1] | 15.4 [5.9 to 30.5] | 5.7 [0.7 to 19.2] | 11.1 [3.1 to 26.1] | 7.5 [1.6 to 20.4] | 7.5 [1.6 to 20.4] | 9.2 [3.8 to 18.1] | 2.6 [0.1 to 13.8] | 5.3 [0.6 to 17.7] | 8.3 [1.8 to 22.5] | 13.5 [4.5 to 28.8] | 4.9 [0.6 to 16.5] | 15.8 [6.0 to 31.3]
  Day 84 | 13.0 [6.4 to 22.6] | 17.9 [7.5 to 33.5] | 14.7 [5.0 to 31.1] | 14.3 [4.8 to 30.3] | 7.7 [1.6 to 20.9] | 10.5 [2.9 to 24.8] | 10.5 [4.7 to 19.7] | 5.3 [0.6 to 17.7] | 5.3 [0.6 to 17.7] | 20.6 [8.7 to 37.9] | 8.1 [1.7 to 21.9] | 14.6 [5.6 to 29.2] | 26.3 [13.4 to 43.1]
  Day 182 | 8.1 [3.0 to 16.8] | 10.3 [2.9 to 24.2] | 2.9 [0.1 to 15.3] | 14.3 [4.8 to 30.3] | 2.6 [0.1 to 13.5] | 7.9 [1.7 to 21.4] | 8.0 [3.0 to 16.6] | 2.7 [0.1 to 14.2] | 2.7 [0.1 to 14.2] | 11.1 [3.1 to 26.1] | 2.6 [0.1 to 13.8] | 2.6 [0.1 to 13.5] | 13.2 [4.4 to 28.1]

76. Secondary Outcome: Microneutralization (MN50) Antibody Responses Specific to Vaccine Homologous Wild-type Influenza A/Brisbane (H1N1 Subtype) Expressed as GMTR
Description: Microneutralization (MN50) antibody responses: neutralizing antibody titers specific to vaccine homologous wild-type Influenza A/Brisbane (H1N1 Subtype) and/or antigenically-drifted influenza strains, as measured by a MN assay , expressed as GMTR.
Time Frame: Day 28 to Day 182
Population: Per Protocol Analysis Set population
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric mean titer ratio
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41
Geometric mean titer ratio
  Day 28 (Comparison to qNIV Reference [Group O] Day 28) | 0.86 [0.62 to 1.19] | 0.70 [0.45 to 1.09] | 0.66 [0.50 to 0.88] | 0.64 [0.49 to 0.85] | 0.74 [0.55 to 1.00] | 0.57 [0.45 to 0.72] | 0.84 [0.62 to 1.14] | 0.63 [0.46 to 0.85] | 0.56 [0.43 to 0.72] | 0.78 [0.55 to 1.11] | 0.70 [0.52 to 0.94] | 0.69 [0.53 to 0.89]
  Day 56 (Comparison to qNIV Reference [Group O] Day 56) | 0.97 [0.70 to 1.36] | 0.76 [0.46 to 1.24] | 0.72 [0.52 to 1.00] | 0.73 [0.53 to 1.00] | 0.76 [0.57 to 1.02] | 0.61 [0.46 to 0.81] | 0.81 [0.60 to 1.10] | 0.64 [0.47 to 0.88] | 0.61 [0.46 to 0.81] | 0.79 [0.55 to 1.13] | 0.77 [0.57 to 1.03] | 0.78 [0.57 to 1.06]
  Day 70 (Comparison to qNIV Reference [Group O] Day 70) | 1.46 [1.04 to 2.05] | 1.27 [0.80 to 2.01] | 1.09 [0.79 to 1.49] | 1.38 [0.96 to 1.99] | 1.33 [0.94 to 1.89] | 0.93 [0.70 to 1.24] | 1.24 [0.92 to 1.66] | 1.08 [0.78 to 1.49] | 0.85 [0.62 to 1.17] | 1.24 [0.86 to 1.79] | 1.16 [0.83 to 1.64] | 1.23 [0.90 to 1.68]
  Day 84 (Comparison to qNIV Reference [Group O] Day 84) | 1.29 [0.90 to 1.86] | 1.24 [0.75 to 2.06] | 0.98 [0.67 to 1.45] | 1.10 [0.74 to 1.64] | 1.18 [0.78 to 1.77] | 0.64 [0.46 to 0.90] | 1.22 [0.90 to 1.67] | 1.12 [0.77 to 1.64] | 0.81 [0.57 to 1.14] | 1.37 [0.88 to 2.13] | 1.06 [0.71 to 1.57] | 1.16 [0.82 to 1.66]
  Day 182 (Comparison to qNIV Reference [Group O] Day 182) | 1.19 [0.83 to 1.71] | 0.89 [0.54 to 1.47] | 0.81 [0.57 to 1.15] | 0.91 [0.63 to 1.31] | 0.98 [0.68 to 1.42] | 0.66 [0.47 to 0.91] | 1.07 [0.78 to 1.49] | 0.85 [0.60 to 1.19] | 0.65 [0.48 to 0.89] | 1.09 [0.72 to 1.63] | 0.65 [0.39 to 1.08] | 1.01 [0.71 to 1.46]
  Day70 (Comparison to qNIV Reference [Group O] Day 28)** | 1.10 [0.79 to 1.53] | 0.94 [0.60 to 1.48] | 0.82 [0.60 to 1.12] | 1.04 [0.72 to 1.49] | 1.00 [0.71 to 1.42] | 0.71 [0.53 to 0.94] | 0.94 [0.70 to 1.26] | 0.82 [0.59 to 1.13] | 0.64 [0.47 to 0.88] | 0.94 [0.66 to 1.35] | 0.93 [0.68 to 1.26] | 1.10 [0.79 to 1.53]

77. Secondary Outcome: Microneutralization (MN50) Antibody Responses Specific to Vaccine Homologous Wild-type Influenza A/Kansas (H3N2 Subtype) Expressed as GMTR
Description: Microneutralization (MN50) antibody responses: neutralizing antibody titers specific to vaccine homologous wild-type Influenza A/Kansas (H3N2 Subtype) and/or antigenically-drifted influenza strains, as measured by a MN assay , expressed as GMTR.
Time Frame: Day 28 to Day 182
Population: Per Protocol Analysis Set population
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric mean titer ratio
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41
Geometric mean titer ratio
  Day 28 (Comparison to qNIV Reference [Group O] Day 28) | 0.73 [0.50 to 1.07] | 0.61 [0.34 to 1.11] | 0.43 [0.28 to 0.64] | 0.52 [0.33 to 0.80] | 0.62 [0.39 to 1.00] | 0.51 [0.33 to 0.77] | 0.70 [0.47 to 1.04] | 0.43 [0.28 to 0.64] | 0.44 [0.29 to 0.68] | 0.73 [0.45 to 1.17] | 0.65 [0.42 to 1.01] | 0.66 [0.42 to 1.05]
  Day 56 (Comparison to qNIV Reference [Group O] Day 56) | 0.81 [0.56 to 1.17] | 0.64 [0.35 to 1.16] | 0.47 [0.30 to 0.74] | 0.57 [0.37 to 0.87] | 0.58 [0.37 to 0.91] | 0.57 [0.37 to 0.88] | 0.75 [0.51 to 1.09] | 0.47 [0.31 to 0.69] | 0.52 [0.34 to 0.80] | 0.72 [0.45 to 1.15] | 0.70 [0.45 to 1.09] | 0.76 [0.48 to 1.20]
  Day 70 (Comparison to qNIV Reference [Group O] Day 70) | 1.16 [0.83 to 1.62] | 1.02 [0.57 to 1.83] | 0.78 [0.50 to 1.20] | 1.00 [0.67 to 1.51] | 0.93 [0.62 to 1.40] | 0.86 [0.55 to 1.33] | 1.11 [0.78 to 1.58] | 0.74 [0.49 to 1.10] | 0.76 [0.50 to 1.16] | 0.96 [0.60 to 1.54] | 0.98 [0.64 to 1.51] | 0.98 [0.64 to 1.50]
  Day 84 (Comparison to qNIV Reference [Group O] Day 84) | 1.29 [0.90 to 1.86] | 1.24 [0.75 to 2.06] | 0.98 [0.67 to 1.45] | 1.10 [0.74 to 1.64] | 1.18 [0.78 to 1.77] | 0.64 [0.46 to 0.90] | 1.22 [0.90 to 1.67] | 1.12 [0.77 to 1.64] | 0.81 [0.57 to 1.14] | 1.37 [0.88 to 2.13] | 1.06 [0.71 to 1.57] | 1.16 [0.82 to 1.66]
  Day 182 (Comparison to qNIV Reference [Group O] Day 182) | 1.19 [0.83 to 1.71] | 0.89 [0.54 to 1.47] | 0.81 [0.57 to 1.15] | 0.91 [0.63 to 1.31] | 0.98 [0.68 to 1.42] | 0.66 [0.47 to 0.91] | 1.07 [0.78 to 1.49] | 0.85 [0.60 to 1.19] | 0.65 [0.48 to 0.89] | 1.09 [0.72 to 1.63] | 0.65 [0.39 to 1.08] | 1.01 [0.71 to 1.46]
  Day70 (Comparison to qNIV Reference [Group O] Day 28)** | 1.19 [0.83 to 1.71] | 0.89 [0.54 to 1.47] | 0.81 [0.57 to 1.15] | 0.91 [0.63 to 1.31] | 0.98 [0.68 to 1.42] | 0.66 [0.47 to 0.91] | 1.07 [0.78 to 1.49] | 0.85 [0.60 to 1.19] | 0.65 [0.48 to 0.89] | 1.09 [0.72 to 1.63] | 0.65 [0.39 to 1.08] | 1.01 [0.71 to 1.46]

78. Secondary Outcome: Microneutralization (MN50) Antibody Responses Specific to Vaccine Homologous Wild-type Influenza A/Wisconsin (H1N1 Subtype) Expressed as GMTR
Description: Microneutralization (MN50) antibody responses: neutralizing antibody titers specific to vaccine homologous wild-type Influenza A/Wisconsin (H1N1 Subtype) and/or antigenically-drifted influenza strains, as measured by a MN assay , expressed as GMTR.
Time Frame: Day 28 to Day 182
Population: Per Protocol Analysis Set population
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric mean titer ratio
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41
Geometric mean titer ratio
  Day 28 (Comparison to qNIV Reference [Group O] Day 28) | 1.02 [0.82 to 1.26] | 0.95 [0.73 to 1.23] | 0.88 [0.71 to 1.08] | 0.88 [0.73 to 1.07] | 0.91 [0.76 to 1.09] | 0.86 [0.71 to 1.04] | 0.99 [0.81 to 1.22] | 0.82 [0.69 to 0.98] | 0.77 [0.64 to 0.92] | 1.16 [0.86 to 1.56] | 0.90 [0.74 to 1.08] | 0.95 [0.76 to 1.19]
  Day 56 (Comparison to qNIV Reference [Group O] Day 56) | 0.99 [0.80 to 1.22] | 0.92 [0.72 to 1.18] | 0.88 [0.71 to 1.09] | 0.83 [0.68 to 1.02] | 0.88 [0.72 to 1.07] | 0.84 [0.69 to 1.01] | 0.88 [0.70 to 1.11] | 0.83 [0.69 to 1.00] | 0.79 [0.65 to 0.95] | 0.98 [0.77 to 1.25] | 0.85 [0.71 to 1.02] | 0.96 [0.76 to 1.22]
  Day 70 (Comparison to qNIV Reference [Group O] Day 70) | 1.20 [0.93 to 1.54] | 1.01 [0.75 to 1.34] | 1.04 [0.80 to 1.35] | 1.13 [0.88 to 1.45] | 1.12 [0.88 to 1.43] | 0.90 [0.72 to 1.12] | 1.09 [0.86 to 1.38] | 0.92 [0.71 to 1.19] | 0.81 [0.65 to 1.01] | 1.19 [0.88 to 1.61] | 1.06 [0.83 to 1.35] | 1.13 [0.87 to 1.47]
  Day 84 (Comparison to qNIV Reference [Group O] Day 84) | 1.16 [0.89 to 1.52] | 0.98 [0.72 to 1.33] | 1.06 [0.80 to 1.41] | 1.04 [0.79 to 1.36] | 1.14 [0.87 to 1.49] | 0.87 [0.67 to 1.14] | 1.07 [0.81 to 1.41] | 0.90 [0.69 to 1.19] | 0.77 [0.60 to 0.98] | 1.38 [0.97 to 1.96] | 1.05 [0.80 to 1.39] | 1.19 [0.88 to 1.61]
  Day 182 (Comparison to qNIV Reference [Group O] Day 182) | 1.08 [0.84 to 1.37] | 0.89 [0.68 to 1.16] | 0.94 [0.72 to 1.22] | 1.01 [0.78 to 1.31] | 1.03 [0.80 to 1.32] | 0.90 [0.70 to 1.15] | 1.06 [0.83 to 1.35] | 0.84 [0.66 to 1.08] | 0.74 [0.57 to 0.95] | 1.26 [0.91 to 1.74] | 0.97 [0.74 to 1.25] | 1.13 [0.86 to 1.49]
  Day70 (Comparison to qNIV Reference [Group O] Day 28)** | 1.18 [0.92 to 1.51] | 1.01 [0.76 to 1.33] | 1.04 [0.81 to 1.34] | 1.13 [0.89 to 1.43] | 1.12 [0.89 to 1.40] | 0.89 [0.72 to 1.10] | 1.08 [0.86 to 1.36] | 0.91 [0.71 to 1.17] | 0.80 [0.65 to 0.98] | 1.18 [0.88 to 1.58] | 1.04 [0.83 to 1.32] | 1.12 [0.88 to 1.44]

79. Secondary Outcome: Microneutralization (MN50) Antibody Responses Specific to Vaccine Homologous Wild-type Influenza A/Cambodia (H3N2 Subtype) Expressed as GMTR
Description: Microneutralization (MN50) antibody responses: neutralizing antibody titers specific to vaccine homologous wild-type Influenza A/Cambodia (H3N2 Subtype) and/or antigenically-drifted influenza strains, as measured by a MN assay , expressed as GMTR.
Time Frame: Day 28 to Day 182
Population: Per Protocol Analysis Set population
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric mean titer ratio
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41
Geometric mean titer ratio
  Day 28 (Comparison to qNIV Reference [Group O] Day 28) | 1.07 [0.78 to 1.46] | 1.13 [0.70 to 1.82] | 0.83 [0.60 to 1.16] | 0.94 [0.66 to 1.34] | 1.21 [0.78 to 1.88] | 0.83 [0.61 to 1.14] | 1.00 [0.73 to 1.38] | 0.78 [0.57 to 1.05] | 0.82 [0.59 to 1.13] | 1.40 [0.91 to 2.15] | 1.09 [0.73 to 1.62] | 0.89 [0.61 to 1.31]
  Day 56 (Comparison to qNIV Reference [Group O] Day 56) | 1.16 [0.88 to 1.54] | 1.17 [0.74 to 1.85] | 0.97 [0.70 to 1.35] | 1.00 [0.72 to 1.38] | 1.08 [0.74 to 1.58] | 0.89 [0.66 to 1.20] | 1.07 [0.80 to 1.44] | 0.84 [0.65 to 1.09] | 0.90 [0.66 to 1.23] | 1.41 [0.93 to 2.13] | 1.15 [0.81 to 1.62] | 1.05 [0.75 to 1.47]
  Day 70 (Comparison to qNIV Reference [Group O] Day 70) | 1.44 [1.09 to 1.89] | 1.61 [1.02 to 2.54] | 1.30 [0.94 to 1.80] | 1.36 [0.96 to 1.92] | 1.61 [1.10 to 2.35] | 1.21 [0.88 to 1.66] | 1.40 [1.04 to 1.88] | 1.12 [0.84 to 1.49] | 1.14 [0.84 to 1.56] | 1.74 [1.14 to 2.67] | 1.52 [1.06 to 2.19] | 1.31 [0.93 to 1.84]
  Day 84 (Comparison to qNIV Reference [Group O] Day 84) | 1.30 [0.97 to 1.74] | 1.50 [0.92 to 2.44] | 1.23 [0.87 to 1.75] | 1.32 [0.92 to 1.90] | 1.39 [0.92 to 2.10] | 1.06 [0.74 to 1.51] | 1.24 [0.90 to 1.70] | 1.10 [0.82 to 1.47] | 1.11 [0.78 to 1.57] | 1.98 [1.25 to 3.14] | 1.53 [1.06 to 2.23] | 1.17 [0.83 to 1.67]
  Day 182 (Comparison to qNIV Reference [Group O] Day 182) | 1.14 [0.89 to 1.47] | 1.27 [0.81 to 2.01] | 1.09 [0.80 to 1.50] | 1.15 [0.83 to 1.61] | 1.16 [0.82 to 1.66] | 0.99 [0.70 to 1.38] | 1.09 [0.82 to 1.45] | 1.03 [0.79 to 1.34] | 0.97 [0.71 to 1.32] | 1.54 [1.03 to 2.32] | 1.29 [0.93 to 1.78] | 1.09 [0.81 to 1.47]
  Day70 (Comparison to qNIV Reference [Group O] Day 28)** | 1.09 [0.82 to 1.46] | 1.24 [0.77 to 1.99] | 0.99 [0.69 to 1.41] | 1.04 [0.72 to 1.51] | 1.22 [0.82 to 1.83] | 0.93 [0.66 to 1.31] | 1.06 [0.78 to 1.45] | 0.86 [0.63 to 1.19] | 0.87 [0.61 to 1.22] | 1.30 [0.83 to 2.04] | 1.16 [0.79 to 1.72] | 0.98 [0.68 to 1.41]

80. Secondary Outcome: Microneutralization (MN50) Antibody Responses Specific to Vaccine Homologous Wild-type Influenza A/Hong Kong (H3N2 Subtype) Expressed as GMTR
Description: Microneutralization (MN50) antibody responses: neutralizing antibody titers specific to vaccine homologous wild-type Influenza A/Hong Kong (H3N2 Subtype) and/or antigenically-drifted influenza strains, as measured by a MN assay , expressed as GMTR.
Time Frame: Day 28 to Day 182
Population: Per Protocol Analysis Set population
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric mean titer ratio
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41
Geometric mean titer ratio
  Day 28 (Comparison to qNIV Reference [Group O] Day 28) | 0.91 [0.64 to 1.31] | 1.07 [0.58 to 1.97] | 0.70 [0.46 to 1.06] | 0.82 [0.53 to 1.26] | 0.95 [0.55 to 1.62] | 0.78 [0.51 to 1.20] | 1.05 [0.71 to 1.55] | 0.66 [0.45 to 0.98] | 0.80 [0.52 to 1.22] | 1.22 [0.76 to 1.96] | 1.00 [0.63 to 1.61] | 0.91 [0.57 to 1.45]
  Day 56 (Comparison to qNIV Reference [Group O] Day 56) | 0.97 [0.69 to 1.36] | 1.07 [0.60 to 1.90] | 0.77 [0.51 to 1.17] | 0.81 [0.53 to 1.24] | 0.88 [0.55 to 1.40] | 0.81 [0.54 to 1.21] | 1.04 [0.71 to 1.52] | 0.72 [0.50 to 1.04] | 0.91 [0.60 to 1.36] | 1.15 [0.74 to 1.78] | 1.09 [0.70 to 1.70] | 0.96 [0.61 to 1.50]
  Day 70 (Comparison to qNIV Reference [Group O] Day 70) | 1.22 [0.86 to 1.74] | 1.52 [0.82 to 2.79] | 1.14 [0.72 to 1.80] | 1.13 [0.72 to 1.79] | 1.29 [0.79 to 2.10] | 1.14 [0.72 to 1.80] | 1.39 [0.95 to 2.04] | 0.94 [0.61 to 1.45] | 1.14 [0.73 to 1.77] | 1.41 [0.88 to 2.25] | 1.34 [0.84 to 2.15] | 1.28 [0.81 to 2.04]
  Day 84 (Comparison to qNIV Reference [Group O] Day 84) | 1.21 [0.83 to 1.77] | 1.72 [0.93 to 3.17] | 1.17 [0.72 to 1.92] | 1.14 [0.70 to 1.84] | 1.29 [0.76 to 2.19] | 1.05 [0.62 to 1.77] | 1.43 [0.97 to 2.09] | 1.15 [0.73 to 1.81] | 1.29 [0.80 to 2.08] | 1.64 [0.99 to 2.71] | 1.41 [0.85 to 2.32] | 1.26 [0.79 to 2.03]
  Day 182 (Comparison to qNIV Reference [Group O] Day 182) | 1.07 [0.76 to 1.53] | 1.42 [0.81 to 2.47] | 0.94 [0.61 to 1.45] | 1.07 [0.70 to 1.65] | 1.18 [0.74 to 1.87] | 1.04 [0.66 to 1.64] | 1.21 [0.86 to 1.71] | 0.99 [0.68 to 1.44] | 1.10 [0.73 to 1.66] | 1.43 [0.91 to 2.24] | 1.11 [0.73 to 1.70] | 1.21 [0.79 to 1.87]
  Day70 (Comparison to qNIV Reference [Group O] Day 28)** | 0.97 [0.69 to 1.37] | 1.20 [0.65 to 2.19] | 0.90 [0.57 to 1.41] | 0.89 [0.57 to 1.40] | 1.02 [0.63 to 1.65] | 0.90 [0.58 to 1.42] | 1.10 [0.76 to 1.59] | 0.75 [0.49 to 1.14] | 0.90 [0.58 to 1.40] | 1.09 [0.69 to 1.73] | 1.07 [0.68 to 1.71] | 1.01 [0.69 to 1.37]

81. Secondary Outcome: Microneutralization (MN50) Antibody Responses Specific to Vaccine Homologous Wild-type Influenza B/Maryland (Victoria Subtype)Expressed as GMTR
Description: Microneutralization (MN50) antibody responses: neutralizing antibody titers specific to vaccine homologous wild-type Influenza B/Maryland (Victoria Subtype) and/or antigenically-drifted influenza strains, as measured by a MN assay , expressed as GMTR.
Time Frame: Day 28 to Day 182
Population: Per Protocol Analysis Set population
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric mean titer ratio
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41
Geometric mean titer ratio
  Day 28 (Comparison to qNIV Reference [Group O] Day 28) | 0.88 [0.68 to 1.15] | 0.78 [0.56 to 1.08] | 0.61 [0.44 to 0.84] | 0.66 [0.46 to 0.95] | 0.85 [0.62 to 1.18] | 0.63 [0.46 to 0.84] | 0.85 [0.65 to 1.12] | 0.66 [0.46 to 0.84] | 0.62 [0.46 to 0.84] | 0.83 [0.59 to 1.116] | 0.76 [0.55 to 1.06] | 0.73 [0.53 to 1.00]
  Day 56 (Comparison to qNIV Reference [Group O] Day 56) | 0.91 [0.70 to 1.19] | 0.77 [0.54 to 1.08] | 0.66 [0.47 to 0.91] | 0.69 [0.48 to 0.99] | 0.83 [0.60 to 1.21] | 0.67 [0.49 to 0.92] | 0.86 [0.66 to 11.3] | 0.69 [0.51 to 0.94] | 0.67 [0.49 to 0.92] | 0.85 [0.60 to 1.21] | 0.78 [0.55 to 1.11] | 00.78 [0.56 to 1.08]
  Day 70 (Comparison to qNIV Reference [Group O] Day 70) | 1.22 [0.92 to 1.60] | 1.10 [0.78 to 1.55] | 0.86 [0.61 to 1.20] | 0.93 [0.65 to 1.33] | 1.15 [0.84 to 1.60] | 0.87 [0.63 to 1.18] | 1.09 [0.84 to 1.43] | 0.84 [0.60 to 1.18] | 0.84 [0.61 to 1.15] | 1.09 [0.74 to 1.59] | 1.01 [0.72 to 1.43] | 1.04 [0.76 to 1.40]
  Day 84 (Comparison to qNIV Reference [Group O] Day 84) | 1.31 [0.96 to 1.78] | 0.99 [0.66 to 1.47] | 0.87 [0.60 to 1.28] | 1.03 [0.68 to 1.56] | 1.02 [0.69 to 1.51] | 0.81 [0.55 to 1.17] | 1.10 [0.81 to 1.49] | 0.88 [0.61 to 1.27] | 0.78 [0.54 to 1.12] | 1.28 [0.82 to 1.98] | 0.85 [0.62 to 1.44] | 1.21 [0.83 to 1.76]
  Day 182 (Comparison to qNIV Reference [Group O] Day 182) | 1.28 [0.95 to 1.72] | 0.86 [0.60 to 1.25] | 0.81 [0.57 to 1.16] | 1.00 [0.67 to 1.50] | 0.91 [0.64 to 1.31] | 0.83 [0.58 to 1.17] | 1.03 [0.76 to 1.40] | 0.76 [0.54 to 1.08] | 0.75 [0.53 to 1.07] | 1.14 [0.77 to 1.69] | 0.88 [0.60 to 1.310] | 1.02 [0.72 to 1.45]
  Day70 (Comparison to qNIV Reference [Group O] Day 28)** | 0.96 [0.73 to 1.25] | 0.87 [0.62 to 1.21] | 0.67 [0.49 to 0.93] | 0.73 [0.51 to 1.03] | 0.91 [0.67 to 1.24] | 0.68 [0.51 to 0.92] | 0.87 [0.67 to 1.12] | 0.67 [0.48 to 0.93] | 0.67 [0.49 to 0.90] | 0.87 [0.60 to 1.25] | 0.80 [0.58 to 1.12] | 0.82 [0.61 to 1.10]

82. Secondary Outcome: Microneutralization (MN50) Antibody Responses Specific to Vaccine Homologous Wild-type Influenza B/Phuket (Yamagata Subtype) Expressed as GMTR
Description: Microneutralization (MN50) antibody responses: neutralizing antibody titers specific to vaccine homologous wild-type Influenza B/Phuket (Yamagata Subtype) and/or antigenically-drifted influenza strains, as measured by a MN assay , expressed as GMTR.
Time Frame: Day 28 to Day 182
Population: Per Protocol Analysis Set population
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric mean titer ratio
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41
Geometric mean titer ratio
  Day 28 (Comparison to qNIV Reference [Group O] Day 28) | 1.01 [0.75 to 1.36] | 0.76 [0.57 to 1.03] | 0.62 [0.46 to 0.83] | 0.72 [0.53 to 0.97] | 0.92 [0.62 to 1.35] | 0.73 [0.55 to 0.96] | 0.85 [0.66 to 1.10] | 0.75 [0.56 to 1.01] | 0.68 [0.52 to 0.89] | 0.95 [0.69 to 1.32] | 0.78 [0.58 to 1.06] | 0.91 [0.66 to 1.26]
  Day 56 (Comparison to qNIV Reference [Group O] Day 56) | 1.01 [0.75 to 1.37] | 0.72 [0.54 to 0.96] | 0.66 [0.50 to 0.87] | 0.74 [0.55 to 1.00] | 0.92 [0.62 to 1.36] | 0.78 [0.60 to 1.02] | 0.84 [0.66 to 1.07] | 0.77 [0.58 to 1.01] | 0.71 [0.54 to 0.92] | 0.88 [0.64 to 1.22] | 0.82 [0.61 to 1.09] | 0.93 [0.68 to 1.27]
  Day 70 (Comparison to qNIV Reference [Group O] Day 70) | 1.32 [0.97 to 1.79] | 0.97 [0.73 to 1.27] | 0.81 [0.61 to 1.08] | 1.03 [0.77 to 1.37] | 1.29 [0.90 to 1.84] | 0.93 [0.71 to 1.21] | 1.06 [0.82 to 1.37] | 0.99 [0.76 to 1.30] | 0.88 [0.67 to 1.14] | 1.37 [0.99 to 1.89] | 0.94 [0.71 to 1.26] | 1.17 [0.86 to 1.58]
  Day 84 (Comparison to qNIV Reference [Group O] Day 84) | 1.39 [1.01 to 1.90] | 0.87 [0.64 to 1.19] | 0.91 [0.66 to 1.25] | 1.03 [0.75 to 1.40] | 1.20 [0.84 to 1.73] | 0.79 [0.60 to 1.04] | 1.12 [0.85 to 1.47] | 0.97 [0.73 to 1.29] | 0.91 [0.67 to 1.23] | 1.37 [0.93 to 2.01] | 0.93 [0.67 to 1.28] | 1.41 [1.02 to 1.95]
  Day 182 (Comparison to qNIV Reference [Group O] Day 182) | 1.28 [0.95 to 1.72] | 0.71 [0.55 to 0.93] | 0.72 [0.54 to 0.98] | 0.98 [0.74 to 1.32] | 1.09 [0.78 to 1.52] | 0.74 [0.58 to 0.96] | 0.95 [0.74 to 1.23] | 0.84 [0.65 to 1.02] | 0.78 [0.60 to 1.02] | 1.16 [0.82 to 1.63] | 0.88 [0.66 to 1.18] | 1.16 [0.85 to 1.57]
  Day70 (Comparison to qNIV Reference [Group O] Day 28)** | 1.14 [0.83 to 1.57] | 0.85 [0.63 to 1.16] | 0.70 [0.51 to 0.96] | 0.89 [0.65 to 1.22] | 1.11 [0.76 to 1.62] | 0.81 [0.60 to 1.09] | 0.91 [0.69 to 1.20] | 0.86 [0.64 to 1.16] | 0.76 [0.56 to 1.02] | 1.19 [0.84 to 1.68] | 0.82 [0.59 to 1.13] | 1.01 [0.73 to 1.40]

83. Secondary Outcome: Microneutralization (MN50) Antibody Responses Specific to Vaccine Homologous Wild-type Influenza B/Washington(VictoriaSubtype) Expressed as GMTR
Description: Microneutralization (MN50) antibody responses: neutralizing antibody titers specific to vaccine homologous wild-type Influenza B/Washington(VictoriaSubtype) and/or antigenically-drifted influenza strains, as measured by a MN assay , expressed as GMTR.
Time Frame: Day 28 to Day 182
Population: Per Protocol Analysis Set population
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric mean titer ratio
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41
Geometric mean titer ratio
  Day 28 (Comparison to qNIV Reference [Group O] Day 28) | 0.85 [0.62 to 1.17] | 0.76 [0.52 to 1.12] | 0.58 [0.40 to 0.84] | 0.73 [0.48 to 1.10] | 0.82 [0.55 to 1.22] | 0.64 [0.44 to 0.94] | 0.81 [0.59 to 1.11] | 0.63 [0.43 to 0.92] | 0.55 [0.38 to 0.81] | 0.76 [0.50 to 1.14] | 0.77 [0.51 to 1.17] | 0.70 [0.48 to 1.01]
  Day 56 (Comparison to qNIV Reference [Group O] Day 56) | 0.91 [0.68 to 1.23] | 0.78 [0.54 to 1.12] | 0.62 [0.44 to 0.89] | 0.74 [0.51 to 1.09] | 0.81 [0.56 to 1.16] | 0.70 [0.49 to 1.00] | 0.83 [0.63 to 1.10] | 0.66 [0.46 to 0.93] | 0.65 [0.46 to 0.93] | 0.79 [0.54 to 1.15] | 0.84 [0.57 to 1.23] | 0.80 [0.54 to 1.17]
  Day 70 (Comparison to qNIV Reference [Group O] Day 70) | 1.16 [0.85 to 1.57] | 1.04 [0.73 to 1.50] | 0.81 [0.57 to 1.15] | 0.97 [0.67 to 1.41] | 1.07 [0.76 to 1.52] | 0.88 [0.62 to 1.25] | 1.01 [0.76 to 1.33] | 0.80 [0.57 to 1.12] | 0.79 [0.56 to 1.11] | 0.97 [0.65 to 1.44] | 1.01 [0.70 to 1.45] | 0.96 [0.70 to 1.32]
  Day 84 (Comparison to qNIV Reference [Group O] Day 84) | 1.11 [0.81 to 1.52] | 0.96 [0.64 to 1.45] | 0.87 [0.59 to 1.29] | 1.07 [0.71 to 1.60] | 1.00 [0.67 to 1.50] | 0.79 [0.53 to 1.18] | 1.01 [0.74 to 1.37] | 0.79 [0.54 to 1.16] | 0.85 [0.58 to 1.25] | 1.19 [0.78 to 1.82] | 0.99 [0.65 to 1.51] | 1.00 [0.69 to 1.46]
  Day 182 (Comparison to qNIV Reference [Group O] Day 182) | 1.10 [0.82 to 1.49] | 0.87 [0.61 to 1.25] | 0.76 [0.54 to 1.08] | 1.11 [0.76 to 1.61] | 0.91 [0.64 to 1.28] | 0.82 [0.57 to 1.18] | 1.06 [0.79 to 1.40] | 0.77 [0.55 to 1.08] | 0.85 [0.60 to 1.20] | 1.08 [0.74 to 1.58] | 1.02 [0.69 to 1.49] | 0.94 [0.67 to 1.33]
  Day70 (Comparison to qNIV Reference [Group O] Day 28)** | 0.91 [0.66 to 1.26] | 0.82 [0.55 to 1.21] | 0.64 [0.43 to 0.94] | 0.76 [0.50 to 1.14] | 0.84 [0.57 to 1.23] | 0.69 [0.47 to 1.02] | 0.79 [0.58 to 1.07] | 0.63 [0.43 to 0.92] | 0.62 [0.42 to 0.91] | 0.77 [0.50 to 1.18] | 0.80 [0.54 to 1.18] | 0.75 [0.53 to 1.08]

84. Secondary Outcome: Serum Immunoglobulin G (IgG) Antibody Concentrations as ELISA Units to the SARS-CoV-2 Wuhan Strain Spike Protein Expressed as Geometric Mean ELISA Unit (GMEU)
Description: IgG geometric mean ELISA unit concentrations (EU/mL) to the SARS-CoV-2 Wuhan Strain spike protein from the matched vaccine construct (and mismatched variant if available), at Days 0, 56, 70, and other follow-up time points.
Time Frame: Day 0 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | SARS-CoV-2 rS With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 40
EU/mL
  Day 0 | 5683.8 [4450.9 to 7258.3] | 4454.2 [2893.6 to 6856.4] | 3856.6 [2822.3 to 5269.9] | 4495.9 [3233.5 to 6251.3] | 4091.0 [2950.8 to 5671.9] | 5180.7 [3838.1 to 6992.9] | 5741.8 [4568.3 to 7216.9] | 3804.2 [2800.4 to 5167.9] | 4523.3 [3465.3 to 5904.5] | 4544.0 [3237.1 to 6378.6] | 4391.3 [3132.1 to 6156.8] | 4626.8 [3265.4 to 6555.7] | 4429.2 [3191.1 to 6147.7]
  Day 28 | 13942.2 [11511.6 to 16885.9] | 7335.6 [4979.4 to 10806.6] | 10956.0 [8766.5 to 13692.2] | 17807.1 [14049.0 to 22570.5] | 9117.3 [6640.0 to 12518.8] | 16742.3 [12369.2 to 22661.5] | 8417.5 [6889.8 to 10284.0] | 8841.9 [6584.3 to 11873.6] | 7891.9 [5957.7 to 10454.0] | 14050.0 [10829.5 to 18228.1] | 7458.5 [5446.8 to 10213.0] | 9746.3 [7411.8 to 12816.3] | 16916.6 [12692.9 to 22545.8]
  Day 56 | 11135.2 [9073.1 to 13666.1] | 5386.6 [3848.3 to 7539.6] | 8964.0 [6963.9 to 11538.5] | 12767.0 [9926.9 to 16419.7] | 6818.0 [5175.7 to 8981.4] | 12182.9 [9259.8 to 16028.8] | 6794.8 [5516.7 to 8369.1] | 6241.6 [4864.5 to 8008.4] | 7333.3 [5785.2 to 9295.7] | 9943.2 [6998.1 to 14127.7] | 5372.8 [4000.2 to 7216.4] | 7345.8 [5496.2 to 9817.9] | 14045.3 [10578.0 to 18649.1]
  Day 70 | 20242.6 [16329.2 to 25093.8] | 10953.8 [8261.7 to 14523.2] | 16790.1 [12876.7 to 21892.9] | 31832.6 [24731.8 to 40972.2] | 14239.8 [11057.4 to 18338.1] | 30516.7 [24805.8 to 37542.3] | 10034.7 [8330.5 to 12087.7] | 14056.4 [11065.9 to 17855.1] | 13323.0 [10080.2 to 17608.9] | 20057.8 [14905.1 to 26991.7] | 9499.5 [7483.6 to 12058.5] | 12008.6 [9222.7 to 15636.0] | 49648.9 [37172.2 to 66313.2]
  Day 84 | 18638.7 [15052.6 to 23079.0] | 9995.0 [7277.5 to 13727.2] | 14734.9 [11353.6 to 19123.2] | 26887.4 [21170.6 to 34147.9] | 13044.7 [10008.3 to 17002.3] | 23187.1 [18124.0 to 29664.6] | 9036.4 [7508.0 to 10875.9] | 13272.6 [9937.1 to 17727.7] | 12165.5 [9252.7 to 15995.5] | 17551.8 [12775.4 to 24114.0] | 8452.8 [6297.0 to 11346.6] | 12333.7 [9385.2 to 16208.7] | 47019.7 [35065.8 to 63048.7]
  Day 182 | 24291.7 [17313.5 to 34082.3] | 30967.6 [20184.3 to 47512.0] | 23902.3 [16449.9 to 34731.0] | 33992.1 [24097.1 to 47950.4] | 17658.7 [12260.0 to 25434.7] | 26514.4 [18000.1 to 39056.1] | 18724.8 [13525.2 to 25923.4] | 27578.7 [18550.2 to 41001.3] | 25514.6 [15700.4 to 41463.6] | 26561.5 [18880.7 to 37366.8] | 15001.9 [8142.9 to 27638.6] | 13145.9 [7396.4 to 23365.0] | 50766.4 [35129.2 to 73364.5]

85. Secondary Outcome: Serum IgG Antibody Concentrations as ELISA Units to the SARS-CoV-2 Omicron BA.1 Variant Spike Protein Expressed as GMEU
Description: IgG geometric mean ELISA unit concentrations (EU/mL) to the SARS-CoV-2 Omicron BA.1 spike protein from the matched vaccine construct (and mismatched variant if available), at Days 0, 56, 70, and other follow-up time points.
Time Frame: Day 0 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | SARS-CoV-2 rS With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 40
EU/mL
  Day 0 | 2509.4 [1957.1 to 3217.4] | 2352.1 [1517.9 to 3644.7] | 1640.8 [1144.5 to 2352.2] | 2223.5 [1602.6 to 3085.0] | 1891.7 [1367.8 to 2616.4] | 2118.1 [1524.3 to 2943.1] | 2338.1 [1833.3 to 2982.1] | 1546.0 [1129.3 to 2116.4] | 2169.7 [1652.6 to 2848.5] | 1836.6 [1239.4 to 2721.6] | 2026.9 [1377.9 to 2981.8] | 1907.4 [1300.7 to 2797.0] | 1924.5 [1411.7 to 2623.7]
  Day 28 | 7178.0 [5886.3 to 8753.2] | 3681.8 [2512.7 to 5395.0] | 5540.0 [4089.2 to 7505.5] | 9164.6 [7181.8 to 11694.8] | 5016.6 [3863.2 to 6514.4] | 9532.8 [7308.3 to 12434.3] | 4771.3 [3897.6 to 5840.8] | 4523.6 [3445.0 to 5939.8] | 4449.2 [3422.2 to 57854.] | 6525.9 [4832.6 to 8812.6] | 3337.6 [2354.9 to 4730.3] | 5146.3 [3778.5 to 7009.2] | 9022.0 [6966.5 to 11684.0]
  Day 56 | 4944.6 [4042.6 to 6047.8] | 2401.9 [1686.2 to 3421.3] | 4066.0 [3129.3 to 5283.1] | 6627.4 [5200.3 to 8446.1] | 3169.4 [2333.5 to 4304.6] | 5695.2 [4018.5 to 8071.5] | 3153.4 [2518.2 to 3948.8] | 3025.0 [2285.5 to 4003.8] | 3104.4 [2409.2 to 4000.2] | 4874.6 [3484.8 to 6818.7] | 2486.6 [1763.6 to 3506.0] | 3418.5 [2490.4 to 4692.4] | 6174.1 [4706.2 to 8099.7]
  Day 70 | 10131.1 [8119.8 to 12640.7] | 5996.7 [4255.9 to 8449.7] | 8505.0 [6469.9 to 11180.4] | 17713.1 [13344.9 to 23511.2] | 7554.2 [5905.9 to 9662.7] | 15278.3 [11882.4 to 19644.8] | 5213.9 [4241.2 to 6409.6] | 8810.1 [6663.7 to 11647.8] | 7595.8 [5620.7 to 10264.9] | 9771.5 [6885.5 to 13867.1] | 4807.0 [3620.2 to 6382.9] | 5959.0 [4480.2 to 7925.9] | 29688.8 [21629.2 to 40751.6]
  Day 84 | 9816.0 [7858.0 to 12261.8] | 5433.7 [3861.9 to 7645.3] | 8251.7 [5870.6 to 11598.5] | 17296.1 [13366.6 to 22380.7] | 7548.7 [5780.4 to 9857.9] | 17095.5 [13534.1 to 21594.1] | 4820.6 [3927.4 to 5916.8] | 9228.5 [6671.3 to 12765.8] | 7392.8 [5384.3 to 10150.6] | 9687.1 [6844.1 to 13711.1] | 4501.4 [3405.1 to 5950.5] | 5899.3 [4311.0 to 8072.9] | 29386.3 [22037.7 to 39185.1]
  Day 182 | 11537.2 [8148.0 to 16336.1] | 13357.2 [8842.6 to 20176.7] | 11651.7 [7261.4 to 18696.5] | 18548.4 [12711.6 to 27065.1] | 8631.2 [6113.1 to 12186.5] | 13600.4 [9274.6 to 19943.7] | 8827.8 [6412.1 to 12153.5] | 14569.4 [9359.6 to 22679.3] | 11423.9 [7309.8 to 17853.3] | 9692.8 [6381.5 to 14722.3] | 6533.1 [3364.0 to 12687.8] | 6134.1 [3521.6 to 10684.7] | 25661.9 [17621.8 to 37370.1]

86. Secondary Outcome: Serum IgG Antibody Concentrations as ELISA Units to the SARS-CoV-2 Wuhan Strain Spike Protein Expressed as GMFR
Description: as for outcome 84
Time Frame: Day 28 to Day 182
Population: Per Protocol Analysis Set population
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean fold rise
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | SARS-CoV-2 rS With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 40
geometric mean fold rise
  Day 28 | 2.5 [2.1 to 2.8] | 1.6 [1.4 to 2.0] | 2.8 [2.2 to 3.4] | 4.0 [2.9 to 5.4] | 2.2 [1.8 to 2.8] | 3.2 [2.6 to 4.1] | 1.5 [1.3 to 1.7] | 2.3 [1.8 to 2.9] | 1.7 [1.4 to 2.2] | 3.2 [2.4 to 4.2] | 1.7 [1.4 to 2.0] | 2.1 [1.7 to 2.6] | 3.8 [2.9 to 5.0]
  Day 56 | 1.9 [1.7 to 2.2] | 1.4 [1.1 to 1.6] | 2.1 [1.7 to 2.6] | 2.8 [2.1 to 3.8] | 1.7 [1.4 to 2.1] | 2.4 [1.9 to 3.0] | 1.2 [1.1 to 1.3] | 1.6 [1.3 to 2.1] | 1.7 [1.3 to 2.1] | 2.3 [1.8 to 2.9] | 1.2 [1.0 to 1.5] | 1.6 [1.3 to 2.0] | 3.2 [2.5 to 4.1]
  Day 70 | 3.5 [2.9 to 4.1] | 2.7 [2.2 to 3.5] | 3.9 [3.0 to 5.0] | 7.1 [4.8 to 10.4] | 3.5 [2.7 to 4.6] | 5.9 [4.4 to 7.9] | 1.8 [1.5 to 2.1] | 3.8 [2.8 to 5.1] | 3.0 [2.3 to 4.0] | 4.8 [3.7 to 6.4] | 2.0 [1.6 to 2.4] | 2.6 [2.0 to 3.3] | 11.2 [8.2 to 15.3]
  Day 84 | 3.3 [2.8 to 3.9] | 2.5 [1.8 to 3.5] | 3.6 [2.8 to 4.6] | 6.2 [4.4 to 8.8] | 3.0 [2.3 to 4.0] | 4.3 [3.2 to 5.7] | 1.6 [1.4 to 1.9] | 3.6 [2.5 to 5.0] | 2.8 [2.1 to 3.7] | 4.3 [3.2 to 5.8] | 1.7 [1.3 to 2.3] | 2.7 [1.9 to 3.7] | 10.6 [7.6 to 14.8]
  Day 182 | 4.5 [3.4 to 5.9] | 6.2 [3.6 to 10.8] | 5.0 [3.4 to 7.5] | 7.6 [4.8 to 12.1] | 4.0 [2.5 to 6.3] | 5.0 [3.4 to 7.3] | 3.0 [2.1 to 4.4] | 7.2 [4.1 to 12.3] | 6.1 [3.9 to 9.6] | 6.5 [4.3 to 9.8] | 3.5 [2.1 to 5.9] | 2.6 [1.6 to 4.1] | 10.7 [6.6 to 17.3]

87. Secondary Outcome: Serum IgG Antibody Concentrations as ELISA Units to the SARS-CoV-2 Omicron BA.1 Variant Spike Protein Expressed as GMFR
Description: IgG geometric mean ELISA unit concentrations (EU/mL) to the SARS-CoV-2 Omicron BA.1 Variant spike protein from the matched vaccine construct (and mismatched variant if available), at Days 0, 56, 70, and other follow-up time points.
Time Frame: Day 28 to Day 182
Population: Per Protocol Analysis Set population
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean fold rise
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | SARS-CoV-2 rS With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 40
geometric mean fold rise
  Day 28 | 2.9 [2.4 to 3.4] | 1.6 [1.3 to 1.9] | 3.3 [2.4 to 4.4] | 4.1 [2.9 to 5.9] | 2.7 [2.0 to 3.6] | 4.5 [3.5 to 5.9] | 2.1 [1.8 to 2.4] | 2.9 [2.2 to 3.8] | 2.1 [1.6 to 2.6] | 3.6 [2.6 to 5.0] | 1.6 [1.3 to 2.2] | 2.7 [2.0 to 3.7] | 4.7 [3.7 to 6.0]
  Day 56 | 2.0 [1.7 to 2.3] | 1.1 [0.9 to 1.4] | 2.2 [1.7 to 2.8] | 3.0 [2.1 to 4.2] | 1.7 [1.3 to 2.2] | 2.7 [2.0 to 3.6] | 1.3 [1.2 to 1.5] | 2.0 [1.5 to 2.5] | 1.5 [1.2 to 1.9] | 2.8 [2.1 to 3.7] | 1.2 [0.9 to 1.5] | 1.8 [1.4 to 2.4] | 3.2 [2.5 to 4.1]
  Day 70 | 4.0 [3.2 to 4.9] | 2.9 [2.2 to 3.8] | 4.4 [3.3 to 5.9] | 8.0 [5.4 to 11.8] | 4.1 [2.9 to 5.8] | 7.2 [5.1 to 10.2] | 2.2 [1.9 to 2.6] | 5.9 [4.1 to 8.6] | 3.6 [2.6 to 5.1] | 5.8 [4.1 to 8.3] | 2.1 [1.6 to 2.8] | 3.1 [2.1 to 4.7] | 15.4 [10.9 to 21.8]
  Day 84 | 3.9 [3.3 to 4.7] | 2.6 [2.0 to 3.4] | 4.6 [3.2 to 6.6] | 8.1 [5.4 to 12.1] | 3.9 [2.7 to 5.6] | 7.6 [5.3 to 10.8] | 2.1 [1.8 to 2.5] | 6.2 [4.1 to 9.5] | 3.5 [2.5 to 4.9] | 5.6 [4.1 to 7.6] | 2.0 [1.5 to 2.6] | 3.1 [2.1 to 4.5] | 15.3 [10.8 to 21.7]
  Day 182 | 4.8 [3.3 to 6.5] | 5.5 [3.3 to 9.2] | 5.7 [3.5 to 9.1] | 8.7 [5.2 to 14.4] | 4.3 [2.8 to 6.6] | 6.3 [4.1 to 9.7] | 3.3 [2.3 to 4.7] | 9.3 [5.2 to 16.6] | 5.7 [3.8 to 8.5] | 6.1 [3.7 to 10.1] | 3.2 [1.9 to 5.5] | 3.2 [1.7 to 5.9] | 13.0 [8.0 to 21.1]

88. Secondary Outcome: Serum IgG Antibody Concentrations as ELISA Units to the SARS-CoV-2 Wuhan Strain Spike Protein Expressed as SCR
Description: as for outcome 84
Time Frame: Day 28 to Day 182
Population: Per Protocol Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | SARS-CoV-2 rS With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 40
Percentage of participants
  Day 28 | 17.7 [10.0 to 27.9] | 10.0 [2.8 to 23.7] | 28.9 [15.4 to 45.9] | 48.6 [31.9 to 65.6] | 12.2 [4.1 to 26.2] | 40.0 [24.9 to 56.7] | 3.9 [0.8 to 11.0] | 30.8 [17.0 to 47.6] | 10.3 [2.9 to 24.2] | 34.2 [19.6 to 51.4] | 5.1 [0.6 to 17.3] | 17.5 [7.3 to 32.8] | 35.9 [21.2 to 52.8]
  Day 56 | 9.0 [3.7 to 17.6] | 5.1 [0.6 to 17.3] | 19.4 [8.2 to 36.0] | 27.8 [14.2 to 45.2] | 12.5 [4.2 to 26.8] | 20.0 [9.1 to 35.6] | 0 [0.0 to 4.7] | 12.8 [4.3 to 27.4] | 10.5 [2.9 to 24.8] | 22.2 [10.1 to 39.2] | 2.6 [0.1 to 13.8] | 7.5 [1.6 to 20.4] | 30.8 [17.0 to 47.6]
  Day 70 | 44.7 [33.3 to 56.6] | 23.1 [11.1 to 39.3] | 54.3 [36.6 to 71.2] | 63.9 [46.2 to 79.2] | 42.5 [27.0 to 59.1] | 62.5 [45.8 to 77.3] | 12.0 [5.6 to 21.6] | 42.1 [26.3 to 59.2] | 31.6 [17.5 to 48.7] | 57.1 [39.4 to 73.7] | 10.8 [3.0 to 25.4] | 25.0 [12.7 to 41.2] | 86.8 [71.9 to 95.6]
  Day 84 | 39.0 [28.0 to 50.8] | 25.6 [13.0 to 42.1] | 32.4 [17.4 to 50.5] | 62.9 [44.9 to 78.5] | 35.9 [21.2 to 52.8] | 55.3 [38.3 to 71.4] | 6.7 [2.2 to 14.9] | 42.1 [26.3 to 59.2] | 21.1 [9.6 to 37.3] | 54.5 [36.4 to 71.9] | 8.1 [1.7 to 21.9] | 30.0 [16.6 to 46.5] | 78.9 [62.7 to 90.4]
  Day 182 | 50.8 [37.7 to 63.9] | 63.6 [45.1 to 79.6] | 60.0 [40.6 to 77.3] | 64.5 [45.4 to 80.8] | 52.8 [35.5 to 69.6] | 60.6 [42.1 to 77.1] | 43.3 [31.2 to 56.0] | 65.5 [45.7 to 82.1] | 64.5 [45.4 to 80.8] | 66.7 [47.2 to 82.7] | 58.6 [38.9 to 76.5] | 32.3 [16.7 to 51.4] | 76.7 [57.7 to 90.1]

89. Secondary Outcome: Serum IgG Antibody Concentrations as ELISA Units to the SARS-CoV-2 Omicron BA.1 Variant Spike Protein Expressed as SCR
Description: as for outcome 87
Time Frame: Day 28 to Day 182
Population: Per Protocol Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | SARS-CoV-2 rS With Matrix-M1 Adjuvant
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41 | 40
Percentage of participants
  Day 28 | 35.4 [25.0 to 47.0] | 7.5 [1.6 to 20.4] | 50.0 [33.4 to 66.6] | 35.1 [20.2 to 52.5] | 29.3 [16.1 to 45.5] | 57.5 [40.9 to 73.0] | 18.2 [10.3 to 28.6] | 30.8 [17.0 to 47.6] | 17.9 [7.5 to 33.5] | 47.4 [31.0 to 64.2] | 12.8 [4.3 to 27.4] | 25.0 [12.7 to 41.2] | 56.4 [39.6 to 72.2]
  Day 56 | 14.1 [7.3 to 23.8] | 0 [0.0 to 9.0] | 19.4 [8.2 to 36.0] | 33.3 [18.6 to 51.0] | 17.5 [7.3 to 32.8] | 35.0 [20.6 to 51.7] | 2.6 [0.3 to 9.1] | 23.1 [11.1 to 39.3] | 10.5 [2.9 to 24.8] | 30.6 [16.3 to 48.1] | 5.3 [0.6 to 17.7] | 10.0 [2.8 to 23.7] | 30.8 [17.0 to 47.6]
  Day 70 | 47.4 [35.8 to 59.2] | 30.8 [17.0 to 47.6] | 60.0 [42.1 to 76.1] | 66.7 [49.0 to 81.4] | 60.0 [43.3 to 75.1] | 72.5 [56.1 to 85.4] | 24.0 [14.9 to 35.3] | 60.5 [43.4 to 76.0] | 36.8 [21.8 to 54.0] | 62.9 [44.9 to 78.5] | 21.6 [9.8 to 38.2] | 30.0 [16.6 to 46.5] | 92.1 [78.6 to 98.3]
  Day 84 | 46.8 [35.3 to 58.5] | 28.2 [15.0 to 44.9] | 52.9 [35.1 to 70.2] | 62.9 [44.9 to 78.5] | 48.7 [32.4 to 65.2] | 71.1 [54.1 to 84.6] | 17.3 [9.6 to 27.8] | 60.5 [43.4 to 76.0] | 34.2 [19.6 to 51.4] | 60.6 [42.1 to 77.1] | 16.2 [6.2 to 32.0] | 32.5 [18.6 to 49.1] | 92.1 [78.6 to 98.3]
  Day 182 | 54.1 [40.8 to 66.9] | 60.6 [42.1 to 77.1] | 53.3 [34.3 to 71.7] | 67.7 [48.6 to 83.3] | 52.8 [35.5 to 69.6] | 66.7 [48.2 to 82.0] | 47.8 [35.4 to 60.3] | 65.5 [45.7 to 82.1] | 58.1 [39.1 to 75.5] | 60.0 [40.6 to 77.3] | 37.9 [20.7 to 57.7] | 45.2 [27.3 to 64.0] | 86.7 [69.3 to 96.2]

90. Secondary Outcome: Serum IgG Antibody Concentrations as ELISA Units to the SARS-CoV-2 Omicron BA.1 Variant Spike Protein Expressed as Geometric Mean ELISA Unit Ratio (GMEUR)
Description: as for outcome 87
Time Frame: Day 28 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41
ratio
  Day 28 (Comparison to SARS-CoV-2 Reference [Group P]) | 0.68 [0.54 to 0.86] | 0.35 [0.27 to 0.46] | 0.66 [0.49 to 0.89] | 0.97 [0.70 to 1.33] | 0.56 [0.41 to 0.76] | 1.01 [0.76 to 1.35] | 0.47 [0.38 to 0.59] | 0.56 [0.42 to 0.75] | 0.46 [0.35 to 0.62] | 0.75 [0.55 to 1.02] | 0.36 [0.26 to 0.49] | 0.57 [0.42 to 0.78]
  Day 56 (Comparison to SARS-CoV-2 Reference [Group P]) | 0.68 [0.54 to 0.87] | 0.37 [0.28 to 0.49] | 0.67 [0.51 to 0.89] | 1.01 [0.74 to 1.39] | 0.52 [0.39 to 0.71] | 0.87 [0.61 to 1.24] | 0.44 [0.35 to 0.56] | 0.55 [0.41 to 0.75] | 0.48 [0.36 to 0.64] | 0.83 [0.61 to 1.13] | 0.38 [0.28 to 0.52] | 0.56 [0.41 to 0.75]
  Day 70 (Comparison to SARS-CoV-2 Reference [Group P]) | 0.30 [0.21 to 0.41] | 0.19 [0.13 to 0.28] | 0.29 [0.20 to 0.41] | 0.57 [0.38 to 0.86] | 0.26 [0.18 to 0.37] | 0.50 [0.34 to 0.72] | 0.16 [0.12 to 0.21] | 0.32 [0.22 to 0.48] | 0.25 [0.17 to 0.37] | 0.35 [0.23 to 0.52] | 0.15 [0.11 to 0.22] | 0.20 [0.14 to 0.30]
  Day 84 (Comparison to SARS-CoV-2 Reference [Group P]) | 0.29 [0.22 to 0.39] | 0.18 [0.12 to 0.26] | 0.29 [0.19 to 0.43] | 0.58 [0.40 to 0.84] | 0.26 [0.18 to 0.37] | 0.56 [0.39 to 0.80] | 0.15 [0.11 to 0.19] | 0.33 [0.22 to 0.51] | 0.24 [0.16 to 0.36] | 0.34 [0.24 to 0.50] | 0.14 [0.10 to 0.20] | 0.20 [0.14 to 0.30]
  Day 182 (Comparison to SARS-CoV-2 Reference [Group P]) | 0.41 [0.25 to 0.68] | 0.50 [0.29 to 0.87] | 0.45 [0.25 to 0.79] | 0.72 [0.42 to 1.21] | 0.33 [0.20 to 0.55] | 0.52 [0.31 to 0.86] | 0.32 [0.19 to 0.54] | 0.58 [0.33 to 1.03] | 0.44 [0.26 to 0.76] | 0.40 [0.23 to 0.68] | 0.25 [0.13 to 0.48] | 0.24 [0.13 to 0.46]

91. Secondary Outcome: Serum IgG Antibody Concentrations as ELISA Units to the SARS-CoV-2 (Wuhan) Spike Protein Expressed as GMEUR
Description: IgG geometric mean ELISA unit concentrations (EU/mL) to the SARS-CoV-2 (Wuhan) spike protein from the matched vaccine construct (and mismatched variant if available), at Days 0, 56, 70, and other follow-up time points.
Time Frame: Day 28 to Day 182
Population: Per-Protocol Analysis Set Population
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation
Number analyzed (Participants) | 80 | 40 | 39 | 37 | 41 | 41 | 81 | 39 | 39 | 40 | 40 | 41
ratio
  Day 28 (Comparison to SARS-CoV-2 Reference [Group P]) | 0.71 [0.56 to 0.89] | 0.43 [0.33 to 0.57] | 0.69 [0.53 to 0.90] | 1.05 [0.77 to 1.43] | 0.57 [0.42 to 0.77] | 0.90 [0.66 to 1.22] | 0.42 [0.34 to 0.52] | 0.57 [0.42 to 0.78] | 0.46 [0.34 to 0.62] | 0.83 [0.61 to 1.12] | 0.44 [0.33 to 0.59] | 0.56 [0.43 to 0.74]
  Day 56 (Comparison to SARS-CoV-2 Reference [Group P]) | 0.67 [0.54 to 0.83] | 0.41 [0.32 to 0.54] | 0.66 [0.51 to 0.85] | 0.90 [0.67 to 1.22] | 0.51 [0.39 to 0.68] | 0.79 [0.59 to 1.05] | 0.40 [0.33 to 0.50] | 0.48 [0.36 to 0.64] | 0.52 [0.40 to 0.69] | 0.72 [0.53 to 0.97] | 0.39 [0.30 to 0.50] | 0.67 [0.54 to 0.83]
  Day 70 (Comparison to SARS-CoV-2 Reference [Group P]) | 0.35 [0.27 to 0.46] | 0.23 [0.17 to 0.32] | 0.34 [0.25 to 0.47] | 0.64 [0.45 to 0.91] | 0.30 [0.22 to 0.41] | 0.58 [0.43 to 0.79] | 0.18 [0.14 to 0.22] | 0.30 [0.22 to 0.42] | 0.27 [0.19 to 0.38] | 0.42 [0.30 to 0.58] | 0.18 [0.14 to 0.25] | 0.24 [0.17 to 0.32]
  Day 84 (Comparison to SARS-CoV-2 Reference [Group P]) | 0.35 [0.26 to 0.46] | 0.22 [0.15 to 0.32] | 0.32 [0.23 to 0.46] | 0.58 [0.41 to 0.82] | 0.28 [0.20 to 0.40] | 0.46 [0.33 to 0.64] | 0.17 [0.13 to 0.22] | 0.30 [0.21 to 0.44] | 0.26 [0.18 to 0.37] | 0.39 [0.27 to 0.55] | 0.17 [0.12 to 0.25] | 0.26 [0.18 to 0.37]
  Day 182 (Comparison to SARS-CoV-2 Reference [Group P]) | 0.45 [0.28 to 0.72] | 0.61 [0.35 to 1.06] | 0.47 [0.29 to 0.77] | 0.68 [0.42 to 1.10] | 0.35 [0.21 to 0.59] | 0.50 [0.30 to 0.82] | 0.35 [0.20 to 0.59] | 0.55 [0.33 to 0.95] | 0.53 [0.30 to 0.94] | 0.54 [0.34 to 0.87] | 0.31 [0.17 to 0.59] | 0.25 [0.13 to 0.46]

ADVERSE EVENTS:
Time Frame: 6 Month
Arm/Group | Group A and Group C - ICC Vaccine Formulation | Group B -ICC Vaccine Formulation | Group D - ICC Vaccine Formulation | Group E - ICC Vaccine Formulation | Group F- ICC Vaccine Formulation | Group G- ICC Vaccine Formulation | Group H and Group N- ICC Vaccine Formulation | Group I- ICC Vaccine Formulation | Group J -ICC Vaccine Formulation | Group K - ICC Vaccine Formulation | Group L - ICC Vaccine Formulation | Group M -ICC Vaccine Formulation | Group O - qNIV With Matrix-M1 Adjuvant | Group P- SARS-CoV-2 rS With Matrix-M1 Adjuvant
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/40 | 0/39 | 0/37 | 0/41 | 0/41 | 0/81 | 0/39 | 0/39 | 0/40 | 0/40 | 0/41 | 0/39 | 0/40
Serious Adverse Events (participants affected / at risk) | 2/80 | 1/40 | 2/39 | 0/37 | 2/41 | 1/41 | 3/81 | 2/39 | 0/39 | 0/40 | 5/40 | 0/41 | 1/39 | 1/40
Other Adverse Events (participants affected / at risk) | 8/80 | 6/40 | 12/39 | 13/37 | 7/41 | 8/41 | 19/81 | 5/39 | 7/39 | 2/40 | 4/40 | 8/41 | 6/39 | 4/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A and Group C - ICC Vaccine Formulation (N=80) | Group B -ICC Vaccine Formulation (N=40) | Group D - ICC Vaccine Formulation (N=39) | Group E - ICC Vaccine Formulation (N=37) | Group F- ICC Vaccine Formulation (N=41) | Group G- ICC Vaccine Formulation (N=41) | Group H and Group N- ICC Vaccine Formulation (N=81) | Group I- ICC Vaccine Formulation (N=39) | Group J -ICC Vaccine Formulation (N=39) | Group K - ICC Vaccine Formulation (N=40) | Group L - ICC Vaccine Formulation (N=40) | Group M -ICC Vaccine Formulation (N=41) | Group O - qNIV With Matrix-M1 Adjuvant (N=39) | Group P- SARS-CoV-2 rS With Matrix-M1 Adjuvant (N=40)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected bite (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sialoadenitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Scapula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint instability (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A and Group C - ICC Vaccine Formulation (N=80) | Group B -ICC Vaccine Formulation (N=40) | Group D - ICC Vaccine Formulation (N=39) | Group E - ICC Vaccine Formulation (N=37) | Group F- ICC Vaccine Formulation (N=41) | Group G- ICC Vaccine Formulation (N=41) | Group H and Group N- ICC Vaccine Formulation (N=81) | Group I- ICC Vaccine Formulation (N=39) | Group J -ICC Vaccine Formulation (N=39) | Group K - ICC Vaccine Formulation (N=40) | Group L - ICC Vaccine Formulation (N=40) | Group M -ICC Vaccine Formulation (N=41) | Group O - qNIV With Matrix-M1 Adjuvant (N=39) | Group P- SARS-CoV-2 rS With Matrix-M1 Adjuvant (N=40)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (3) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 3 (3) | 3 (3) | 2 (2) | 4 (4) | 3 (3) | 7 (7) | 1 (1) | 4 (4) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are NOT employed by the organization sponsoring the study.

There IS an agreement between the Principal Investigator and the Sponsor (or its agents) that restricts the PI's rights to discuss or publish trial results after the trial is completed.

DOCUMENTS (2):
  • Study Protocol (2022-05-06): https://cdn.clinicaltrials.gov/large-docs/41/NCT04961541/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-28): https://cdn.clinicaltrials.gov/large-docs/41/NCT04961541/SAP_001.pdf